Page: 1

Protocol Number: CA139387

Date: 25-May-2005

# **Clinical Protocol CA139387**

Rollover Study of weekly Paclitaxel (BMS-181339) in Patients with Breast Cancer







This protocol contains information that is confidential and proprietary to Bristol-Myers Squibb (BMS)/Bristol-Myers K.K. (BMKK).

# **SYNOPSIS**

# **Clinical Protocol CA139387**

| <b>Title of Study:</b> Protocol CA139387: Rollover Study of Weekly Paclitaxel (BMS-181339) in Patients with Advanced Breast Cancer. |
|---|
| Estimated Number of Study Centers and Countries/Regions: 5 sites/Japan |
| Study Phase: II |
| Primary Objective: The primary objective is to provide an access to Paclitaxel therapy to all subjects who have completed previous and are deemed to be benefiting from this treatment (and should continue on this therapy) as assessed by the treating investigator(s). Cond study (CA 139-387) will also evaluate the frequency and the severity of observed adverse events in treated study subjects. |
| Study Design: This study is a rollover study designed to provide an access to Paclitaxel therapy to breast cancer subjects who have completed previous and are believed to be benefiting from this treatment as assessed by the treating investigator(s). Only breast cancer patients who have participated in a previous can enroll in this rollover weekly Paclitaxel trial (CA139387) provided that they meet all eligibility criteria. Study subjects will receive weekly Paclitaxel at the dose consistent with their last dose in the previous Phase II weekly Paclitaxel trial. Paclitaxel will be given as a one hour intravenous (iv) infusion on Days 1, 8 15,22, 29, 36 followed by 2 weeks of no treatment (observation). One treatment course will consist of 49 days. Safety assessment required in the protocol should be done at each of these weekly visits. Tumor response will be assessed at the completion of at least every 7 weeks. |
| Number of Subjects per Group: Approximately 10 subjects. |
| Study Population: Patients with advanced breast cancer that have completed therapy in a previous and are proven to be benefiting from it with recommendation of continuation of this treatment, as assessed by the treating investigator(s). |
| Test Product, Dose and Mode of Administration, Duration of Treatment: Paclitaxel will be administered intravenously by a 1-hour infusion for the first week of each treatment course. All patients will receive premedication with Paclitaxel given at the last dose that each individual patient was receiving on the previous The day of the initial drug dose administration on the given course is defined as Day 1 of the treatment course. Subsequent Paclitaxel administrations will be given on Days 8, 15, 22, 29 and 36 followed by two weeks of rest (i.e. until Day 49). One treatment course consists of 49 days total. |
| Reference Therapy, Dose and Mode of Administration, Duration of Treatment: Not applicable. |
| <b>Criteria for Evaluation:</b> Every adverse event shall be evaluated and its severity be graded according to the NCI- Common Toxicity Criteria (NCI-CTC) Ver.2.0 (see Appendix 10; It also includes Japanese-language version translated by the JCOG.). |
| Responses will be assessed according to the "Evaluation Criteria on the Therapeutic Effects in Patients with Advanced or Recurrent Breast Cancer "(Extract) and RECIST criteria (See Appendix 7). |
| Statistical Methods: Demographic data and safety will be summarized using descriptive statistics. |

# **TABLE OF CONTENTS**

| TITLE PAGE | 1 |
|-------------------------------|----|
| SYNOPSIS | 2 |
| TABLE OF CONTENTS | 3 |
| 2 STUDY OBJECTIVES 1 | 11 |
| 2.1 Primary Objective | 11 |
| 2.2 Secondary Objectives | 12 |
| 3 STUDY DESIGN AND EVALUATION | 12 |
| 3.1 Study Design | 12 |
| 3.2 Study Population | |
| 3.3 Criteria for Evaluation | 12 |
| 3.4 Sample Size Determination | 13 |
| 3.5 Interim Analyses | 13 |
| 4 STATISTICAL METHODOLOGY | 13 |
| 4.1 Data Set Descriptions | 13 |

| 4.2 Analyses | 13 |
|---|---|
| 4.2.1 Demographics and Baseline Characteristics | 13 |
| 4.2.2 Efficacy Analyses | 14 |
| 4.2.3 Safety Analyses | 14 |
| 4.2.5 Other Analyses | 14 |
| 5 SUBJECT SELECTION CRITERIA | 14 |
| 5.1 Inclusion Criteria | 14 |
| 5.2 Exclusion Criteria | 16 |
| 6 STUDY CONDUCT | 17 |
| 6.1 Ethics | 17 |
| 6.2 Study Therapy | 19 |
| 6.2.2 Treatment Group Assignment | 19 |
| 6.2.2 Treatment Group Assignment | |
| | 20 |
| 6.2.3 Treatment Administration | 20 |
| 6.2.3 Treatment Administration | <ul><li>20</li><li>20</li><li>21</li></ul> |
| 6.2.3 Treatment Administration | <ul><li>20</li><li>20</li><li>21</li></ul> |
| 6.2.3 Treatment Administration | <ul><li>20</li><li>20</li><li>21</li></ul> |
| 6.2.3 Treatment Administration 6.2.3.1 Method 6.2.3.2 Criteria for re-treatment within the course of therapy 6.2.3.3 Re-treatment Criteria for Course 2 and thereafter. | <ul><li>20</li><li>20</li><li>21</li><li>22</li></ul> |
| 6.2.3 Treatment Administration 6.2.3.1 Method 6.2.3.2 Criteria for re-treatment within the course of therapy 6.2.3.3 Re-treatment Criteria for Course 2 and thereafter. 6.2.4 Dose Modifications | <ul><li>20</li><li>20</li><li>21</li><li>22</li><li>23</li></ul> |
| <ul> <li>6.2.3 Treatment Administration</li> <li>6.2.3.1 Method</li> <li>6.2.3.2 Criteria for re-treatment within the course of therapy</li> <li>6.2.3.3 Re-treatment Criteria for Course 2 and thereafter</li> <li>6.2.4 Dose Modifications</li> <li>6.2.5 Discontinuation of Therapy</li> </ul> | <ul><li>20</li><li>20</li><li>21</li><li>22</li><li>23</li><li>23</li></ul> |
| <ul> <li>6.2.3 Treatment Administration</li> <li>6.2.3.1 Method</li> <li>6.2.3.2 Criteria for re-treatment within the course of therapy</li> <li>6.2.3.3 Re-treatment Criteria for Course 2 and thereafter</li> <li>6.2.4 Dose Modifications</li> <li>6.2.5 Discontinuation of Therapy</li> <li>6.2.6 Treatment Compliance</li> </ul> | <ul><li>20</li><li>20</li><li>21</li><li>22</li><li>23</li><li>23</li><li>24</li></ul> |
| <ul> <li>6.2.3 Treatment Administration</li> <li>6.2.3.1 Method</li> <li>6.2.3.2 Criteria for re-treatment within the course of therapy</li> <li>6.2.3.3 Re-treatment Criteria for Course 2 and thereafter</li> <li>6.2.4 Dose Modifications</li> <li>6.2.5 Discontinuation of Therapy</li> <li>6.2.6 Treatment Compliance</li> <li>6.2.7 Other Guidance</li> </ul> | 20<br>20<br>21<br>22<br>23<br>23<br>24<br>24 |

| 6.5 Non-therapy Precautions and Restrictions | 26 |
|---|---|
| 6.5.1 Precautions | 26 |
| 6.5.2 Restrictions | 27 |
| 6.6 Withdrawal of Subjects from Study | 28 |
| 7 STUDY PROCEDURES AND OBSERVATIONS | 28 |
| 7.1 Flow Chart/Time and Events Schedule | 28 |
| 7.2 Procedures by Visit | 30 |
| 7.2.1 Screening evaluation | 30 |
| 7.2.2 Day 1 of the first therapy course (before infusion) | 30 |
| 7.2.3 Evaluations during each therapy course (on Days 8, 15, 22, 29, 36, 43 of each course) | 31 |
| 7.2.4 Evaluations on Day 1 of Course 2 and thereafter (excluding the first course) | 31 |
| 7.2.5 Discharge evaluations | 32 |
| 7.3 Details of Procedures | 32 |
| 7.3.1 Study Materials | 32 |
| 7.3.2 Safety Assessments | 32 |
| 7.3.2.1 Subjective/objective findings | 32 |
| 7.3.2.2 Blood Pressure | 33 |
| 7.3.2.3 Chest X-ray and PaO2 | 33 |
| 7.3.3 Laboratory Test Assessments | 33 |
| 7.3.4 Efficacy Assessments | 34 |
| 7.3.4.1 Primary Efficacy Assessments | 34 |
| 7.3.4.2 Secondary Efficacy Assessments | 34 |
| 8 INVESTIGATIONAL PRODUCT | 34 |

| aclitaxel CA139387<br>BMS-181339 Clinical Protocol |
|----------------------------------------------------------------|
| 8.1 Investigational Product Identification |
| 8.2 Packaging and Labeling |
| 8.3 Handling and Dispensing of Investigational Product |
| 8.4 Investigational Product Records at Investigational Site(s) |
| 8.5 Return and Destruction of Investigational Product . 36 |
| 8.5.1 Return of Investigational Product |
| 8.5.2 Destruction of Investigational Product 37 |
| 8.6 Retained Samples for |

9.1 Importance of Adverse Event Reporting . 37

9.3 Adverse Events Related to Study Conditions . . . . . 40

9.7 Handling of Serious Adverse Events (SAEs)..... 41

9.8 Laboratory Test Abnormalities . 44

9.9 Other Safety Considerations . 44

40

9.6 Reporting of AE Information Following Study

9 ADVERSE EVENT REPORTING IN CLINICAL TRIALS

| 10.1 Compliance with the Protocol and Protocol | |
|------------------------------------------------|----|
| Revisions | 46 |
| 10.2 Informed Consent | 47 |

| 10.2.1 Informed Consent Procedures | 47 |
|------------------------------------------------------|------------|
| 10.2.2 Subjects Unable to Give Informed Consent | 47 |
| 10.2.2.1 Miscellaneous Circumstances | 47 |
| 10.2.3 Illiterate Subjects | 48 |
| 10.2.4 Update of Informed Consent | 48 |
| 10.3 Monitoring for Protocol Compliance | 48 |
| 10.4 Records and Reports | 49 |
| 10.5 Institutional Review Board/Independent Ethics | |
| Committee (IRB/IEC) | 50 |
| 10.6 Records Retention | 50 |
| 10.7 Study Completion, Termination and Suspension | |
| Study Completion | 50 |
| 10.7.1 Study Completion | 50 |
| 10.7.2 Termination or Suspension of an Entire Study | 51 |
| 10.7.3 Termination or Suspension of the Study at the | <b>5</b> 4 |
| Medical Institution | 51 |
| 11 GLOSSARY OF TERMS AND LIST OF | |
| ABBREVIATIONS | 52 |
| 11.1 Glossary of Terms | 52 |
| 11.2 List of Abbreviations | 52 |
| APPENDIX 1 INFORMED CONSENT ELEMENT | 56 |

| APPENDIX 4 ROLES AND RESPONSIBILITIES OF STUDY RELATED PERSONNEL AND STUDY PERIODD | 63 |
|---|---|
| APPENDIX 5 DEFINITION OF ABNORMAL CHANGES AND OUTCOME OF LABORATORY TESTS | 66 |
| APPENDIX 6 DIRECT ACCESS TO SOURCE DOCUMENTS AND DEFINITION THEREOF | 68 |
| APPENDIX 7 CRITERIA FOR RESPONSEE | 69 |
| APPENDIX 8 PERFORMANCE STATUS | 77 |
| APPENDIX 9 THERAPEUTIC ACTIONS FOR ACUTE ALLERGIC SYMPTOMS, ARRHYTHMIA, HYPOTENSION OR INTERSTITIAL PNEUMONIAA | 78 |
| APPENDIX 10 COMMON TOXICITY CRITERIA | 82 |

Paclitaxel CA139387 BMS-181339 Clinical Protocol







## 2 STUDY OBJECTIVES

# 2.1 Primary Objective

The primary study objectives are as follow:

- 1) To provide the access to Paclitaxel therapy to breast cancer subjects who have completed at least 2 course on the previous conducted in Japan and are believed to be benefiting from this treatment, as assessed by the treating investigator(s).
- 2) To evaluate the frequency and the severity of observed adverse reactions in treated subjects.

# 2.2 Secondary Objectives

The secondary objective is to obtain additional data on the response rate and duration of responses to complement information collected on the previous

#### 3 STUDY DESIGN AND EVALUATION

## 3.1 Study Design

Only subjects who participated in the previous Phase II study may enroll in this rollover study provided that they meet all specified in this protocol inclusion and exclusion criteria. Subjects will receive weekly Paclitaxel at the dose that was their last dose on the previous delivered as a one hour iv infusion on Days 1,8,15,22,29,36 followed by 2 weeks of rest (no therapy). One course of therapy consists of 49 days. The range of doses on this study are expected to be decided based on dose reductions seen in Safety assessment required in the protocol should be done at each of these weekly visits. Response to therapy will be assessed at least every 7 weeks, if clinically indicated.

# 3.2 Study Population

Patients with advanced breast cancer who have completed weekly Paclitaxel dosing in previous and are believed to benefit from this treatment with recommendation to continue this regimen, as assessed by the treating investigator(s).

#### 3.3 Criteria for Evaluation

Observed responses should be evaluated according to the "Evaluation Criteria on the Therapeutic Effects in Patients with Advanced or Recurrent Breast Cancer "(Extracts) and the "RECIST" criteria (See Appendix 7).

Every observed adverse event shall be evaluated according to the NCI Common Toxicity Criteria (NCI-CTC) Ver.2.0 (see Appendix 10, translated by the JCOG Japanese language version will also be available). For any toxicity not defined by the NCI-CTC criteria, it must be classified into the category of "Other toxicity" with detailed description on the toxicity observed and be graded according to the following criteria:

Paclitaxel CA139387 BMS-181339 Clinical Protocol

Grade 0: Normal, normal/within normal range, no toxicity

Grade 1: Minor/Mild toxicity

Grade 2: Medium/Moderate toxicity

Grade 3: Severe/High-grade toxicity

Grade 4: Life-threatening toxicity

Grade 5: Death due to toxicity

# 3.4 Sample Size Determination

Sample size will be determined by the number of appropriate subjects who have completed previous and are eligible to participate in this rollover (CA139387) study. At the present time 9 patients remain on . It is estimated that less than 10 patients will be rolled over to this study from .

## 3.5 Interim Analyses

There are no planned interim analyses. If requested by Japanese regulatory agencies, an interim analysis of this trial may be performed to support the Japanese regulatory filing.

#### 4 STATISTICAL METHODOLOGY

# 4.1 Data Set Descriptions

Subjects who receive at least one dose of weekly Paclitaxel treatment will be included in the baseline, dosing and safety summaries. Data from the previous will be utilized for the demographic data and baseline values in enrolled patients for this rollover trial. To obtain an additional data on a response rate and duration of responses, efficacy data will be collected in this rollover CA139387 study.

# 4.2 Analyses

# 4.2.1 Demographics and Baseline Characteristics

Demographic data, performance status, diagnosis, stage, disease locations, prior treatment(s), and selected baseline laboratory results will be summarized using

Paclitaxel CA139387 BMS-181339 Clinical Protocol

descriptive statistics for all patients who received at least one dose of study medication.

Baseline laboratory measurements will be collected from the data obtained for the participation in a previous

## 4.2.2 Efficacy Analyses

Duration of response will be summarized using descriptive statistics for all responders among response-evaluable patients.

## 4.2.3 Safety Analyses

All patients who received at least one dose of study medication will be included in the safety analysis. Worst toxicity grades per patient will be tabulated for adverse events and laboratory measurements.

# .

## 4.2.5 Other Analyses

Not applicable.

### 5 SUBJECT SELECTION CRITERIA

For entry into the study, the following criteria MUST be met.

#### 5.1 Inclusion Criteria

Only patients enrolled in the previous who have completed dosing and are believed to be benefiting from this treatment with advice to continue this regimen, as assessed by the treating investigator(s), may be considered for this rollover study after meeting study eligibility criteria as listed below.

## Signed written informed consent

1) Give written and voluntary informed consent.

## **Target population**

- 2) Patients should receive at least 2 courses, or more, of \_\_\_\_\_ in the previous study (\_\_\_\_\_) and the efficacy evaluation should be completed and confirmed by the treating investigator(s).
- 3) Patients who maintain bone marrow function and meet the following standards at the time of laboratory test obtained prior to the 1<sup>st</sup> Paclitaxel administration in this rollover study;
- WBC count of 3,000/μL or higher, or absolute neutrophile count (ANC) of 1,500/μL or above.
- Platelet count of 75,000/μL or above.
- 4) Performance Status (PS) of 0 2 (according to Classification Criteria of Performance Status by the Eastern Cooperative Oncology Group-ECOG. (See Appendix 8).

#### Age and Sex

5) Women, ages 20 or older.

Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 2 weeks after the study in such a manner that the risk of pregnancy is minimized.

WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea ≥ 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35mIU/mL]. Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential.

WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication.



## 5.2 Exclusion Criteria

## **Sex and Reproductive Status**

- 1) WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 2 weeks after the study.
- 2) WOCBP using a prohibited contraceptive method (however, prohibited contraceptive methods are not specified in this protocol).
- 3) Women who are pregnant or breastfeeding
- 4) Women with a positive pregnancy test on enrollment or prior to study drug administration.

#### **Target Disease Exceptions**

5) Patients with cerebral metastasis that are associated with clinical symptoms, and/or are associated with surrounding edema, or that require ongoing therapy with steroids or anti-convulsants.

#### **Medical History and Concurrent Diseases**

6) Patients with serious uncontrolled medical illness despite optimal therapy i.e. uncontrolled cardiac disease, unstable angina, cerebrovascular disorder, diabetes mellitus etc; active infection, active gastric ulcer etc.

#### **Allergies and Adverse Drug Reactions**

7) Patients with previous history of serious hypersensitivity reaction to Paclitaxel.

## **Prohibited Therapies and/or Medications**

| 8) | Patients who following their last dose of given on the previous |
|---|---|
| | study received chemotherapy other than, surgical procedure |
| | hormonal therapy, immunotherapy, radiotherapy, physiotherapy and/or othe |
| | therapies against their cancer that may prohibit appropriate evaluation of the |
| | efficacy and safety of Paclitaxel on this rollover study. |

#### **Other Exclusion Criteria**

- 9) Subjects who are compulsorily detained for legal reasons or treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.
- 10) Patients whose final efficacy evaluation is judged as Progressive Disease (PD) by the treating investigator(s) based on the CT or any other images taken within 4 weeks prior to the enrollment in this study.
- 11) Patients with grade 2 or higher peripheral neuropathy and/or grade 2 or higher arthralgia/myalgia despite optimal medical therapy that, in the opinion of treating investigator(s), will make unsafe to continue further Paclitaxel therapy.
- 12) Any serious, clinically unmanageable by standard medical therapy (i.e. G-CSF for neutropenia, blood transfusion for anemia, etc.) adverse event(s), subjective/objective findings, abnormal laboratory values etc. that occur prior to initiation of Paclitxel therapy on this rollover study that, in the opinion of treating investigator(s), will make unsafe to continue further Paclitaxel therapy.



#### 6 STUDY CONDUCT

## 6.1 Ethics

This study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki and will be consistent with International Conference on Harmonization Good Clinical Practice (ICH GCP), Japan GCP and regulatory requirements.

The study will be conducted in compliance with the protocol. The protocol and any Amendments and the subject informed consent will receive Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approval/favorable opinion prior to initiation of the study.

Freely given written informed consent must be obtained from every subject prior to clinical trial participation, including informed consent for any screening procedures conducted to establish subject eligibility for the trial.

Subjects unable to give their written consent (e.g., stroke patients, or subjects with severe dementia) may only be enrolled in the study with the consent of their legally acceptable representatives. The subject must also be informed about the nature of the study to the extent compatible with the subject's understanding, and should they become capable, personally sign and date the consent form as soon as possible.

For further details on informed consent, see Section 10.2.

The rights, safety and well-being of the trial subjects are the most important considerations and should prevail over interests of science and society.

Study personnel involved in conducting this trial will be qualified by education, training, and experience to perform their respective task(s).

This trial will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (e.g., loss of medical licensure, debarment).

Systems with procedures that assure the quality of every aspect of the study will be implemented.

Study site personnel involved in this study must bear in mind that study subjects are at a risk of experiencing adverse events as a result of administration of the investigational product and study-related procedures. Anticipated benefits of the investigational products and anticipated disadvantages to the subjects must be described in the informed consent form and explained to subjects prior to enrollment in this study. During and following a subject's participation in the trial, the head of the medical institution or the investigator should ensure that adequate medical care is provided to a subject for any adverse events, including clinically significant laboratory values, related to the clinical trial.

When serious unexpected events occur in a subject during the course of this study, the investigators should promptly evaluate whether the study should be discontinued, in collaboration with the Sponsor.

All study site and sponsor personnel involved in this study must take the necessary actions to ensure that all information collected about study subjects throughout the study appropriately protects subjects' privacy according to the requirements specified in the criminal law and the pharmaceutical affairs law. This applies, but is not limited to, information collected on the written informed consent, CRFs, source documents,

and publication of study results. Consequently, study subjects should, wherever possible, be identified by subject number.

A detailed summary of the applicable regulatory requirements is provided in Appendix 2.

## 6.2 Study Therapy



## **6.2.2** Treatment Group Assignment

Every potential study patient shall, when she/he fully meets all the eligibility criteria and submits a signed freely given informed consent, be eligible for this study registration. For each study participant, an Investigator/Sub-investigator is required to fill in all necessary items on a case registration form and send it to the Case Registration Center via facsimile as specified below. The Case Registration Center shall confirm that the data described in a registration card sent by an Investigator/Sub-investigator fulfills all inclusion criteria and does not meet any of the exclusion criteria before a case registration. The Case Registration Center shall inform an Investigator/Sub-investigator of the registration number for a registered case by telephone or facsimile. If the data described in a registration card does not fulfill the inclusion criteria or does meet any of the exclusion criteria, the Case Registration Center shall confirm the data in question by discussing it with an Investigator/Sub-investigator and, if the case is ineligible for the study, inform an Investigator/Sub-investigator of this decision by telephone and facsimile.



#### 6.2.3 Treatment Administration

#### 6.2.3.1 Method

The firs Paclitaxel dose on a given course is defined as Day 1 of therapy with subsequent drug administrations being given on Days 8, 15, 22, 29 and 36 followed by 2 weeks of rest (no drug given). One course of treatment will therfore consist of total of 49 days.

1) Pre-medications (also see Section 6.5.1)

The following premedications must be given before each paclitaxel infusion

- Dexamethasone 8 mg i.v.(\*: Dose can be reduced to 4mg → 2mg → 1mg) administered 1 hour before and completed 30 minutes prior to the initiation of the paclitaxel infusion
- Ranitidine 50 mg i.v.- administered 1 hour before and completed 30 minutes prior to the initiation of the paclitaxel infusion
- Diphenhydramine 50 mg p.o.

#### (\*): Dexamethasone:

Dexamethasone dose at the initial administration day (Day 1) shall be the same as the last dose in the previous . If any hypersensitivity reaction was observed at the last dose in the previous Phase II study, a dosage of dexamethasone shall be double of the last dose. During the observation period (Days 1-7), if there are no specific clinical problems, dexamethasone dose for the subsequent week (Day 8) would be allowed to be decreased by half the dose from the previous week (i.e.4mg), if necessary. Consequently, if no clinically significant hypersensitivity reaction is observed in a week following the drug administration, it would be possible to use again a half of the previous dexamethasone dose (i.e. 2mg), if necessary. The minimum dexamethasone dosage however, can not be less then 1 mg). If clinically significant hypersensitivity reaction develops, and it is judged that further continuation of weekly Paclitaxel is in the best patient's interest, dexamethasone dose shall be double the previous dose (e.g. if 8 mg was given and there was an event observed then, the next dexamethasone should be 16 mg) for the subsequent Paclitaxel administrations.

2) Paclitaxel (Day1, 8, 15, 22, 29, 36) (see Section 6.5.1)

After administration of the pre-medications, the patient should receive Paclitaxel dose that is consistent with the last dose(\*) of Paclitaxel that the given patient has received in the previous study

1. This Paclitaxel dose shall be mixed with 250 mL of a saline solution or 5% glucose solution for intravenous infusion given over 1-hour.

(\*) weekly Paclitaxel dose should be reduced, if appropriate, according to the severity of adverse effect(s) observed at the last Paclitaxel treatment in the previous Phase II study according to the "Dose Modification" criteria (See Section 6.2.3)".

Administration of weekly Paclitaxel dose should be given on the expected date of treatment + one day.

| | course 1 | | | | | | | | e 2 |
|---|---|---|---|---|---|---|---|---|---|
| Days | Day1 | Day1 Day8 Day15 Day22 Day29 Day36 Day43 | | | | | | | +++ |
| Paclitaxel | О | О | О | О | О | О | ~ | О | +++ |

## 6.2.3.2 Criteria for re-treatment within the course of therapy

(Days: 8, 15, 22, 29, 36 of a therapy course)

An in-course repeated dosing could be allowed only when the laboratory test values and clinical assessments in the previous week or immediately before Paclitaxel administration meet the following requirements;

- WBC count of 2,000/μL or above, or absolute neutrophile count (ANC) of 1,000/μL or above.
- Platelet count of <u>75,000/μL</u> or above.
- No Grade 2 or higher peripheral neuropathy and/or Grade 2 arthralgia/myalgia despite optimal medical therapy which, in the opinion of treating investigator(s), will make further Paclitaxel therapy unsafe.
- Any serious, clinically unmanageable by standard medical therapy (i.e. G-CSF for neutropenia, blood transfusion for anemia, etc.) adverse event(s), subjective/objective findings, abnormal laboratory values etc. occur that, in the opinion of treating investigator(s), will make unsafe to continue further Paclitaxel therapy.

If the patient does not meet above requirements or if the investigator/sub-investigator judges that, it is in the best patient's interest to delay Paclitaxel dosing, the drug administration shall be postponed by one week. Reasons for this decision should be described in a case report form. A dose modification, if appropriate, should be

performed for a successive in-course dosing. (See Section 6.2.3 "Dose Modification").

The study should be discontinued if more than two consecutive Paclitaxel administrations or more than three out of six doses total within the given treatment course are not delivered. However, in patients with evidence of Paclitaxel anti-tumor effects, as judged by the treating investigator(s), subsequent Paclitaxel therapy following longer than allowed suspension of treatment may be allowed. The reasons for this decision shall be described in a case report form and all safety precautions should be observed.

#### 6.2.3.3 Re-treatment Criteria for Course 2 and thereafter

The second and consequent courses of therapy should be started after confirmation that the following criteria are all met prior to the drug administration.

- WBC count of  $3,000/\mu$ L or above, or ANC of  $1,500/\mu$ L or above.
- Platelet count of <u>75,000/µ</u>L or above.
- No Grade 2 or higher peripheral neuropathy and/or Grade 2 arthralgia/myalgia despite optimal medical therapy which, in the opinion of treating investigator(s), will make further Paclitaxel therapy unsafe.
- Any serious, clinically unmanageable by standard medical therapy (i.e. G-CSF for neutropenia, blood transfusion for anemia, etc.) adverse event(s), subjective/objective findings, abnormal laboratory values etc. occur that, in the opinion of the treating investigator(s), will make unsafe to continue further Paclitaxel therapy.
- No Grade 3 or higher non-hematological toxicity despite optimal medical therapy.

When any one of the criteria is not met, administration should not be started (a dose modification should be performed for a successive in-course repeated dosing. See Section 6.2.3 "Dose Modification"). Paclitaxel therapy should be started as soon as the laboratory test values and the symptoms are recovered to the acceptable level. However, if the re-treatment criteria are not met following 2 weeks after the scheduled initiation date of the given treatment course, the study therapy shall be discontinued in a given patient. When the initiation of the treatment course is delayed, the delayed initiation date shall be set as Day 1 of the given course with the subsequent treatment schedule adjusted accordingly.

However, in the given patient (i.e. in case of electrolytes abnormalities, etc.), if in the opinion of the treating investigator(s) it is still safe and in the best patient's interest to

continue Paclitaxel therapy (with dose adjustment, if clinically indicated), the treatment may continue but the reasons for this decision must be described in the case report form.

#### 6.2.4 Dose Modifications

Paclitaxel dose shall be reduced according to the severity of an adverse event using criteria listed below. Paclitaxel dose should be decreased by the increment of  $20 \text{mg/m}^2$ /dose. Patients who require a decrease below the total of  $60 \text{mg/m}^2$ /dose will be discontinued from treatment..

- WBC count: less than 1000/µL (\*1)
- Grade 3 neutropenia (neutrophils count  $<1000/\mu$ L but  $\ge 500//\mu$ L) or higher, neutropenia associated with fever ( $\ge 38^{\circ}$ C) or infection
- Grade 3 or higher non-hematological toxicity (\*2)
- Development of Grade 2 or higher peripheral neuropathy and/or Grade 2 arthralgia/myalgia despite optimal medical therapy which, in the opinion of treating investigator(s), will make further Paclitaxel therapy clinically difficult.
- When an investigator/sub-investigator judges to be clinically appropriate to skip a scheduled drug administration and/or to require a dose reduction.
- In the opinion of the treating investigator/sub-investigator there is a need for dose modification. Reasons for this decision should be described in a case report form.
- (\*1) Dose reduction based on the WBC count being less than  $1,000/\mu L$  shall depend on a decision of treating investigator/sub-investigator (taking into consideration the time of bone marrow recovery, clinical scenario for a given patient, etc.).
- (\*2): For the given patient, if in the opinion of the treating investigator/sub-investigator it is not clinically necessary to reduce the Paclitaxel dose (including Grade 3 or higher electrolyte abnormality, etc.) the dose may stay the same however, the reason for this decision must be described in a case report form.

# 6.2.5 Discontinuation of Therapy

Study therapy MUST be immediately discontinued for the following reasons:

- If the clinical efficacy evaluation reveals progressive disease (PD).
- Withdrawal of informed consent (subject's decision to withdraw for any reason).
- Any clinical adverse event, laboratory abnormality or intercurrent illness which, in the opinion of the investigator, indicates that continued treatment with study therapy is not in the best interest of the subject.

Paclitaxel CA139387 BMS-181339 Clinical Protocol

- Pregnancy.
- Termination of the study by BPKK.
- The compulsory detention for legal reasons or for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
- If a patient becomes ineligible after registration for the study.

Also, the study subject should be discontinued from the study therapy for the following reasons:

- A treatment delay of > 2-weeks because of paclitaxel related toxicity
- If in the opinion of the treating investigator(s) further continuation of Paclitaxel therapy is judged to be unsafe or clinically inappropriate based on the development of new or worsening of previous symptoms.
- If any clinical findings consistent with the Grade 1 or higher interstitial pneumonia, pneumonia, pulmonary fibrosis or severe infection develops.
- If there is a need for dose reduction below the total of  $60 \text{mg/m}^2/\text{dose}$  which violates the dose-reduction criteria.
- If an alternative systemic or local anti-cancer therapy is initiated.
- If the patient has moved away from the area during the study participation that makes the continuation of the study therapy no longer feasible.
- If the treating investigator/sub-investigator judges that the discontinuation of study therapy is in the best patient's interest..

For discontinuation of the study see Section 6.6.

#### 6.2.6 Treatment Compliance

Each study drug administration must be conducted under the supervision of an investigator/sub-investigator and the following data must be described in the case report form (CRF); date of paclitaxel administration, dosage, infusion time, body weight, and the pre-medications given.

#### 6.2.7 Other Guidance

Not applicable.

# 6.3 Blinding/Unblinding

Not applicable.

# 6.3.1 Blinding

Not applicable.

# 6.3.2 Unblinding

Not applicable.





# 6.5 Non-therapy Precautions and Restrictions

#### 6.5.1 Precautions

#### 1) Pre-medication drugs:

Based on the foreign literature, prolonged use of dexamethasone as pre-medication for the weekly Paclitaxel regimen appears is utilized. Compared with the dosing method for every 3 weeks Paclitaxel schedule, the total volume of steroids administered with the weekly regimen(s) appears to be fairly large. Therefore, it is considered highly likely that this may cause suppression of the adrenocortical function hence, lower doses of dexamethasone are permitted based on tolerance of the individual patient.

A clinical study reported by using decreasing doses of dexamethasone demonstrated that the dose of 20mg of dexamethasone (administered twice: 12 hours and 6 hours before Paclitaxel infusion) was gradually decreased to 2mg and only 1/22 patients developed skin rash but others tolerated Paclitaxel therapy well. Another report by revealed following results: 16mg of dexamethasone was administered as pre-medication to 43 patients. There was one patient with apnea that resolved without treatment but other 42 patients had no evidence of any hypersensitivity reaction.

Based on these reports, in the Japanese Phase I weekly Paclitaxel study, dexamethasone was initially administered at the 16mg dose, which was lower than the approved 20 mg dose, with subsequent decrease to a total of 2 mg. During this study dexamethasone dosing was further changed to the initial dose of 8 mg with subsequent dose decrease to a total of 1mg. With this last dexamethasone pre-medication regimen there were no hypersensitivity reaction observed.

Based on these data, the pre-medication regimen shall be used as described in the Section 6.2.2.1 (1).

- 2) Paclitaxel
- 2-1) Preparation and i.v. infusion time

Immediately prior to the infusion, Paclitaxel shall be mixed with 250 ml of a saline solution or 5% glucose solution and administered as a 1-hour IV infusion.

Containers for the solution MUST be made of glass, polyethylene or polypropylene. Paclitaxel is known to dissolve the container if it is made of polyvinyl chloride (PVC) and the plasticizer, DEHP[di-(2-ethylhexyl)phthalate], in the container may cause leaching.

#### 2-2) Injection kit

An injection kit made of PVC should NOT be used because of a possible leaching caused by plasticizer (DEHP). For the Paclitaxel injection, an in-line filter must be used.

#### 2-3) Other Caution Items

Paclitaxel is reconstituted with ethanol as a solvent. For any patient with alcoholic sensitivity, administration shall be made with full care. Upon administration, a patient's subjective and objective symptoms shall be carefully monitored and a patient should be carefully monitored during the time-points specified below;

- a) First-at 30 minutes following initiation of IV infusion for possible development of immediate allergy-like symptom or arrhythmia
- b) Subsequently- during and immediately after completion of IV infusion for possible hypotension.

For treatment of immediate allergy-like symptoms, arrhythmia or hypotension, refer to Appendix 9.





# 6.6 Withdrawal of Subjects from Study

Subjects MUST be discontinued from the study therapy AND withdrawn from the study participation for the reasons described in Section 6.2.5.

## 7 STUDY PROCEDURES AND OBSERVATIONS

## 7.1 Flow Chart/Time and Events Schedule

Clinical laboratory testing and monitoring during the study period shall be conducted at every appropriate time-point as detailed in Table 1. For those tests conducted after the final course of treatment on a previous please follow instructions shown in Table 1.

Any adverse event that does not recover to a baseline level by the 14<sup>th</sup> day of observation a follow-up shall be done, as much as possible, until the recovery to baseline or symptoms stabilization.

Table.7.1: X: required measurement point, XX: Conduct, if possible, at the time of clinic visit.

| | | | Rollover study (CA139387) | | | | | |
|---|---|---|---|---|---|---|---|---|
| Procedure | As needed after 2 <sup>nd</sup> course | | | 2nd- course | | | | |
| | Last | Observation | 1 <sup>st</sup> v | week (Day | 1) | Day8, | 7w | 1w |
| | dose | | Pre-dose <sup>a</sup> | Infusion | Post-<br>infusion | 15,22,<br>29,36 | Day43<br>(off) | Day1 |
| Patient background | | X | | | | | | |
| Body weight (BW),<br>Height, and BSA | | | X | | | | | X |
| Subjective/objective findings and P.S. | X | X | | X | | X | X | X |
| Blood Test (clinical laboratory) | X | X | X | | | X | X | X |
| Ca <sup>b</sup> | | | X | | | | | X <sup>b</sup> |
| Chest CT-scan <sup>c</sup> | Coı | nduct wh | en acute lur | ng disorde | r or interst | itial pneur | nonia wer | e suspected |
| Chest X-ray <sup>d</sup> | | | | Condu | ct if neces | sary | | |
| PaO <sub>2</sub> <sup>e</sup> | | | | Condu | ct if neces | sary | | |
| ECG <sup>f</sup> | | | | Condu | ct if neces | sary | | |
| Blood pressure <sup>g</sup> | | | X | | X | X | | X |
| Urine test h | | | X | | | | | X <sup>h</sup> |
| Pregnancy test <sup>i</sup> | | | X | | | | | XX |
| Observation of lesion for efficacy | | | C | onduct at l | east every | 7 weeks <sup>j</sup> | | |
| evaluation evaluation evaluation | | | | | | | | |

<sup>\*</sup> A day that a study drug is administered is Day 1.

<sup>\*</sup> Each laboratory test (except for tumor marker test) must be completed prior to administration of each weekly drug administration.

<sup>\*</sup> Administration of weekly Paclitaxel doses and initiation of successive treatment courses must be done within an expected date of treatment + one day.

Each required examination before the administration of a 1st course shall be conducted within 2 days before the first dose. Tumor status evaluation (tumor measurements, tumor markers) could be conducted within one month prior to the scheduled 1st Paclitaxel dose.

Once a course evaluation is required.

<sup>&</sup>lt;sup>c</sup> Conduct when acute lung disorder or interstitial pneumonia is suspected.

Can be done for evaluation of clinical symptoms such as fever, cough, shortness of breath or dyspnea. Can be repeated as clinically indicated.

e Conduct if clinically indicated i.e. if any respiratory symptoms such as cough or shortness of breath develops.

Done for patients with suspected cardiac-related toxicity. ECG monitoring during subsequent treatments shall be done when clinically indicated. with strong consideration given to safety of further Paclitaxel therapy.

- Frequent monitoring shall be performed. Patients should be closely monitored during and after the study drug infusion. Patients who will be going home following completion of Paclitaxel infusion (outpatient clinic practice) should be thoroughly evaluated for any side effects including vital signs and performance status.
- Should be done once prior to each treatment course. If the drug safety can be adequately judged from other evaluation(s) i.e. serum creatinine, etc., this test may not have to be done routinely.
- A pregnancy test shall be conducted within 72 hours prior to Day 1 of a 1st course for a WOCBP (WOCBP must have a negative serum or urine pregnancy test which has minimum sensitivity 25 IU/L or equivalent units of HCG). For successive treatment courses, it will be conducted prior to a Day 1 of each treatment course(as much as possible).
- To objectively evaluate the anti-tumor effect, an identical imaging diagnostic method shall be utilized for the individual patient. More than one diagnostic method could be applied, if clinically indicated. In addition, lesion(s) that can be evaluated only clinically i.e. skin or chest wall lesions, should be, as much as possible, photographed and lesion measurements should be documented.
- \* A day that a study drug is administered is Day 1.
- \* Each laboratory test (except for tumor marker test) must be completed prior to administration of each weekly drug administration.
- \* Administration of weekly Paclitaxel doses and initiation of successive treatment courses must be done within an expected date of treatment + one day.

# 7.2 Procedures by Visit

## 7.2.1 Screening evaluation

The following tests should be performed within 14 days prior to a first dose of study drug administration. If data (i.e. laboratory test values, etc.) from the time prior to obtaining the informed consent is used for study enrollment, the study subject shall agree to this herself/himself.

- Subjective/objective findings(including Performance Status-PS)
- Clinical efficacy from
- ECG (see Table 1)
- Blood test (Hb, WBC, ANC, Plt, T-Bil, AST(GOT), ALT(GPT), BUN, S-Cr, Ca)
- Serum or Urine pregnancy test: in case of WOCBP(minimum sensitivity 25IU/L or equivalent units of HCG)

## 7.2.2 Day 1 of the first therapy course (before infusion)

The following evaluation shall be conducted on Day1 of the 1<sup>st</sup> treatment course prior to a study drug administration;

• Body weight and height. Body Surface Area (BSA)

Paclitaxel CA139387 BMS-181339 Clinical Protocol

- Subjective/objective findings(including PS)
- Blood test and urine test (see Section 7.3.3 for details)
- Blood pressure (pre-dose and post- infusion)
- Serum or Urine pregnancy test: in case of WOCBP (minimum sensitivity 25IU/L or equivalent units of HCG within 72 hours prior to the start of study medication. However, if a pregnancy test is already conducted within 72 hours prior to the study drug administration during the enrollment period the repeated test is not needed.

# 7.2.3 Evaluations during each therapy course (on Days 8, 15, 22, 29, 36, 43 of each course)

The following items shall be examined;

- Subjective/objective findings (including PS)
- Blood test and urine test (see Section 7.3.3 for details)
- Blood pressure (pre-dose and post- infusion)

See Table 1 for details of evaluation on day 43 (7<sup>th</sup> week of each course of treatment)

# 7.2.4 Evaluations on Day 1 of Course 2 and thereafter (excluding the first course)

Following evaluation should be done on Day1 of the second therapy course and each subsequent treatment course(excluding the first course).

• Body weight, BSA.

Serum calcium and urine test shall be conducted at least once a course. When safety of further Paclitaxel therapy is adequately judged from i.e. serum creatinine values, etc., the urine test may not to be done routinely.

Tumor status evaluation should be done after completion of each treatment course (i.e. every 4~7 weeks or sooner, if clinically indicated)

• Measurements of lesion(s) for efficacy evaluation should be done using the same imagining method for each tumor status evaluation i.e. CT and/or MRI and/or bone scan etc. Lesions that can be evaluated only clinically i.e. skin and/or chest wall lesions should be photographed and measurement(s) of such lesions should be documented (as much as possible)

CA139387 Clinical Protocol

• Tumor marker (at least one type regardless of marker type)

## 7.2.5 Discharge evaluations

When the patient is discontinued from the study therapy (taken off the study) either due to a progressive disease or toxicity, or other (please see Section 6.2.5 for details), the following evaluation shall be done at the 14<sup>th</sup> day from the last dose (it may also be done on the 15<sup>th</sup> day or later, if necessary i.e. subject's personal matters or unexpected inconvenience at a study site,etc).

- Subjective/objective findings (including PS)
- Blood test, urine test (see Section 7.3.3)

#### 7.3 Details of Procedures

## 7.3.1 Study Materials

The Sponsor will provide the Paclitaxel(BMS-181339) Investigator Brochure, any relevant safety addendum, protocol and any amendments to the protocol, Case Report Forms(CRF), instructions for completing CRFs, case registration forms and Severe Adverse Reaction (SAE) forms etc.

#### 7.3.2 Safety Assessments

#### 7.3.2.1 Subjective/objective findings

It shall be conducted weekly on a day of the drug administration and, if possible, during the week when therapy is suspended (during the patient visit at the clinic or in the hospital). Instruct all patients to inform the investigator immediately if the patient develops fever, dry cough, shortness of breath for early detection and diagnosis of acute lung disorder or interstitial pneumonia. Investigator must evaluate carefully each study patient (i.e.auscultation, etc) even without clinical symptoms. Conduct chest CT-scan immediately, if clinically indicated, for proper diagnosis and treatment. Conduct A-aDO2 or DLCO, if necessary.

#### 7.3.2.2 Blood Pressure

It should be measured pre-dose and post-dose on every drug administrations. Frequent monitoring should be performed, fully observing the patients during and after the study drug IV infusion. If the patient is treated in the outpatient clinic settings, she/he should be thoroughly evaluated ( i.e. for any side effects, performance status, vital signs, etc) prior to discharge to home.

## 7.3.2.3 Chest X-ray and PaO2

Monitor carefully for the clinical symptoms such as fever, cough, shortness of breath or dyspnea, and if any of these symptoms develop, chest x-ray and/or PaO<sub>2</sub> may be conducted, if clinically indicated. If acute lung disorder or interstitial pneumonia is suspected, a chest CT-scan and, if necessary, additional A-aDO<sub>2</sub> or DL<sub>CO</sub> can be done (cf. 6.2.4 and Appendix 9). Consider consult with experts on respiratory diseases, if needed.

## 7.3.3 Laboratory Test Assessments

The following laboratory tests shall be conducted at the time of registration and prior to the scheduled Paclitaxel administration at each study site (corrected Ca test shall be conducted at least once a course);

- 1) Hematology
  - RBC count, hemoglobin, WBC count, neutrophil count, and platelet count.
- 2) Serum Chemistry
  - Total protein, albumin, total bilirubin, ALP, AST, ALT, LDH, BUN, S-Cr, Na, K, Cl and Ca.
- 3) Others
  - CRP (C-reactive protein)
  - The following tests will be done at least once for each course prior to Paclitaxel administration.
- 4) Urine test: urine protein, urine sugar, urobilinogen
  - The following obligatory evaluation should be done prior to the administration of a first drug dose on the first treatment course and subsequently, every  $\sim 7$  weeks.
- 5) Tumor marker
  - Appropriate type (at least one type regardless of marker type)
  - For WOCBP, a pregnancy test must be conducted within 72 hours prior to an initial study drug administration on a 1<sub>st</sub> course and prior to the1st dose on subsequent treatment courses (as much as possible).

Paclitaxel CA139387 BMS-181339 Clinical Protocol

6) Pregnancy test

Appropriate test (Serum or Urine pregnancy test [minimum sensitivity 25 IU/L or equivalent units of HCG]).

Results of all laboratory tests required by this protocol must be recorded on the laboratory pages of the CRF or by another method as agreed upon between the Investigator/Sub-investigator and this, too must be recorded in the CRF (see Section 9.8 Laboratory Test Abnormalities).

The following evaluation should be conducted if any respiratory symptoms such as cough or shortness of breath develop.

7) PaO<sub>2</sub>

7.3.4 Efficacy Assessments

7.3.4.1 Primary Efficacy Assessments

The primary efficacy endpoint will not be set in this study.

7.3.4.2 Secondary Efficacy Assessments

Not applicable.

8 INVESTIGATIONAL PRODUCT

Investigational product is defined as a pharmaceutical form of an active ingredient or placebo being tested or used as a reference in the study, whether blinded or unblinded.

8.1 Investigational Product Identification

The sponsor will provide Paclitaxel and pre-medication drugs as study drugs.

# Study Drug:

Code name: BMS-181339 Generic name: Paclitaxel

Dosage form/content: Each vial (16.7 mL) contains 100 mg of paclitaxel.

| CA13938 | 7 |
|------------------|----|
| Clinical Protoco | ol |

| Pac | ita | xel | |
|-----|-----|-----|-----|
| BM | S-1 | 81 | 339 |

| # Premedication | s: | | |
|---|---|---|---|
| Drug Name Formulation | | Contents | Packaging |
| Dexamethasone | vial | One vial (2 mL) contains 8 mg<br>dexamethasone sodium phosphate (6.6 mg<br>as dexamethasone) | 50 vials/box |
| Diphenhydramine | tablet | One tablet contains 10 mg diphenhydramine hydrochloride | 500 tablets/bottle |
| Ranitidine | ampule | One ampule contains 50 mg ranitidine | 10 ampules/box |

# 8.2 Packaging and Labeling

A label bearing the following information will be placed on the container or the package of the investigational product (see Appendix 3):

- The fact that the drug is for clinical study use
- Name of the investigational product (code name)
- Lot number
- Dosage form and content
- Storage condition
- Name and address of the sponsor
- Use date, if necessary

# 8.3 Handling and Dispensing of Investigational Product

After study contract between the sponsor and the medical institution is finalized, the sponsor will supply the investigational drug to the investigational product storage manager designated by the head of the medical institution. The investigational product storage manager will store and manage the investigational product appropriately, according to the written procedures prepared and provided by the sponsor, and follow up the status of dispensing by keeping the record of the investigational product management sheet.

Investigational product should be stored in a secure area according to local regulations. It is the responsibility of the Investigator to ensure that investigational product is only dispensed to study subjects. The investigational product must be dispensed only from official study sites by authorized personnel according to local regulations.

# 8.4 Investigational Product Records at Investigational Site(s)

It is the responsibility of the investigational product storage manager designated by the head of the medical institution to ensure that a current record of investigational product disposition is maintained at each study site where investigational product is inventoried and disposed. Records or logs must comply with applicable regulations and guidelines, and should include:

- Amount received and placed in storage area.
- Amount currently in storage area.
- Label ID number or batch number.
- Dates and initials of person responsible for each investigational product inventory entry/movement.
- Amount dispensed to and returned by each subject, including unique subject identifiers.
- Amount transferred to another area for dispensing or storage.
- Non-study disposition (e.g., lost, wasted, broken).
- Amount returned to Sponsor.

Sponsor will provide forms to facilitate inventory control if the staff at the investigational site does not have an established system that meets these requirements.

Sponsor should also provide procedures stipulating instructions for the handling, storage and management of investigational products and recording thereof.

# 8.5 Return and Destruction of Investigational Product

# 8.5.1 Return of Investigational Product

Upon completion or termination of the study, all unused and/or partially used investigational product must be returned to BMKK, if not authorized by BMKK to be destroyed at the site.

All investigational products returned to BMKK must be accompanied by the appropriate documentation and be clearly identified by protocol number and study site name. Empty containers should not be returned to BMKK. It is the responsibility of the medical institution to arrange for disposal of all empty containers, provided that procedures for proper disposal have been established according to applicable local
and institutional guidelines and procedures. The return of unused investigational product(s) should be arranged by the responsible Study Monitor.

Upon completion or termination of the study, all unused and/or partially used investigational product must be returned to BMKK, if not authorized by BMKK to be destroyed at the site.

All investigational products and empty containers returned to BMKK must be accompanied by the appropriate documentation and be clearly identified by protocol number and study site name. The return of unused investigational product(s) should be arranged by the responsible Study Monitor.

### 8.5.2 Destruction of Investigational Product

All unused investigational products must be returned to BMKK and therefore, the product can not be destroyed at the site without appropriate reasons. The investigational product storage manager must provide a detailed explanation to BMKK if the drug is destroyed at the site. BMKK will ensure appropriate destruction of investigational product.

# 8.6 Retained Samples for Bioavailability/Bioequivalence Studies

Not Applicable.

#### 9 ADVERSE EVENT REPORTING IN CLINICAL TRIALS

### 9.1 Importance of Adverse Event Reporting

Timely and complete reporting of safety information assists BMS/BMKK in identifying any untoward medical occurrence, thereby allowing: (1) protection of safety of study subjects; (2) a greater understanding of the overall safety profile of the investigational product; (3) recognition of dose-related investigational product toxicity; (4) appropriate modification of study protocols; (5) improvements in study design or procedures; and (6) adherence to worldwide regulatory requirements.

# 9.2 Collection of Safety Information

In BMS/BMKK clinical trials, an *Adverse Event (AE)* is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a patient or clinical investigation subject administered a medicinal product and which

does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal (investigational or marketed) product, whether or not considered related to the medicinal (investigational or marketed) product.

During clinical trials, adverse events can be spontaneously reported or elicited during open-ended questioning, examination, or evaluation of a subject. (In order to prevent reporting bias, patients should not be questioned regarding the specific occurrence of one or more adverse events.)

Following the subject's written consent to participate in the study, all serious AEs should be collected. The collection of non-serious AE information should begin at initiation of investigational product. Non-serious AE information should also be collected from the start of a placebo lead-in period or other observational period intended to establish a baseline status for the patient.

All identified AEs must be recorded and described on the appropriate Non-serious or Serious AE page of the CRF. If known, the diagnosis of the underlying illness or disorder should be recorded, rather than its individual symptoms. The following information should be captured for all AEs: date (and time) of onset and resolution, severity of the event (see definitions), investigator's opinion of the relationship to investigational product (see definitions), treatment required for the AE (see categories), cause of the event (if known), and information regarding resolution/outcome (see definitions).

Severity will be graded according to the... NCI-CTC

The following categories and definitions of severity should be used for AEs in this clinical trial:

- Mild (Grade I) Awareness of event but easily tolerated
- Moderate (Grade II) Discomfort enough to cause some interference with usual activity
- Severe (Grade III) Inability to carry out usual activity
- Very Severe (Grade IV) Debilitating, significantly incapacitates subject despite symptomatic therapy

The following categories and definitions of causal relationship to study drug should be used for all BMS/BMKK clinical trial AEs:

• Certain: There is a reasonable causal relationship between the study drug and the AE. The event responds to withdrawal of study drug (dechallenge), and recurs with rechallenge when clinically feasible.

- Probable: There is a reasonable causal relationship between the study drug and the AE. The event responds to dechallenge. Rechallenge is not required.
- Possible: There is reasonable causal relationship between the study drug and the AE. Dechallenge information is lacking or unclear.
- Not likely: There is a temporal relationship to study drug administration, but there is not a reasonable causal relationship between the study drug and the AE.
- Unrelated: There is not a temporal relationship to study drug administration (too early, or late, or study drug not taken), or there is a reasonable causal relationship between another drug, concurrent disease, or circumstance and the AE.

The adverse event will be regarded as related to study drug if the causal relationship is assessed as either "1. Certain ","2. Probable" or "3. Possible".

If a causal relation of an adverse event is assessed as "4. Not likely" or "5. Unrelated," reasons for the evaluation are to be described.

The following categories and definitions of outcome /resolution should be used for all BMS/BMKK clinical trial AEs

- 1) Did not resolve (Persisted or Aggravated)
- 2) Resolved (Recovered)
- 3) Resolved, but residual effects(s) persist (Relieved)
- 4) Unknown
- 5) Subject Died\*
- \* "Subject Died" category applies to reporting of Serious AEs only.

The following categories and definitions on action taken with respect to investigational product administration should be used for all BMS/BMKK clinical trial AEs

- 1) None
- 2) Dose reduced\*
- 3) Interrupted
- 4) Discontinued
- 5) Dose Increased\*

<sup>\* &</sup>quot;Dose reduced" and "dose increased" should be deleted if not applicable

The following categories on treatment required should be used for all BMS/BMKK clinical trial AEs

- 1) No
- 2) Yes (If Yes, comment on the treatment.)

A detailed explanation of the categories and definitions applicable to AEs due to laboratory abnormalities is provided in Appendix 5.

# 9.3 Adverse Events Related to Study Conditions

If the investigator believes that an SAE is not related to the investigational product, but is potentially related to the conditions of the study, (such as withdrawal of previous therapy, or complication of a diagnostic procedure), the relationship should be specified in the narrative section of the SAE page of the CRF.

#### 9.4 Overdose

An overdose is defined as the accidental or intentional ingestion of any dose of a product that is considered both excessive and medically important. For reporting purposes, BMS considers an overdose, regardless of adverse outcome, as an important medical event (see Serious Adverse Events).

### 9.5 AE Follow-up

AEs should be followed to resolution or stabilization, and reported as SAEs if they become serious. This also applies to subjects experiencing AEs that cause interruption or discontinuation of investigational product, or those experiencing AEs that are present at the end of their participation in the study; such subjects should receive post-treatment follow-up as appropriate. If an ongoing AE changes in its severity or in its perceived relationship to study drug, a new AE entry for the event should be completed.

# 9.6 Reporting of AE Information Following Study Completion

Collection of safety information following the end of investigational product administration is important in assisting in the identification of possible delayed toxicities or withdrawal effects. In BMS/BMKK trials, all SAEs must be collected which occur within 30 days of discontinuation of dosing or completion of the patient's participation in the study if the last scheduled visit occurs at a later time. In

addition, the investigator should notify BMS/BMKK of any SAE which may occur after this time period which they believe to be certainly, probably or possibly related to investigational product.

# 9.7 Handling of Serious Adverse Events (SAEs)

A *serious AE* is any untoward medical occurrence that at any dose:

- results in death,
- is life-threatening (defined as an event in which the subject or patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe),
- requires inpatient hospitalization or causes prolongation of existing hospitalization,
- results in persistent or significant disability/incapacity,
- is a cancer,
- is a congenital anomaly/birth defect,
- results in the development of drug dependency or drug abuse,
- is an important medical event (defined as a medical event(s) that may not be immediately life-threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the patient/subject or may require intervention (e.g., medical, surgical) to prevent one of the other serious outcomes listed in the definition above.) Examples of such events include, but are not limited to, intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization.) For reporting purposes, BMS/BMKK also considers the occurrences of pregnancy or overdose (regardless of adverse outcome) as events which must be reported as important medical events.

Adverse events classified as "serious" must be recorded on the SERIOUS AE (SAE) page of the CRF and require expeditious handling and reporting to BMKK as well as to the head of the medical institutions to comply with regulatory requirements.

All serious AEs whether related or unrelated to investigational product, must be immediately reported to BMKK as well as to the head of the medical institution (or designee) by confirmed facsimile transmission. A documented telephone call may be used in lieu of a facsimile. If only limited information is initially available, follow-up reports are required. The original BMKK SAE form must be kept on file at the sponsor. In selected circumstances, the protocol may specify conditions which require additional telephone reporting.

Cases of pregnancy must be reported on Pregnancy Surveillance Forms in lieu of SAE pages (see Section 9.10).

Collection of complete information concerning SAEs is extremely important. Thus, follow-up information which becomes available as the SAE evolves, as well as supporting documentation (e.g., hospital discharge summaries and autopsy reports), should be collected subsequently, if not available at the time of the initial report, and immediately sent using the same procedure as the initial SAE report.



As required, BMKK will notify Investigators and the heads of the medical institutions of all AEs that are serious, unexpected, and certainly, probably, or possibly related to the investigational product. This notification will be in the form of a Safety Update.

Upon receiving such notices, the Investigator must review and retain the notice with the Investigator Brochure. At the same time sponsor will immediately submit a copy of this information to the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) according to local regulations, via the head of the medical institution. The Investigator and IRB/IEC will determine if the informed consent requires revision. The Investigator should also comply with the IRB/IEC procedures

42

Date: 25-May-2005

for reporting any other safety information. Where required, submission of Safety Updates by the Investigator to Health Authorities, should be handled according to local regulations.

Serious adverse events whose causal relationship to the investigational product cannot be ruled out (adverse drug reactions) and that meet the criteria as specified in Article 273 of the Enforcement Regulations of the Pharmaceutical Affairs Law are to be reported on an expedited basis. The sponsor will report the adverse drug reactions to the regulatory authority. The time limit of reporting varies according to whether the reported adverse drug reactions are expected or unexpected.

- i. Unexpected "Death" or "cases which might result in death": within 7 days
- ii. Unexpected events other than those listed above: within 15 days
- iii. Expected "Death" or "Cases which might result in death": within 15 days

When necessary, the sponsor will consult with the medical expert on the actions to be taken regarding the conduct of the study, including whether this study is to be continued or not. Procedures for termination or suspension of this study are described in Section 10.7.



#### Reporting of Serious Adverse Events Seen in the Other Studies

When serious adverse events possibly related to the investigational product (adverse drug reactions) are reported in other studies, the sponsor will take the following actions.

For an unexpected serious adverse drug reaction, the sponsor will consult with the medical expert, if necessary, and the sponsor will notify Investigator and the head of the medical institution promptly. Any serious adverse drug reactions specified in Section 9.7 Serious Adverse events (SAEs) will be reported to the regulatory authority on an expedited basis within the specified time limits.

Periodically, according to the Investigator Brochure SOP, the Investigator Brochure will be updated to include new and relevant safety information. Until such time that

an AE becomes identified in the Investigator Brochure, it will continue to be reported to Investigators and to health authorities in line with local regulations.

### 9.8 Laboratory Test Abnormalities

All laboratory test values captured as part of the study should be recorded on the appropriate laboratory test results pages of the CRF, or be submitted electronically from a central lab. In addition, in order for BMKK to collect additional information about clinically important laboratory abnormalities, at a minimum, the following laboratory abnormalities should be captured on the non-serious or serious AE pages of the CRF as appropriate:

- Any laboratory test result that meets the criteria for a Serious Adverse Event
- Any laboratory abnormality that required the patient to have investigational product discontinued or interrupted
- Any laboratory abnormality that required the patient to receive specific corrective therapy.

It is expected that wherever possible, the clinical, rather than the laboratory term would be used by the reporting investigator (e.g., anemia versus low hemoglobin value).

A detailed definition of abnormal laboratory changes and outcome is provided in Appendix 5.

# 9.9 Other Safety Considerations

Any clinically significant changes noted during interim or final physical examinations, electrocardiograms, x-rays, and any other potential safety assessments, whether or not these procedures are required by the protocol, should also be recorded on the appropriate AE page of the CRF (i.e., NON-SERIOUS).

# 9.10 Pregnancy

Sexually active women of childbearing potential must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. (See Section 5.1 for definition of WOCBP).

Before enrolling women of childbearing potential (WOCBP) in this clinical trial, Investigators must review the guideline about study participation for WOCBP which can be found in the GCP Manual for Investigators. The topics include the following:

- General Information
- Informed Consent Form
- Pregnancy Prevention Information Sheet
- Drug Interactions with Hormonal Contraceptives
- Contraceptives in Current Use
- Guidelines for the Follow-up of a Reported Pregnancy

Prior to study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. The subject must sign an informed consent form documenting this discussion.

All WOCBP MUST have a **negative** pregnancy test within 72 hours **prior** to receiving investigational product. The minimum sensitivity of the pregnancy test must be 25 IU/L or equivalent units of HCG. If the pregnancy test is positive, the subject must not receive investigational product and must not be enrolled in the study.

Pregnancy testing must also be performed throughout the study as specified in Section 7.3.3 and the results of all pregnancy tests (positive or negative) recorded on the case report form.

# In addition, all WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation.

If following initiation of study treatment, it is subsequently discovered that a trial subject is pregnant or may have been pregnant at the time of investigational product exposure, including during at least 6 half-lives after product administration, the investigational product will be permanently discontinued in an appropriate manner (e.g., dose tapering if necessary for subject safety). Exceptions to investigational product discontinuation may be considered for life-threatening conditions only after consultation with the BMKK Medical Monitor or as otherwise specified in this protocol. The Investigator must immediately notify the BMKK Medical Monitor of this event and record the pregnancy on the Pregnancy Surveillance Form. Pregnancy Surveillance Forms are forwarded to BMKK as described in Section 9.7 (SAEs).

Protocol-required procedures for study discontinuation and follow-up must be performed on the subject unless contraindicated by pregnancy (e.g., x-ray studies). Other appropriate pregnancy follow-up procedures should be considered if indicated. In addition, the Investigator must report to BMKK, on the appropriate BMKK pregnancy surveillance forms(s), follow-up information regarding the course of the pregnancy, including perinatal and neonatal outcome. Infants should be followed for a minimum of eight weeks.

#### 10 ADMINISTRATIVE SECTION

## 10.1 Compliance with the Protocol and Protocol Revisions

The study shall be conducted as described in this approved protocol. All revisions to the protocol must be discussed with, and be prepared by, BMKK. The Investigator should not implement any deviation or change to the protocol without prior review and documented approval/favorable opinion from the IRB/IEC of an Amendment, except where necessary to eliminate an immediate hazard(s) to study subjects. Any significant deviation must be documented in the CRF or in the specific sheet provided to record these deviations.

If a deviation or change to a protocol is implemented to eliminate an immediate hazard(s) prior to obtaining IRB/IEC approval/favorable opinion, as soon as possible the deviation or change will be submitted to:

- IRB/IEC, via the head of the medical institution, for review and approval/favorable opinion;
- Bristol-Myers K.K.;
- The head of the medical institution;
- Regulatory Authority(ies), if required by local regulations.

Documentation of approval signed by the chairperson or designee of the IRB(s)/IEC(s) must be sent to BMKK.

If the revision is an Administrative Letter, the Sponsor must inform their IRB(s)/IEC(s) via the head of the medical institution.

If an Amendment substantially alters the study design or increases the potential risk to the subject: (1) the consent form must be revised and submitted to the IRB(s)/IEC(s) for review and approval/favorable opinion; (2) the revised form must be used to

obtain consent from subjects currently enrolled in the study if they are affected by the Amendment; and (3) the new form must be used to obtain consent from new subjects prior to enrollment.

#### 10.2 Informed Consent

Investigators must ensure that subjects are clearly and fully informed about the purpose, potential risks and other critical issues regarding clinical trials in which they volunteer to participate.

#### 10.2.1 Informed Consent Procedures

Preparation of the consent form is the responsibility of the Investigator and must include all elements required by ICH, GCP and applicable regulatory requirements, and must adhere to GCP and to the ethical principles that have their origin in the Declaration of Helsinki. The consent form must also include a statement that BMKK and regulatory authorities have direct access to subject records. Prior to the beginning of the study, the Investigator must have the IRB/IEC's written approval/favorable opinion of the written informed consent form and any other information to be provided to the subjects.

The Investigator must provide the subject with a copy of the consent form and written information about the study in the language in which the subject is most proficient. The language must be non-technical and easily understood. The Investigator should allow time necessary for subject to inquire about the details of the study, then informed consent must be signed and personally dated by the subject and by the person who conducted the informed consent discussion. The subject should receive a copy of the signed informed consent and any other written information provided to study subjects prior to subject's participation in the trial.

### 10.2.2 Subjects Unable to Give Informed Consent

#### 10.2.2.1 Miscellaneous Circumstances

Subjects who are compulsorily detained for legal reasons or treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

In circumstances where a subject's only access to treatment is through enrollment in a clinical trial, e.g., for subjects in developing countries with limited resources or for

subjects with no marketed treatment options, the investigator must take special care to explain the potential risks and benefits associated with the trial and ensure that the subject is giving informed consent.

When a subject may be in a dependent relationship with the investigator, a subinvestigator who is completely independent of the relationship between the subject and investigator should obtain the subject's informed consent.

#### 10.2.3 Illiterate Subjects

If the subject is unable to read, a reliable and independent witness should be present during the entire informed consent discussion. The choice of the witness must not breach the subject's rights to confidentiality. A reliable independent witness is defined as one not affiliated with the institution or engaged in the investigation. A family member or acquaintance are appropriate independent witnesses. After the subject orally consents and has signed, if capable, the witness should sign and personally date the consent form attesting that the information is accurate and that the subject has fully understood the content of the informed consent agreement and is giving true informed consent.

#### 10.2.4 Update of Informed Consent

The informed consent and any other information provided to subjects, should be revised whenever important new information becomes available that is relevant to the subject's consent, and should receive IRB/IEC approval/favorable opinion prior to use. The Investigator, or a person designated by the head of the medical institution, should fully inform the subject of all pertinent aspects of the study and of any new information relevant to the subject's willingness to continue participation in the study. This communication should be documented.

During a subject's participation in the trial, any updates to the consent form and any updates to the written information will be provided to the subject.

# 10.3 Monitoring for Protocol Compliance

Representatives of BMKK/BMS must be allowed to visit all study site locations periodically to assess the data, quality and study integrity. On site they will review study records and directly compare them with source documents and discuss the conduct of the study with the Investigator, and verify that the facilities remain acceptable.

In addition, the study may be evaluated by BMS/BMKK internal auditors and government inspectors who must be allowed access to CRFs, source documents and other study files. BMS/BMKK audit reports will be kept confidential.

THE HEAD OF THE MEDICAL INSTITUTION MUST NOTIFY BMKK PROMPTLY OF ANY INSPECTIONS SCHEDULED BY REGULATORY AUTHORITIES, AND PROMPTLY FORWARD COPIES OF INSPECTION REPORTS TO BMKK.

### 10.4 Records and Reports

An Investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the investigation on each individual treated with the investigational product or entered as a control in the investigation. Data reported on the CRF, that are derived from source documents, must be consistent with the source documents or the discrepancies must be explained.

The CRF must be completed legibly in ink. Subjects are to be identified by birth date and subject number, if applicable. All requested information must be entered on the CRF in the spaces provided. If an item is not available or is not applicable, it must be documented as such; do not leave a space blank.

The confidentiality of records that could identify subjects must be protected, respecting the privacy and confidentiality rules in accordance with the applicable regulatory requirement(s).

The Investigator will maintain a copy of the Signature Sheet to document signatures and seals of all persons authorized to make entries and/or corrections on CRFs. The original of this sheet will be kept by the sponsor. A correction must be made by striking through the incorrect entry with a single or double line and entering the correct information adjacent to the incorrect entry. The correction must be dated, signed or sealed and explained (if necessary) by the person making the correction and must not obscure the original entry.

The completed CRF must be promptly reviewed, signed or sealed, and dated by a qualified physician who is an Investigator or Subinvestigator. The Investigator must retain a copy of the CRFs including records of the changes and corrections.

# 10.5 Institutional Review Board/Independent Ethics Committee (IRB/IEC)

Before study initiation, the Sponsor must have written and dated approval/favorable opinion from the IRB/IEC, via the head of the medical institution, for the protocol, consent form, subject recruitment materials/process (e.g., advertisements), and any other written information to be provided to subjects. The Sponsor should also provide the IRB/IEC, via the head of the medical institution, with a copy of the Investigator Brochure or product labeling, information to be provided to subjects and any updates.

The Investigator and Sponsor should provide the IRB/IEC, via the head of the medical institution, with reports, updates, and other information (e.g., Safety Updates, Amendments, Administrative Letters) according to regulatory requirements or Institution procedures.

#### 10.6 Records Retention

The head of the medical institution must retain investigational product disposition records, copies of CRFs (or electronic files), and source documents for the maximum period required by applicable regulations and guidelines, or Institution procedures, or for the period specified by the Sponsor, whichever is longer. The head of the medical institution must contact BMKK prior to destroying any records associated with the study.

BMKK will notify the head of the medical institution when the trial records are no longer needed.

# 10.7 Study Completion, Termination and Suspension Study Completion

#### 10.7.1 Study Completion

When this study is completed, the investigator will notify the head of the medical institution in writing of the completion and provide a written overview of the study results.

The head of the medical institution will in turn notify the Sponsor and the IRB in writing of the completion and send a copy of the written overview of the study results.

#### 10.7.2 Termination or Suspension of an Entire Study

For an event that may require termination of this study, the sponsor will consult with the medical expert before deciding on the termination or suspension of this study. The sponsor will provide to the medical expert any relevant safety, efficacy or other available information that may justify the need for terminating or suspending the study. The termination or suspension of this study will be decided by the sponsor, taking in consideration the advice given by the medical expert.

When the termination of this study is decided, the sponsor will promptly notify the investigator and the head of the medical institution in writing of the decision and reasons for the termination.

# 10.7.3 Termination or Suspension of the Study at the Medical Institution

When the investigator considers it necessary to terminate or suspend this study, the investigator will promptly report the fact and reasons in writing to the head of the medical institution to which the investigator belongs.

The head of the medical institution will in turn promptly notify the Sponsor and the IRB in writing of the fact and explain in detail the events and rationale which required the termination or suspension of the study.

# 11 GLOSSARY OF TERMS AND LIST OF ABBREVIATIONS

# 11.1 Glossary of Terms

Not applicable.

# 11.2 List of Abbreviations

| Term | Definition |
|--------------------|----------------------------------------------------|
| d.i.v. | drip infusion in vein |
| 3w1q | 3 weeks administration, 1week quit |
| 6w1q | 6 weeks administration, 1 week quit |
| 6w2q | 6 weeks administration, 2week quit |
| °C | degrees centigrade |
| μL | microliters |
| μm | micrometers |
| A-aDO <sub>2</sub> | Alveolar to arterial oxygen gradient |
| ADM | doxorubicin |
| AE(s) | adverse event(s) |
| Alb | Albumin |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| (GOT) | (Glutamic Oxaloacetic Transaminase) |
| ANC | Absolute Neutrophil Count |
| AST | aspartate aminotransferase |
| (GPT) | (Glutamin Pyruvic Transaminase) |
| A-V | atrioventricular |
| BMKK | Bristol Myers K.K. |
| BRM | biological response modifiers |
| BUN | blood urea nitrogen |
| Ca | Calcium |
| CAP | cyclophosphamide, doxorubicin, cisplatin |
| CHF | congestive heart failure |
| Cl | Chloride |
| cm3 | centimeters cubed |
| CPA | cyclophosphamide |
| CR | complete response |
| CRF | case report form |
| CRP | C-reactive protein |
| CT | computed tomography |
| DL <sub>CO</sub> | Diffusing capacity of the lung for carbon monoxide |

| Term | Definition |
|------------------|------------------------------|
| DLT | dose-limiting toxicity |
| ECG | electrocardiogram |
| ER | estrogen receptor |
| GCP | Good Clinical Practice |
| Hb | Hemoglobin |
| IC50 | 50% inhibitory concentration |
| IEC | Independent Ethics Committee |
| IND | Investigational New Drug |
| IRB | Institutional Review Board |
| IV | intravenous |
| K | potassium |
| LDH | lactosedehydrogenase |
| mg/m2 | milligrams per square meter |
| mL | mililiters |
| MRI | magnetic resonance imaging |
| MTD | maximum tolerated dose |
| Na | sodium |
| NCI | National Cancer Institute |
| ng/mL | nanograms per milliliter |
| NSCLC | Non-small cell lung cancer |
| PaO <sub>2</sub> | Partial pressure oxygen |
| PD | progressive disease |
| PgR | Progesterone receptor |
| Plt | Platelet |
| PO, p.o. | orally |
| PR | partial response |
| PS | performance status |
| PVC | polyvinyl chloride |
| RBC | red blood cells |
| SAE(s) | serious adverse event(s) |
| S-Cr | Serum Creatinine |
| SD | stable disease |
| T-Bil | Total Bilirubin |
| TP | Total Protein |
| WBC | white blood cells |

53





#### APPENDIX 1 INFORMED CONSENT ELEMENT

The informed consent discussion and the written informed consent form and any other written information to be provided to subjects should include explanations of the following mandatory topics:

- 1 That the study involves research.
- 2 The purpose of the study.
- The expected duration of the subject's participation in the study.
- The study treatment(s) and the probability for random assignment to each treatment.
- 5 The study procedures to be followed, including all invasive procedures.
- 6 Those aspects of the study that are experimental.
- The reasonably foreseeable risks or inconveniences to the subject, and when applicable, to an embryo, fetus, or nursing infant.
- 8 The reasonably expected benefits. When there is no intended clinical benefit to the subject, the subject should be made aware of this.
- The alternative procedure(s) or course(s) of treatment that may be available to the subject, and their important potential benefits and risks.
- That records identifying the subject will be kept confidential and, to the extent permitted by the applicable laws and/or regulations, will not be made publicly available. If the results of the study are published, the subject's identity will remain confidential.
- That the BPKK/BMS monitor and/or BPKK/BMS representative, IRB/IEC, and regulatory authority(ies) will be granted direct access to the subject's original medical records for verification of clinical study procedures and/or data, without violating the confidentiality of the subject, to the extent permitted by the applicable laws and regulations and that, by signing and dating a written informed consent form, the subject or the subject's legally acceptable representative is authorizing such access.
- 12 The subject's responsibilities.

The compensation and/or treatment available to the subject in the event of study-related injury.

- The anticipated prorated payment, if any, to the subject for participating in the study.
- The person(s) to contact for further information regarding the study and the rights of study subject's, and whom to contact in the event of study-related injury.
- That the subject's participation in the trial is voluntary and that the subject may refuse to participate or withdraw from the study, at any time, without penalty or loss of benefits to which the subject is otherwise entitled.
- The foreseeable circumstances and/or reasons under which the subject's participation in the study may be terminated.
- The anticipated expenses, if any, to the subject for participating in the study.
- The consequences of a subject's decision to withdraw from the research and procedures for orderly termination of participation by the subject.
- That the subject or the subject's legally acceptable representative will be informed in a timely manner if information becomes available that may be relevant to the subject's willingness to continue participation in the study.
- 21 The approximate number of subjects involved in the study.
- The name, title and address of the Investigator or the subinvestigator to contact.

Additional mandatory topics for inclusion in the informed consent of studies enrolling Women of Child Bearing Potential (WOCBP):

#### 1 General Statement

The subject must not be, and should not become pregnant during exposure to the investigational product. Subjects should be instructed to contact the Investigator if they plan to change their pregnancy avoidance method or if they need to take any prescription drug or other medication not prescribed by Investigator. Sexually active subjects must use an effective method of pregnancy avoidance during the course of the study, in a manner such that risk of failure is minimized. The informed consent must indicate that information on pregnancy prevention for women of child-bearing potential has been reviewed with the subject by the Investigator or study designee.

#### 2 Laboratory & Animal Reproductive Toxicology

A statement addressing what is known about the investigational product from laboratory and animal reproductive toxicity studies concerning possible mutagenic and/or teratogenic effects should be included in the consent. The consent should indicate that this information has limited predictive value for humans.

#### 3 Unforeseeable Risks

The consent must indicate that exposure to the investigational product may involve currently unforeseeable risks to the subject (or embryo or fetus, if the subject is or may become pregnant).

#### 4 Occurrence of Pregnancy or Suspected Pregnancy

The informed consent must include study contact name(s) and telephone number(s) for the subject to call if she becomes pregnant or suspects pregnancy, has missed her period or it is late, or she has a change in her usual menstrual cycle (e.g., heavier bleeding during her period or bleeding between periods).

#### 5 Discontinuation from the Study

Any subject who becomes pregnant during the course of the study will be immediately withdrawn (unless allowed or stated differently in the protocol) and referred for obstetrical care. All financial aspects of obstetrical, child or related care are the responsibility of the subject.

#### 6 Pregnancy Follow-up

If a subject becomes pregnant, BMS will seek access to the subject's and/or infant's clinic/hospital records through the pregnancy, and for a minimum of 8 weeks following delivery.

#### 7 Use of a Study-prohibited Contraceptive Method

When applicable, the informed consent should clearly indicate if a contraceptive method is prohibited (e.g., when hormonal contraceptive interaction with the investigational product(s) is known or suspected). In this situation, a study participant should be instructed to notify the Investigator or study designee if a prohibited contraceptive method is initiated during the course of the study so that additional precautions can be taken or the subject discontinued from the study.

#### 8 Non-investigational product Interactions with Hormonal Contraceptives

Women using a hormonal method of contraception (oral contraceptives, implantable or injectable agents) must be instructed to notify the Investigator or study designee of the need to take any prescription drug or other medication not prescribed by the Investigator. The purpose of this statement is to identify any potential non-investigational product interaction with the contraceptive which might reduce the effectiveness of the contraceptive method.





62

#### **APPENDIX 4 ROLES AND RESPONSIBILITIES OF STUDY** RELATED PERSONNEL AND STUDY PERIOD

CA139387

The study system is described below.

#### 4.1 **SPONSOR**

#### 4.1.1 **Sponsor**



#### 4.1.2 **Study Director**

Taku Seriu, M.D., Director



#### 4.1.3 **Medical Expert and Roles Thereof**



#### **Roles**

The medical expert will, as occasion demands, advise about the following matters etc. from a medical point of view:

- Examination of the Protocol
- Preparation for and participation, if necessary, at KIKO Consultations
- Examination of the Case Report Form (CRF)
- Examination of the informed consent form and explanatory document
- Examination of investigator's brochure
- Examination of handling for adverse events (AEs) and safety information
- Examination of continuation, change, termination and suspension of the study
- Review of the clinical study report

Date: 25-May-2005 63



# 4.2 PK/PD ANALYST

Not applicable.

Date: 25-May-2005

64

#### 4.3 COORDINATING INVESTIGATOR AND ROLES THEREOF



### [Roles]

- Coordinate the details of the protocol between the study sites.
- Coordinate troubles on interpretations of the protocol occurring during the study.
- Opinion co-adjustment between the study coordinating investigators and investigators at Evaluation Committee Meeting and other occasions.
- Advise about the preparation and revision of the protocol and others.

#### 4.4 COORDINATION COMMITTEE AND ROLES THEREOF

Not applicable

### 4.5 EFFICACY AND SAFETY COMMISSIONER

#### [Roles]

- 1) The efficacy/safety evaluation commissioner shall evaluate the progress of the study, safety information and others, when appropriate, and advise the sponsor about continuation, change and termination or suspension of the study. The efficacy/safety evaluation committee consists of members independent of the sponsor and the investigator.
- 2) At the request of the sponsor, the efficacy/safety evaluation committee shall conduct the following tasks;
- The committee shall advise the sponsor about the appropriateness of study plan concerning safety assurance and others. The committee shall examine whether the protocol is to be revised or not and, if required, advise the sponsor about the revision.
- When a serious adverse event possibly affecting the conduct of the entire study is reported by the sponsor (see 8.2), the committee shall hold a meeting (or handed-round decision-making system\*) and advise about continuation of the study, changes of the study plan and termination or suspension of the study.

• Each committee member shall review the minutes of the meeting (if a handed-round decision-making system is used, replies from each committee member are handled as the minutes) and affix his or her signature or seal.

Supplemental information on the handed-round decision-making system. The chairman shall decide whether handed-round decision-making is to be required or not. When it is considered necessary to use a handed-round decision-making system from the standpoint of the items of discussion or because of expedited nature of discussion, the chairman shall ask each member to deliberate the matters in writing, and each member shall report the results of deliberation to the chairman in writing. The sponsor shall receive the report of each member from the chairman and retain the report as the minutes of the committee meeting.

#### 4.6 INVESTIGATORS

Refer to an Attachment, "List of Clinical Trial Sites and Investigators"

### 4.7 ASSIGNMENT MANAGER AND ROLES THEREOF

Not applicable.

#### 4. 8 STUDY PERIOD

June/2005- Approval

# APPENDIX 5 DEFINITION OF ABNORMAL CHANGES AND OUTCOME OF LABORATORY TESTS

Laboratory values will be monitored, and their significance will be evaluated by the investigator/subinvestigator taking in consideration how they evolve throughout the study. Any abnormal change observed, per the definition below, shall be recorded in the appropriate form as an "Adverse Event", together with its severity, actions taken and causal relationship to study drug, to be evaluated as described Section 9 in this protocol For details on the follow-up of AEs please refer to Section 9 in this protocol.

On laboratory test values: The abnormal values shall be evaluated according to the NCI Common Toxicity Criteria (NCI-CTC) ver.2.0 (Translated version into Japanese

by the JCOG will also be available in Appendix 10). For the item that is not listed in the NCI-CTC, a normal value at each study site shall be applied).

#### 1) Definition of abnormal changes

For laboratory test parameters, an "abnormal value" is defined as a value deviated from the normal range specified at the medical institution. When a laboratory value is initially "normal" and becomes "abnormal" during the treatment period or is initially "abnormal" and further "aggravates," such a change in laboratory values, if it is clinically significant (adverse event), is considered to be an "abnormal change."

If the investigator/subinvestigator did not assess such a change in laboratory values as an "abnormal change," the investigator/subinvestigator must provide details of and reasons for the assessment in column "Comment" on the laboratory pages of the CRF.

#### 2) Outcome

The outcome of an abnormal change will be recorded according to the following criteria:

- 1) Did not resolve: The value remained outside the normal range and continued to be clinically significant (or worsened with a consequent increase in severity)
- 2) Resolved: The value was reversed to the pretreatment level or returned to a normal range
- 3) Resolved, but residual effect(s) persist: The value was not reversed to a normal range but improved to a clinically insignificant level
- 4) Unknown: Use of an alternative therapeutic method or failure of following-up (the reasons should be described)

# APPENDIX 6 DIRECT ACCESS TO SOURCE DOCUMENTS AND DEFINITION THEREOF

The head of the medical institution and the investigator must permit monitoring and auditing to be performed by the sponsor, reviews by the IRB, and inspection by the regulatory authorities. Direct access to all the study-related records such as source documents should be provided upon request by the monitors and the auditors of the sponsor, the IRB, or the regulatory authorities. In this particular study, source documents, and the CRF data deemed as source data are defined as follows:

#### 1) Source documents

- Subject identification code sheet
- Medical records
- Written consent
- Study drug management sheet
- Laboratory examination data
- Electrocardiography (ECG) charts
- Image that can identify the lesion (MRI, CT, etc.).

#### 2) CRF data deemed as source data

Of the data directly recorded in the CRFs, the following data are deemed as source data: various comments described in the CRFs, study drug relation to abnormal laboratory test finding, comments of adverse events (event, severity, date of onset, actions taken regarding study drug, treatment required for event, outcome, causal relationship to study drug, comments), comments of discontinuation or drop-outs due to any safety problem, comments of protocol compliance status). The data directly described in the margin area of CRF, they are also deemed as source data.

#### APPENDIX 7 CRITERIA FOR RESPONSE

# 7.1 Evaluation Criteria on Therapeutic Effects in Patients with Advanced or Recurrent Breast Cancer(Extracts)

CA139387

Clinical Protocol

#### 7.1.1 Measurement of a Lesion

- 1-1 Tumor lesion sites are divided into 13, as shown in Table 1, and individually measured site-by-site. These lesions include the 3 categories; 1) bi-directional measurable lesions, 2) one-directional measurable lesions and 3) immeasurable (evaluable) lesions. However, if two or more categories of lesions co-exist in one identical lesion site, these lesions shall independently be measured for records. The measurement shall in principle be made every 4 weeks.
- 1-2 A bi-directional lesion represents a product multiplying the largest diameter by its vertical counterpart diameter. (cm2) If a plural number of lesions exist in one identical lesion site, a product for each lesion must separately be figured out. In case only one directional measurement could be available in a front view image by X-ray, etc., a measured value of lateral view that is assumed to be vertical to the front view could be allowable for use.
- 1-3 One directional lesion measurement must always be done on one identical site. (cm) If a plural number of lesions exist in one identical lesion site, a product for each lesion must separately be figured out.
- 1-4 In an immeasurable (evaluable) lesion, an evaluation must be made as much as possible on a dose-response reaction using various parameters (radiography, diagnostic imaging methods and other useful means to trace the post-dose progresses) before and during the therapeutic period.
- 1-5 An efficacy evaluation on radiotherapy shall be applied only to the limited area of irradiated lesion.

#### 7.1.2 Definition of Objective Effects

- 2-1 CR(Complete Response): A disappearance of all tumor lesions confirmed lasts at lest 4 weeks or longer.
  - 2-1-1 For each skeletal (osseous) lesion, a definition shall be made as follows;
    - 1) In osteolytic lesions prior to this study drug therapy, it shall be defined as a fluoroscopically completely hardened or a recovered back-to-normal.
    - 2) In osteogenic lesions prior to this study drug therapy, it shall be defined as a fluoroscopically significant decrease in concentration level.
      - Note 1:Bone scintigraphy findings could be available for use as an auxiliary tool for diagnostics.

Note 2:For the spinal bones, a diagnosis by CT or MRI is better.

- 2-2 Partial Response(PR): defined as a decrease by 50% or more in a total product of measurable lesions. In an immeasurable (evaluable) lesion, defined as a clear improvement. As for any bone metastasis, defined as a calcification of bone-soluble lesion or a decrease in concentration of an osteogenic lesion. These phenomena must last at least 4 weeks or longer. During the course, either one of the lesions (secondary lesions included) shall not be increased by 25% or more and not bear any new lesion.
- 2-3 No Change (NC): defined as a decrease by 50% or less or as an increase by 25% or more in a total product of measurable lesions. In immeasurable (evaluable) and secondary lesions, neither clear improvement nor clear increase is shown and no new lesion appears in either case. These phenomena must last at least 4 weeks or longer, and for a bone lesion 8 weeks or more.
- 2-4 Progressive Disease(PD): defined as an increase by 25% or more in a total product of measurable lesions; a significant increase of measurable (evaluable) and secondary lesions, or a development of new lesion. However, in case of bone metastasis, a pathological fracture or necrosis (or weakness) will not always be interpreted as an evidence for progressive disease.
- 2-4-1 Though an improvement seen in some lesions and a total product of lesions reveals a shrinkage, if any one of the lesions that shows an increase by 25% or more at the time of the most shrunken compared with the baseline value, it shall be defined as PD. However, even if any one of the lesions that shows an increase by 25% or more at the time of the most shrinkage compared with the baseline value in patients with PR, it shall be interpreted as PR as long as thr shrinkage rate stays at 50% or lower compared with the baseline values. (Actual cases seen below)

O A

CR period

CR period

D

Trerapeutic Period

Figure 1. the case of CR

A: Day of study therapy initiation B: Day that CR is first confirmed C: Day that CR is last confirmed

D: Day that PD is confirmed

B-C: CR period

Note: Though Point D shows a shrinkage of 50% or more, compared with Point A, but since it shows 25% or more increase in the value at start of study therapy compared with Point C, it shall be interpreted as PD.

Figure 2. the case of PR



A: Day of study therapy initiation
B: Day that PR is first confirmed
C: Day that PR is last confirmed
D: Day that PD is confirmed

B-C: PR period

Note: Points C & D show 25% or more increase in the value at start of study therapy compared with Point B. However, since Point C shows 50% or more in shrinkage compared with Point A, it will be PR; in the same manner, Point D 50% or less in shrinkage compared with Point D, be interpreted as PD.

Figure 3. the case of NC



- A: Day of study therapy initiation
- B: Day that the most tumor shrinkage is first confirmed
- C: Day that NC is last confirmed
- D: Day that PD is confirmed
- A-C: NC period

Note: Point D shows an increase of 25% or less compared with Point A, but

it shows 25% or more increase in baseline values compared with Point B, be interpreted as PD.

- Note 1: CR: Complete Response(Complete or significant response), PR: Partial Response(partial or responsed), NC: No Change (Not any changed), PD: Progressive Disease
- Note 2: A total product of lesions means a total product of the largest diameter and its vertical largest diameter multiplied (cm2) for bi-directional lesions and a product of measured values for one-directional lesions in plural number of lesions of one identical site.
- Note 3: When a progressive disease stays as NC for long (24 weeks or longer) by the study drug therapy, it will be recorded separately as long NC in efficacy. However, it will not be added to "9. Calculation of Response Rate".
- Note 4: Cases that a decrease of 50% or more in a total product of measurable lesions lasts for 4 weeks or less and those that a decrease of 25% or more to 50% or less lasts for 4 weeks or longer could be recorded separately as

MR(Minor Response). However, it will not be added to "9. Calculation of Response Rate"

- Note 5: Upon evaluating the effects in a therapeutic plan that a minimum dosage or a minimum dosing period is specified, it requires a regulated observation period of 4 weeks or more and that of 8 weeks or more for bone lesions. However, for a clarified PD, it will not be applied.
- Note 6: Evaluations for radiotherapy, they will be recorded immediately after, 4 weeks and 12 weeks after radiotherapy.
- Note 7: For successively planned surgery, etc., an evaluation of objective effects in case of not enough observation period given after study therapy(topical arterial injection therapy, etc.) could well be made by only changes of concerned lesions according to the specifications, regardless of duration. However, it must be described separately to other treatment methods.
| | Table 1: Total Evaluation of Objective Effects for Lesions | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Ca | te- | Sites | Disease Type | bi-directionally<br>measurable | | one-directionally measurable | | immea- | Total |
| go | ry | Sites | Disease Type | measured values | Judg-<br>ments | measured values | Judg-<br>ments | surable | Evaluation |
| | | Primary breast | a. tumor | | | | | | |
| | 1 | and opposite side of breast | b. diffuse infiltration | | | | | | |
| <b>S</b> | | D 1/G1: ) | a. node | | | | | | |
| oft | 2 | Dermal(Skin) and | b. disperse | | | | | | |
| Soft tissues | _ | Subcutaneous | c. diffuse infiltration | | | | | | |
| ues | | | d. distal | | | | | | |
| | 3 | lymphatic<br>node | a. topical/local | | | | | | |
| | 3 | | b. distal | | | | | | |
| | 4 | mediastinal hila | ar tumor | | | | | | |
| bone | 5 | bone | a. bone | | | | | | |
| ne | 3 | bone | b. bone marrow | | | | | | |
| | | | a. node type | | | | | | |
| | 6 | lung | b. disperse type | | | | | | |
| | | | c. funicular type | | | | | | |
| | 7 | pleura | a. node/thickness | | | | | | |
| V <sub>10</sub> | | • | b. pleural effusion | | | | | | |
| Viscera | 8 | pericardial hun | nor | | | | | | |
| а | 9 | hepatic | tic | | | | | | |
| | 10 intra-abdominal | | l tumor | | | | | | |
| | 11 | ascites | | | | | | | |
| | central nervous system(CNS, brain, eyes, etc.) | | | | | | | | |
| | 13 | Others ( | ) | | | | | | |

Note 1:Topical area for skin and subcutaneous tissue means an anterior ipsilateral thorax and others distal.

- Note 2:A topical/local area of lymphatic node includes ipsilateral axilla, supra- and sub-clavicular and parasternal, and others distal.
- Note 3:For pleural effusion, pericardial humor and ascites, it requires to be sytologically diagnosed as positive. A cytological negativity without use of diuretics and complete disappearance of lesion with no humoral retention; this is the only one case for PR.
- Note 4:For hepatic and cerebral tests, lesions must be identified by angiography, scintigraphy, echography and CT, etc. Measurement for hepatic hypertrophy shall be made vertically from the costal end in identical site.

Note 5:See Text 2-1,2 and 4.

Paclitaxel CA139387 BMS-181339 Clinical Protocol

Note 6:No CR evaluation will be made in these lesions.

# 7.2 Response Evaluation Criteria in Solid Tumors (RECIST; Outlines)

#### 7.2.1 Measurability of Tumor Lesions at Baseline

At baseline, tumor lesions will be categorized as:

measurable lesions: lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as 20 mm with conventional techniques or as 10 mm with spiral CT scan.

non- measurable lesions: all other lesions, including small lesions (longest diameter 20 mm with conventional techniques or 10 mm with spiral CT scan) and truly non-measurable lesions.

All measurements should be recorded in metric notation, using a ruler or calipers.

All baseline evaluations should be performed as close as possible to the treatment start and never more than 4 weeks before the beginning of the treatment.

Lesions that are considered as truly non-measurable include the following:

- bone lesions;
- leptomeningeal disease;
- ascites;
- pleural/pericardial effusion;
- inflammatory breast disease;
- lymphangitis cutis/pulmonis;
- abdominal masses that are not confirmed and followed by imaging techniques;
- cystic lesions;

Paclitaxel CA139387 BMS-181339 Clinical Protocol

#### 7.2.2 Tumor response evaluation

## 7.2.2.1 Baseline Documentation of "Target" and "Non-Target" Lesions

All measurable lesions up to a maximum of 10 lesions representative of all involved organs should be identified as target lesions and will be recorded and measured at baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repetitive measurements (either by imaging techniques or clinically). A sum of the longest diameter (LD) for all target lesions will be calculated and reported as the baseline sum LD. The baseline sum LD will be used as reference to further characterize the objective tumor response of the measurable dimension of the disease.

All other lesions (or sites of disease) should be identified as non-target lesions and should also be recorded at baseline. Measurements are not required and these lesions should be followed as "Present" or "Absent".

#### 7.2.2.2 Response Criteria

#### 7.2.2.2.1 Evaluation of Target Lesions

Complete Response CR disappearance of all target lesions.

Partial response PR at least a 30% decrease in the sum of LD of target

lesions taking as reference the baseline sum LD.

Progression PD at least a 20% increase in the sum of LD of target

lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of

one and more new lesions.

Stable Disease SD neither sufficient shrinkage to qualify for PR nor

sufficient increase to qualify for PD taking as references

the smallest sum LD since the treatment started.

#### 7.2.2.2.2 Evaluation of non target lesions

Complete Response CR disappearance of all non-target lesions and

normalization of tumor marker level.

Non-Complete Response CR/

| Paclitaxel | CA139387 |
|------------|-------------------|
| BMS-181339 | Clinical Protocol |

| Non-Progression(non-PD): | rogression(non-PD): persistence of one | | | | | |
|---|---|---|---|---|---|---|
| | or/and | maintenance | of | tumor | marker | level |
| | above the normal limits. | | | | | |

Progression PD appearance of one and more new lesions.

Unequivocal progression of existing non-target lesions.

#### 7.2.2.2.3 Evaluation of best overall response

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence. The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria (see Section 9.2.3)

| Target lesions | Non-Target lesions | New Lesions | Overall response |
|----------------|--------------------|-------------|------------------|
| CR | CR | No | CR |
| CR | Non-CR/Non-PD | No | PR |
| PR | Non-PD | No | PR |
| SD | Non-PD | No | SD |
| PD | Any | Yes or N | lo PD |
| Any | PD | Yes or N | lo PD |
| Any | Any | Yes | PD |

#### 7.2.3 Confirmation Criteria

To be assigned a status of PR or CR, the size changes in tumor measurements must be confirmed by repeat studies that should be performed no less than 4 weeks after the criteria for response are first met.

In the case of SD, the follow-up measurements conducted at least 6 weeks and longer after registration must have met the SD criteria at least once.

### **APPENDIX 8 PERFORMANCE STATUS**

CLASSIFICATION OF PERFORMANCE STATUS (GENERAL CONDITIONS) SPECIFIED BY THE EASTERN COOPERATIVE ONCOLOGY GROUP

| Grade | Performance Status |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of walking hours |
| 3 | Capable of only limited selfcare, confined to bed or chair more than 50% of walking hours |
| 4 | Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair |

# APPENDIX 9 THERAPEUTIC ACTIONS FOR ACUTE ALLERGIC SYMPTOMS, ARRHYTHMIA, HYPOTENSION OR INTERSTITIAL PNEUMONIA

Careful monitoring should be made, especially during the first 30 minutes after initiation of infusion when hypersensitivity reactions (immediate type allergy-like symptoms) or arrhythmia possibly appear, during, and after, the infusion when hypotension may appear.

#### [Hypersensitivity Reactions (Immediate type Allergy-like Symptoms)]

In the U.S. clinical studies, the reported hypersensitivity reactions (immediate type allergy-like symptoms) attributed to paclitaxel administration included dyspnea, bronchospasm, decreased blood pressure, increased blood pressure, angioedema (laryngeal stridor, epiglottic swelling, periorbital edema, etc.), urticaria, flushing, erythematous rash, abdominal pain, pain of extremities, vomiting, fever, and rigidity.

In the event of clear evidence of hypersensitivity reaction (immediate type allergy-like reactions), paclitaxel should immediately be discontinued, and the following actions should be taken while close cardiopulmonary monitoring:

- 1) Diphenhydramine-calcium bromide (5 ml; containing 20 mg of diphenhydramine) should be intravenously administered (the dose should be adjusted appropriately according to the patient<sup>TM</sup>s status).
- 2) Epinephrine (not greater than 0.25 mg) should be diluted with saline or other solvents and administered intravenously as slowly as possible. This course should be repeated at 5- to 15-minute intervals at its need (alternatives are dobutamine and dopamine preparations).
  - a) Hypotension not responding to epinephrine: Central venous pressure and other cardiovascular parameters should be monitored, and intravenous fluid should be given, if necessary.
  - b) Stridor not responding to epinephrine: bronchodilators such as salbutamol sulfate (1.5 2.5 mg of salbutamol or equivalent doses of other drugs) should be given by inhalation, using a nebulizer.
- 3) It is known that corticosteroids are effective in blocking allergic reactions of delayed type due to various antigens. Sodium methylprednisolone succinate

125 mg may be administered intravenously for prevention of recurrence or allergic symptoms.

#### [Arrhythmia]

The following therapeutic actions may be taken for arrhythmia:

- 1) Asymptomatic bradycardia: paclitaxel may be continued.
- 2) Symptomatic bradycardia: paclitaxel should be discontinued.
- 3) Marked sinus bradycardia: paclitaxel should be discontinued, and atropine should be administered intravenously at 5-minute intervals (0.5 mg per administration) until the total dose reaches 2.0 mg.
- 4) Atrioventricular block: paclitaxel should be discontinued. Class I block and block of Mobitz Type I will usually disappear spontaneously. Atropine produces transient improvement of atrioventricular conduction. For severe bradycardia and others (block of Mobitz Type II or complete atrioventricular block), pacing therapy should be used.
- 5) Marked ventricular ectopy (PVC, non-sustained VT, etc.) and marked tachycardia: paclitaxel should be discontinued, and lidocaine should be used. Intravenous lidocaine therapy should be started with 1 2 mg/kg/min and, if effective, followed by drip infusion of 1 2 mg/min.

#### [Hypotension]

The following therapeutic actions may be taken for hypotension:

- 1) Mild: Fluid therapy should be used, if necessary, for keeping blood pressure.
- 2) Moderate or severe: Persistent intravenous infusion of dopamine should immediately be started. Doses (5 15 ∝g/kg/min) should be adjusted according to the severity. The infusion should be continued until blood pressure is stabilized. If necessary, norepinephrine should be administered. After confirming that blood pressure remains stable, the dose of dopamine should be reduced, or the use of this drug should be discontinued.

#### [Interstitial pneumonia]

The following therapeutic measures may be taken for interstitial pneumonia diagnosed with clinical symptoms and diagnostic imaging after failure of antibiotics treatment:

It is reported that following treatment is effective: Discontinue the drug therapy, and apply corticosteroid pulse therapy (methylprednisolone 1000mg in 5% glucose solution or saline solution 200mL for intravenous over 1-hour for consecutive three days (1 course). Repeat 3 courses at maximum with an interval of 1 to 2 week. Following prednisolon 40-60 mg/day p.o. with dose reduction every 1 to 2 weeks).

Consult with doctors who are expert in respiratory disease in time of need.

Date: 25-May-2005

# APPENDIX 10 NATIONAL CANCER INSTITUTE CTC VERSION 2

PDF file can be found at

## **COMMON TOXICITY CRITERIA (CTC)**

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| | | ALLERGY/IM | <b>IMUNOLOGY</b> | | |
| Allergic reaction/<br>hypersensitivity<br>(including drug fever) | none | transient rash, drug<br>fever <38°C (<100.4°F) | urticaria, drug fever<br>≥38°C (≥100.4°F),<br>and/or asymptomatic<br>bronchospasm | symptomatic<br>bronchospasm,<br>requiring parenteral<br>medication(s), with or<br>without urticaria;<br>allergy-related<br>edema/angioedema | anaphylaxis |
| Note: Isolated urticaria, in the Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) | none | nanifestations of an allergic or hy<br>mild, not requiring<br>treatment | persensitivity reaction, is gr<br>moderate, requiring<br>treatment | raded in the DERMATOLO | GY/SKIN category. |
| Autoimmune reaction | none | serologic or other<br>evidence of<br>autoimmune reaction<br>but patient is<br>asymptomatic (e.g.,<br>vitiligo), all organ<br>function is normal and<br>no treatment is required | evidence of<br>autoimmune reaction<br>involving a non-<br>essential organ or<br>function (e.g.,<br>hypothyroidism),<br>requiring treatment<br>other than<br>immunosuppressive<br>drugs | reversible autoimmune reaction involving function of a major organ or other adverse event (e.g., transient colitis or anemia), requiring short-term immunosuppressive treatment | autoimmune reaction<br>causing major grade 4<br>organ dysfunction;<br>progressive and<br>irreversible reaction;<br>long-term<br>administration of high-<br>dose immuno-<br>suppressive therapy<br>required |
| Also consider Hypothyroidism | | bin, Hemolysis. | | | |
| Serum sickness | none | - | - | present | - |
| Urticaria is graded in the DER<br>hypersensitivity reaction, grad | | N category if it occurs as an isol ion/hypersensitivity above. | ated symptom. If it occurs | with other manifestations of | allergic or |
| Vasculitis | none | mild, not requiring treatment | symptomatic, requiring medication | requiring steroids | ischemic changes or requiring amputation |
| Allergy/Immunology - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | AUDITORY | //HEARING | | |
| Conductive hearing loss is grad | ded as Middle ear/l | nearing in the AUDITORY/HEA | RING category. | | |
| Earache is graded in the PAIN | category. | | | | |
| External auditory canal | normal | external otitis with<br>erythema or dry<br>desquamation | external otitis with<br>moist desquamation | external otitis with<br>discharge, mastoiditis | necrosis of the canal soft tissue or bone |
| Note: Changes associated with | radiation to exterr | nal ear (pinnae) are graded under | r Radiation dermatitis in the | DERMATOLOGY/SKIN | category. |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Inner ear/hearing | normal | hearing loss on<br>audiometry only | tinnitus or hearing loss,<br>not requiring hearing<br>aid or treatment | tinnitus or hearing loss,<br>correctable with hearing<br>aid or treatment | severe unilateral or<br>bilateral hearing loss<br>(deafness), not<br>correctable |
| Middle ear/hearing | normal | serous otitis without<br>subjective decrease in<br>hearing | serous otitis or infection<br>requiring medical<br>intervention; subjective<br>decrease in hearing;<br>rupture of tympanic<br>membrane with<br>discharge | otitis with discharge,<br>mastoiditis or<br>conductive hearing loss | necrosis of the canal<br>soft tissue or bone |
| Auditory/Hearing - Other (Specify,) | normal | mild | moderate | severe | life-threatening or disabling |
| | | BLOOD/BON | IE MARROW | | |
| Bone marrow cellularity | normal for age | mildly hypocellular or<br>≤25% reduction from<br>normal cellularity for<br>age | moderately hypocellular<br>or >25 - ≤50%<br>reduction from normal<br>cellularity for age or >2<br>but <4 weeks to<br>recovery of normal<br>bone marrow cellularity | severely hypocellular or >50 - <75% reduction in cellularity for age or 4 - 6 weeks to recovery of normal bone marrow cellularity | aplasia or >6 weeks to<br>recovery of normal<br>bone marrow cellularity |
| Normal ranges: | | | | | |
| children (≤18 years) | 90% cellularity<br>average | | | | |
| younger adults (19-59) | 60 - 70%<br>cellularity average | | | | |
| older adults (≥60 years) | 50% cellularity average | | | | |
| Note: Grade Bone marrow cell | ularity only for change | s related to treatment not dis | sease. | | |
| CD4 count | WNL | <lln -="" 500="" mm<sup="">3</lln> | 200 - <500/mm <sup>3</sup> | 50 - <200/mm <sup>3</sup> | <50/mm <sup>3</sup> |
| Haptoglobin | normal | decreased | - | absent | - |
| Hemoglobin (Hgb) | WNL | <lln -="" 10.0="" dl<br="" g=""><lln -="" 100="" g="" l<br=""><lln -="" 6.2="" l<="" mmol="" td=""><td>8.0 - &lt;10.0 g/dL<br/>80 - &lt;100 g/L<br/>4.9 - &lt;6.2 mmol/L</td><td>6.5 - &lt;8.0 g/dL<br/>65 - &lt;80 g/L<br/>4.0 - &lt;4.9 mmol/L</td><td>&lt;6.5 g/dL<br/>&lt;65 g/L<br/>&lt;4.0 mmol/L</td></lln></lln></lln> | 8.0 - <10.0 g/dL<br>80 - <100 g/L<br>4.9 - <6.2 mmol/L | 6.5 - <8.0 g/dL<br>65 - <80 g/L<br>4.0 - <4.9 mmol/L | <6.5 g/dL<br><65 g/L<br><4.0 mmol/L |
| For leukemia studies or bone marrow infiltrative/<br>myelophthisic processes, if specified in the protocol. | WNL | 10 - <25% decrease<br>from pretreatment | 25 - <50% decrease from pretreatment | 50 - <75% decrease from pretreatment | ≥75% decrease from pretreatment |
| Hemolysis (e.g., immune<br>hemolytic anemia, drug-<br>related hemolysis, other) Also consider Haptoglobin, He | none | only laboratory<br>evidence of hemolysis<br>[e.g., direct antiglobulin<br>test (DAT, Coombs*)<br>schistocytes] | evidence of red cell<br>destruction and ≥2gm<br>decrease in hemoglobin,<br>no transfusion | requiring transfusion<br>and/or medical<br>intervention (e.g.,<br>steroids) | catastrophic<br>consequences of<br>hemolysis (e.g., renal<br>failure, hypotension,<br>bronchospasm,<br>emergency<br>splenectomy) |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

CTC Version 2.0 Publish Date: April 30, 1999

| | Grade | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Leukocytes (total WBC) | WNL | <lln -="" 10<sup="" 3.0="" x="">9 /L<br/><lln -="" 3000="" mm<sup="">3</lln></lln> | ≥2.0 - <3.0 x 10 <sup>9</sup> /L<br>≥2000 - <3000/mm <sup>3</sup> | ≥1.0 - <2.0 x 10 <sup>9</sup> /L<br>≥1000 - <2000/mm <sup>3</sup> | <1.0 x 10 <sup>9</sup> /L<br><1000/mm <sup>3</sup> |
| For BMT studies, if specified in the protocol. | WNL | ≥2.0 - <3.0 X 10 <sup>9</sup> /L<br>≥2000 - <3000/mm <sup>3</sup> | ≥1.0 - <2.0 x 10 <sup>9</sup> /L<br>≥1000 - <2000/mm <sup>3</sup> | ≥0.5 - <1.0 x 10 <sup>9</sup> /L<br>≥500 - <1000/mm <sup>3</sup> | <0.5 x 10 <sup>9</sup> /L<br><500/mm <sup>3</sup> |
| For pediatric BMT studies (using age, race and sex normal values), if specified in the protocol. | | ≥75 - <100% LLN | ≥50 - <75% LLN | ≥25 - 50% LLN | <25% LLN |
| Lymphopenia | WNL | <lln -="" 1.0="" 10<sup="" x="">9 /L<br/><lln -="" 1000="" mm<sup="">3</lln></lln> | ≥0.5 - <1.0 x 10 <sup>9</sup> /L<br>≥500 - <1000/mm <sup>3</sup> | <0.5 x 10 <sup>9</sup> /L<br><500/mm <sup>3</sup> | - |
| For pediatric BMT studies (using age, race and sex normal values), if specified in the protocol. | | ≥75 - <100%LLN | ≥50 - <75%LLN | ≥25 - <50%LLN | <25%LLN |
| Neutrophils/granulocytes (ANC/AGC) | WNL | ≥1.5 - <2.0 x 10 <sup>9</sup> /L<br>≥1500 - <2000/mm <sup>3</sup> | $\geq 1.0 - < 1.5 \times 10^9 / L$<br>$\geq 1000 - < 1500 / mm^3$ | ≥0.5 - <1.0 x 10 <sup>9</sup> /L<br>≥500 - <1000/mm <sup>3</sup> | <0.5 x 10 <sup>9</sup> /L<br><500/mm <sup>3</sup> |
| For BMT studies, if specified in the protocol. | WNL | $\geq 1.0 - < 1.5 \times 10^9 / L$<br>$\geq 1000 - < 1500 / mm^3$ | ≥0.5 - <1.0 x 10 <sup>9</sup> /L<br>≥500 - <1000/mm <sup>3</sup> | ≥0.1 - <0.5 x 10 <sup>9</sup> /L<br>≥100 - <500/mm <sup>3</sup> | <0.1 x 10 <sup>9</sup> /L<br><100/mm <sup>3</sup> |
| For leukemia studies or bone marrow infiltrative/<br>myelophthisic process, if specified in the protocol. | WNL | 10 - <25% decrease<br>from baseline | 25 - <50% decrease from baseline | 50 - <75% decrease from baseline | ≥75% decrease from baseline |
| Platelets | WNL | <lln -="" 10<sup="" 75.0="" x="">9 /L<br/><lln -="" 75,000="" mm<sup="">3</lln></lln> | ≥50.0 - <75.0 x 10 <sup>9</sup> /L<br>≥50,000 - <75,000/mm <sup>3</sup> | ≥10.0 - <50.0 x 10 <sup>9</sup> /L<br>≥10,000 - <50,000/mm <sup>3</sup> | <10.0 x 10 <sup>9</sup> /L<br><10,000/mm <sup>3</sup> |
| For BMT studies, if specified in the protocol. | WNL | ≥50.0 - <75.0 x 10 <sup>9</sup> /L<br>≥50,000 - <75,000/mm <sup>3</sup> | ≥20.0 - <50.0 x 10 <sup>9</sup> /L<br>≥20,000 - <50,000/mm <sup>3</sup> | ≥10.0 - <20.0 x 10 <sup>9</sup> /L<br>≥10,000 - <20,000/mm <sup>3</sup> | <10.0 x 10 <sup>9</sup> /L<br><10,000/mm <sup>3</sup> |
| For leukemia studies or bone<br>marrow infiltrative/<br>myelophthisic process, if<br>specified in the protocol. | WNL | 10 - <25% decrease<br>from baseline | 25 - <50% decrease from baseline | 50 - <75% decrease from baseline | ≥75% decrease from baseline |
| Transfusion: Platelets | none | - | - | yes | platelet transfusions and<br>other measures required<br>to improve platelet<br>increment; platelet<br>transfusion<br>refractoriness associated<br>with life-threatening<br>bleeding. (e.g., HLA or<br>cross matched platelet<br>transfusions) |
| For BMT studies, if specified in the protocol. | none | 1 platelet transfusion in<br>24 hours | 2 platelet transfusions in<br>24 hours | ≥3 platelet transfusions<br>in 24 hours | platelet transfusions and<br>other measures required<br>to improve platelet<br>increment; platelet<br>transfusion<br>refractoriness associated<br>with life-threatening<br>bleeding. (e.g., HLA or<br>cross matched platelet<br>transfusions) |
| Also consider Platelets. | | | | | |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Transfusion: pRBCs | none | - | - | yes | - |
| For BMT studies, if specified in the protocol. | none | ≤2 u pRBC in 24 hours<br>elective or planned | 3 u pRBC in 24 hours<br>elective or planned | ≥4 u pRBC in 24 hours | hemorrhage or<br>hemolysis associated<br>with life-threatening<br>anemia; medical<br>intervention required to<br>improve hemoglobin |
| For pediatric BMT studies, if specified in the protocol. | none | ≤15mL/kg in 24 hours<br>elective or planned | >15 - ≤30mL/kg in 24<br>hours elective or<br>planned | >30mL/kg in 24 hours | hemorrhage or<br>hemolysis associated<br>with life-threatening<br>anemia; medical<br>intervention required to<br>improve hemoglobin |
| Also consider Hemoglobin. | | | | | |
| Blood/Bone Marrow - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | CA | RDIOVASCULA | R (ARRHYTHM | IIA) | |
| Conduction abnormality/<br>Atrioventricular heart block | none | asymptomatic, not<br>requiring treatment<br>(e.g., Mobitz type I<br>second-degree AV<br>block, Wenckebach) | symptomatic, but not<br>requiring treatment | symptomatic and<br>requiring treatment<br>(e.g., Mobitz type II<br>second-degree AV<br>block, third-degree AV<br>block) | life-threatening (e.g.,<br>arrhythmia associated<br>with CHF, hypotension,<br>syncope, shock) |
| Nodal/junctional<br>arrhythmia/dysrhythmia | none | asymptomatic, not requiring treatment | symptomatic, but not<br>requiring treatment | symptomatic and requiring treatment | life-threatening (e.g.,<br>arrhythmia associated<br>with CHF, hypotension,<br>syncope, shock) |
| Palpitations | none | present | - | - | - |
| Note: Grade palpitations only i | n the absence of a docu | mented arrhythmia. | | | |
| Prolonged QTc interval<br>(QTc>0.48 seconds) | none | asymptomatic, not requiring treatment | symptomatic, but not<br>requiring treatment | symptomatic and requiring treatment | life-threatening (e.g.,<br>arrhythmia associated<br>with CHF, hypotension,<br>syncope, shock) |
| Sinus bradycardia | none | asymptomatic, not requiring treatment | symptomatic, but not<br>requiring treatment | symptomatic and requiring treatment | life-threatening (e.g.,<br>arrhythmia associated<br>with CHF, hypotension,<br>syncope, shock) |
| Sinus tachycardia | none | asymptomatic, not requiring treatment | symptomatic, but not requiring treatment | symptomatic and<br>requiring treatment of<br>underlying cause | - |
| Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) | none | asymptomatic, not requiring treatment | symptomatic, but not<br>requiring treatment | symptomatic and requiring treatment | life-threatening (e.g.,<br>arrhythmia associated<br>with CHF, hypotension,<br>syncope, shock) |
| Syncope (fainting) is graded in | the NEUROLOGY cat | egory. | | | |
| Vasovagal episode | none | - | present without loss of consciousness | present with loss of consciousness | - |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| | Gr | ade | | |
|---|---|---|---|---|
| 0 | 1 | 2 | 3 | 4 |
| none | asymptomatic, not requiring treatment | symptomatic, but not<br>requiring treatment | symptomatic and requiring treatment | life-threatening (e.g.,<br>arrhythmia associated<br>with CHF, hypotension,<br>syncope, shock) |
| none | asymptomatic, not requiring treatment | symptomatic, but not requiring treatment | symptomatic, and<br>requiring treatment of<br>underlying cause | life-threatening (e.g.,<br>arrhythmia associated<br>with CHF, hypotension,<br>syncope, shock) |
| | CARDIOVASCU | LAR (GENERAL | ) | |
| absent | - | symptomatic, but not<br>requiring fluid support | respiratory compromise<br>or requiring fluids | life-threatening;<br>requiring pressor<br>support and/or<br>ventilatory support |
| none | non-specific T - wave<br>flattening or changes | asymptomatic, ST - and<br>T - wave changes<br>suggesting ischemia | angina without evidence of infarction | acute myocardial infarction |
| normal | asymptomatic decline<br>of resting ejection<br>fraction of ≥10% but<br><20% of baseline value;<br>shortening fraction<br>≥24% but <30% | asymptomatic but<br>resting ejection fraction<br>below LLN for<br>laboratory or decline of<br>resting ejection fraction<br>>20% of baseline value;<br><24% shortening<br>fraction | CHF responsive to treatment | severe or refractory<br>CHF or requiring<br>intubation |
| is graded in the l | NEUROLOGY category. | | | |
| normal | - | - | levels consistent with<br>unstable angina as<br>defined by the<br>manufacturer | levels consistent with<br>myocardial infarction as<br>defined by the<br>manufacturer |
| normal | ≥0.03 - <0.05 ng/mL | ≥0.05 - <0.1 ng/mL | ≥0.1 - <0.2 ng/mL | ≥0.2 ng/mL |
| none | asymptomatic, not requiring therapy | symptomatic, requiring<br>therapy | symptomatic edema<br>limiting function and<br>unresponsive to therapy<br>or requiring drug<br>discontinuation | anasarca (severe<br>generalized edema) |
| none | asymptomatic, transient<br>increase by >20 mmHg<br>(diastolic) or to<br>>150/100* if previously<br>WNL; not requiring<br>treatment | recurrent or persistent<br>or symptomatic increase<br>by >20 mmHg<br>(diastolic) or to<br>>150/100* if previously<br>WNL; not requiring<br>treatment | requiring therapy or<br>more intensive therapy<br>than previously | hypertensive crisis |
| | none none absent none normal is graded in the N normal normal | none asymptomatic, not requiring treatment CARDIOVASCU absent - none non-specific T - wave flattening or changes normal asymptomatic decline of resting ejection fraction of≥10% but <20% of baseline value; shortening fraction ≥24% but <30% is graded in the NEUROLOGY category. normal - normal ≥0.03 -<0.05 ng/mL none asymptomatic, not requiring therapy none asymptomatic, transient increase by>20 mmHg (diastolic) or to >150/100* if previously WNL; not requiring theraping treating fraction increase by>20 mmHg (diastolic) or to >150/100* if previously WNL; not requiring | none asymptomatic, not requiring treatment Symptomatic, but not requiring treatment | none asymptomatic, not requiring treatment symptomatic, but not requiring treatment requiring treatment symptomatic, and requiring treatment symptomatic, and requiring treatment of underlying cause CARDIOVASCULAR (GENERAL) |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

CA139387

| | Grade | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Hypotension | none | changes, but not<br>requiring therapy<br>(including transient<br>orthostatic hypotension) | requiring brief fluid<br>replacement or other<br>therapy but not<br>hospitalization; no<br>physiologic<br>consequences | requiring therapy and<br>sustained medical<br>attention, but resolves<br>without persisting<br>physiologic<br>consequences | shock (associated with<br>acidemia and impairing<br>vital organ function due<br>to tissue hypoperfusion) |
| Also consider Syncope (fainti | ng). | | | | |
| Notes: Angina or MI is graded | l as Cardiac-ischemia/in | farction in the CARDIOVA | SCULAR (GENERAL) cate | egory. | |
| For pediatric patients, or three measurements | | r less in infants up to 1 year | old and 70 mmHg or less in | n children older than 1 year | of age, use two successive |
| Myocarditis | none | - | - | CHF responsive to treatment | severe or refractory<br>CHF |
| Operative injury of vein/artery | none | primary suture repair<br>for injury, but not<br>requiring transfusion | primary suture repair<br>for injury, requiring<br>transfusion | vascular occlusion<br>requiring surgery or<br>bypass for injury | myocardial infarction;<br>resection of organ (e.g.,<br>bowel, limb) |
| Pericardial effusion/<br>pericarditis | none | asymptomatic effusion,<br>not requiring treatment | pericarditis (rub, ECG<br>changes, and/or chest<br>pain) | with physiologic consequences | tamponade (drainage or<br>pericardial window<br>required) |
| Peripheral arterial ischemia | none | - | brief episode of<br>ischemia managed non-<br>surgically and without<br>permanent deficit | requiring surgical intervention | life-threatening or with<br>permanent functional<br>deficit (e.g.,<br>amputation) |
| Phlebitis (superficial) | none | - | present | - | - |
| Notes: Injection site reaction i | s graded in the DERMA | TOLOGY/SKIN category. | | | |
| Thrombosis/embolism | is graded in the CARDI | OVASCULAR (GENERAL | .) category. | | |
| Syncope (fainting) is graded in | n the NEUROLOGY ca | tegory. | | | |
| Thrombosis/embolism | none | - | deep vein thrombosis,<br>not requiring<br>anticoagulant | deep vein thrombosis,<br>requiring anticoagulant<br>therapy | embolic event including<br>pulmonary embolism |
| Vein/artery operative injury is | Vein/artery operative injury is graded as Operative injury of vein/artery in the CARDIOVASCULAR (GENERAL) category. | | | | |
| Visceral arterial ischemia<br>(non-myocardial) | none | - | brief episode of<br>ischemia managed non-<br>surgically and without<br>permanent deficit | requiring surgical intervention | life-threatening or with<br>permanent functional<br>deficit (e.g., resection of<br>ileum) |
| Cardiovascular/ General - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998

Revised March 23, 1998

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| | | COAGU | LATION | | |
| Note: See the HEMORRHAG | E category for grading | the severity of bleeding ever | nts. | | |
| DIC<br>(disseminated intravascular<br>coagulation) | absent | - | - | laboratory findings<br>present with <u>no</u><br>bleeding | laboratory findings <u>and</u><br>bleeding |
| Also consider Platelets. | | | | | |
| Note: Must have increased fibr | rin split products or D- | limer in order to grade as D | IC. | | |
| Fibrinogen | WNL | ≥0.75 - <1.0 x LLN | ≥0.5 - <0.75 x LLN | ≥0.25 - <0.5 x LLN | <0.25 x LLN |
| For leukemia studies or bone marrow infiltrative/<br>myelophthisic process, if specified in the protocol. | WNL | <20% decrease from<br>pretreatment value or<br>LLN | ≥20 - <40% decrease<br>from pretreatment value<br>or LLN | ≥40 - <70% decrease<br>from pretreatment value<br>or LLN | <50 mg |
| Partial thromboplastin time (PTT) | WNL | >ULN - ≤1.5 x ULN | >1.5 - ≤2 x ULN | >2 x ULN | - |
| Phlebitis is graded in the CAR | DIOVASCULAR (GE | NERAL) category. | | | |
| Prothrombin time (PT) | WNL | >ULN -≤1.5 x ULN | >1.5 - ≤2 x ULN | >2 x ULN | - |
| Thrombosis/embolism is grade | ed in the CARDIOVAS | CULAR (GENERAL) categ | gory. | | |
| Thrombotic<br>microangiopathy (e.g.,<br>thrombotic<br>thrombocytopenic<br>purpura/TTP or hemolytic<br>uremic syndrome/HUS) | absent | - | - | laboratory findings<br>present without clinical<br>consequences | laboratory findings and<br>clinical consequences,<br>(e.g., CNS hemorrhage/<br>bleeding or thrombosis/<br>embolism or renal<br>failure) requiring<br>therapeutic intervention |
| For BMT studies, if specified in the protocol. | - | evidence of RBC<br>destruction<br>(schistocytosis) without<br>clinical consequences | evidence of RBC<br>destruction with<br>elevated creatinine (≤3<br>x ULN) | evidence of RBC<br>destruction with<br>creatinine (>3 x ULN)<br>not requiring dialysis | evidence of RBC<br>destruction with renal<br>failure requiring<br>dialysis and/or<br>encephalopathy |
| Also consider Hemoglobin, Pla | atelets, Creatinine. | | | | |
| Note: Must have microangiopa | thic changes on blood | smear (e.g., schistocytes, he | lmet cells, red cell fragments | s). | |
| Coagulation - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | CONSTITUTION | NAL SYMPTOMS | | |
| Fatigue<br>(lethargy, malaise, asthenia) | none | increased fatigue over<br>baseline, but not<br>altering normal<br>activities | moderate (e.g., decrease in performance status by 1 ECOG level or 20% Karnofsky or Lansky) or causing difficulty performing some activities | severe (e.g., decrease in<br>performance status by<br>≥2 ECOG levels <u>or</u> 40%<br>Karnofsky or <i>Lansky</i> ) <u>or</u><br>loss of ability to<br>perform some activities | bedridden or disabling |
| Note: See Appendix III for per | formance status scales. | | | | |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Fever (in the absence of neutropenia, where neutropenia is defined as AGC <1.0 x 10 <sup>9</sup> /L) | none | 38.0 - 39.0°C (100.4 - 102.2°F) | 39.1 - 40.0°C (102.3 - 104.0°F) | >40.0°C (>104.0°F ) for<br><24hrs | >40.0°C (>104.0°F) fo<br>>24hrs |
| Also consider Allergic reaction | n/hypersensitivity. | | | | |
| Note: The temperature measur | rements listed above a | re oral or tympanic. | | | |
| Hot flashes/flushes are graded | in the ENDOCRINE | category. | | | |
| Rigors, chills | none | mild, requiring<br>symptomatic treatment<br>(e.g., blanket) or non-<br>narcotic medication | severe and/or<br>prolonged, requiring<br>narcotic medication | not responsive to narcotic medication | - |
| Sweating<br>(diaphoresis) | normal | mild and occasional | frequent or drenching | - | - |
| Weight gain | <5% | 5 - <10% | 10 - <20% | ≥20% | - |
| Also consider Ascites, Edema | , Pleural effusion (nor | n-malignant). | | | |
| Weight gain associated with<br>Veno-Occlusive Disease<br>(VOD) for BMT studies, if<br>specified in the protocol. | <2% | ≥2 - <5% | ≥5 - <10% | ≥10% or as ascites | ≥10% or fluid retention<br>resulting in pulmonary<br>failure |
| Also consider Ascites, Edema | , Pleural effusion (nor | n-malignant). | | | |
| Weight loss | <5% | 5 - <10% | 10 - <20% | ≥20% | - |
| Also consider Vomiting, Dehy | dration, Diarrhea. | | | | |
| Constitutional Symptoms -<br>Other<br>(Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | DERMATO | LOGY/SKIN | | |
| Alopecia | normal | mild hair loss | pronounced hair loss | - | - |
| Bruising (in absence of grade 3 or 4 thrombocytopenia) | none | localized or in<br>dependent area | generalized | - | - |
| Note: Bruising resulting from HEMORRHAGE categ | | ocytopenia is graded as Petech<br>IATOLOGY/SKIN category. | iae/purpura <u>and</u> Hemorrhag | e/bleeding with grade 3 or 4 | thrombocytopenia in the |
| Dry skin | normal | controlled with emollients | not controlled with emollients | - | - |
| Erythema multiforme (e.g.,<br>Stevens-Johnson syndrome,<br>toxic epidermal necrolysis) | absent | 2 | scattered, but not<br>generalized eruption | severe or requiring IV<br>fluids (e.g., generalized<br>rash or painful<br>stomatitis) | life-threatening (e.g.,<br>exfoliative or ulcerating<br>dermatitis or requiring<br>enteral or parenteral<br>nutritional support) |
| Flushing | absent | present | - | - | - |
| Hand-foot skin reaction | none | skin changes or<br>dermatitis without pain<br>(e.g., erythema, peeling) | skin changes with pain,<br>not interfering with<br>function | skin changes with pain,<br>interfering with<br>function | - |
| Injection site reaction | none | pain or itching or<br>erythema | pain or swelling, with<br>inflammation or<br>phlebitis | ulceration or necrosis<br>that is severe or<br>prolonged, or requiring<br>surgery | - |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| Nail changes normal discoloration or ridging (kolonychia) or pitting of auti(s) or pain in anilbeds Petechnice is graded in the HEMORRHAGE category. Photosensitivity none painless crythema painful crythema crythema with desquamation changes (e.g., none changes changes changes changes pigmentation changes pigmentation changes pigmentation changes primary trivilia. Pruritus none mild or localized, relieved spontaneously or by local measures or by systemic measures. Purpura is graded in the HEMORRHAGE category. Radiation demantities and category as Pain due to radiation. Radiation recall reaction category as Pain due to radiation. Radiation recall reaction problem category as Pain due to radiation. Radiation recall reaction problem category as Pain due to radiation. Radiation recall reaction problem category as Pain due to radiation. Radiation recall reaction problem category as Pain at the recall problem category as Pain at the recall problem category as Pain at the recall problem category as Pain at the recall problem category as Pain | | Grade | | | | |
|---|---|---|---|---|---|---|
| Petechiae is graded in the HEMORRHAGE category. Photosenstitivity none painless erythema erythema erythema or dry desquamation changes (e.g., none mild or localized, releved spontaneously or hypothema encaures or hypothema erythema or dry desquamation or hypothema erythema or dry desquamation or hone faint erythema or dry desquamation or easily confined to skin folds; noticed by mildress destination or absence or discharged and poorty controlled or hypothema or a patchy moist desquamation. Note: Pain associated with radiation dermatitis is graded separately in the PAIN extragory as Pain due to radiation. Note: Pain associated with radiation dermatitis is graded separately in the PAIN extragory as Pain due to radiation. Note: Pain associated with radiation dermatitis is graded separately in the PAIN extragory as Pain due to radiation. Note: Pain associated with radiation dermatitis is graded separately in the PAIN extragory as Pain due to radiation. Radiation recall reaction (reaction following chemosherapy in the absence of additional radiation demandation therapy that excess radiation port) Ranhi desquamation none macular or papular eruption or erythema with practice or cheared and the confined to skin folds; noted associated symptoms existed expursion or erythema with practice or cheared and the confined to skin folds; noted associated symptoms existed expursion or erythema with practice or cheared and the confined to skin folds; noted expursion or erythema with practice or cheared and the confined to skin folds; noted associated symptoms expursion or erythema with practice or cheared and the confined to skin folds; noted associated symptoms or erythema with practice or cheared and the confined to skin folds; noted associated symptoms or erythema erythema or a patchy noted associated with radiation dermatics or patchy noted associated with radiation dermatics or patchy noted associated with radia | Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Photosensitivity none painless crythema painful crythema crythema with desquamation Pigmentation changes (e.g., none localized pigmentation changes mild or localized, relieved spontaneously or by local measures Pruritus none mild or localized, relieved spontaneously or by systemic measures Purpura is graded in the HEMORRHAGE category. Radiation dermatitis none faint crythema or dry desquamation, mostly confined to skin folds and creases; moderate dema such as the confined most crythema or a patchy mostl desquamation ≥1.5 cm dameter and not confined to skin folds; and creases; moderate dema none faint crythema or dry desquamation none faint crythema or dry desquamation none faint crythema or dry desquamation none macular or papular crythem or or grythema with purities or other associated symptoms associated and poorly controlled despite treatment such and poorly c | Nail changes | normal | | of nail(s) or pain in | - | - |
| Pigmentation changes (e.g., none localized pigmentation changes principle of changes localized pigmentation changes principle changes localized pigmentation changes principle changes mild or localized. Purpura is graded in the HEMORRHAGE category. Radiation dermatitis none laint crythema or dry desquamation local consider Allergic reaction hypersensitivity. Note: Pain associated with pradiation dermatitis is graded separately as Erythema or dry desquamation none law provious radiation port) Rashi desquamation none law provious radiation port) Rashi desquamation none macular or papular cruption or crythema with purities or other associated symptoms associated with gradiation port) Rashi desquamation none macular or papular cruption or crythema with purities or other associated symptoms associated with gradiation port) Rashi desquamation none macular or papular cruption or crythema with purities or other associated symptoms associated with gradiation or other lesions covering ≤50% of body surface are localized desquamation or other lesions covering ≤50% of body surface are localized with gradial or other lesions covering ≤50% of body surface are localized desquamation or other lesions covering ≤50% of body surface are localized desquamation or other lesions covering ≤50% of body surface are localized desquamation explored by the local provious and local provious area are localized desquamation or other lesions covering ≤50% of body surface or localized desquamation learned area area without private | Petechiae is graded in the HE | MORRHAGE category. | | | | |
| Pruritus none mild or Iocalized, relieved spontaneously or by Iocal measures or Purpura is graded in the HEMORRHAGE category. Radiation dermatitis none finit erythema or dry desquamation mostly confined to skin folds and creases; moderate colema modification following chemotherapy in the absence of additional radiation port) Rash/desquamation none macular or papular eruption or erythema without associated symptoms Rash/desquamation none macular or papular eruption or erythema with puritures or other associated with graded separately as Erythema multiforme in the DERMATOLOGY/SKIN category. Rash/dematitis associated with graded separately as Erythema multiforme in the DERMATOLOGY/SKIN category. Rash/desquamation associated with graded separately as Erythema multiforme in the DERMATOLOGY/SKIN category. Rash/desquamation associated with graded separately as Erythema multiform or other lesions covering <50% of body surface area without associated with graded expansion provided sequamation associated with graded separately as Erythema multiform or other lesions covering <50% of body surface area without associated with graded expansion provided sequamation or other lesions covering <50% of body surface area without associated with grade desquamation associated with grade view of the graded sequamation associated with grade view of the graded sequamation or other lesions covering <50% of body surface area without associated with grade view of the graded sequamation associated with grade view of the graded sequamation or other lesions covering <50% of body surface area without associated with grade view of the graded sequamation or other lesions covering <50% of body surface area without associated symptoms covering <50% of body surface area without associated symptoms covering <50% of body surface area without associated symptoms covering <50% of body surface area without associated symptoms covering <50% of body surface area without associated symptoms covering <50% of body surface area without associated with | Photosensitivity | none | painless erythema | painful erythema | | - |
| Purpura is graded in the HEMORRHAGE category. Radiation dermatitis none faint crythema or dry desquamation monely confined to skin folia and creases; moderate colema monely confined to skin folia and creases; moderate colema monely confined to skin folia and creases; moderate colema monely confined to skin folia and creases; moderate colema monely confined to skin folia and creases; moderate colema moderate colema monely confined to skin folia and creases; moderate colema with purultus or other section of purpular cruption or crythema with purultus or other section of purpular cruption or crythema with purultus or other section of purpular cruption or crythema with purultus or other section of purpular cruption or crythema with purultus or other section of purpular cruption or crythema covering <50% of body surface area without associated with graft versus home section of faill thickness dermitis or utlerative department or crythema with purultus or other section of purpular cruption or crythema covering <50% of body surface area without associated with graft versus home section or crythema confined to skin folia by purpular crythema or a patchy confined to skin folia to skin folia by purpular crythema or a patchy confined to skin folia by purpular crythema or a patchy confined to skin folia by purpular crythema or a patchy confined to skin folia by purpular crythema or a p | | none | | | - | - |
| Radiation dermatitis none faint erythema or dry desquamation moist desquamation ≥1.5 cm dischessed sermis; may include bleeding not of trauma or abrasion. Note: Pain associated with radiation dermatitis is graded separately in the PAIN category as Pain due to radiation. Note: Pain associated with radiation dermatitis is graded separately in the PAIN category as Pain due to radiation. Note: Pain associated with radiation dermatitis is graded separately in the PAIN category as Pain due to radiation. Note: Pain associated with radiation dermatitis is graded separately in the PAIN category as Pain due to radiation. Radiation recall reaction none faint erythema or dry desquamation mostly confined to skin folds; pitting edema sinclude bleeding not induced by minor trauma or abrasion therapy that occurs in a previous radiation port) Rash/desquamation none macular or papular eruption or erythema without associated symptoms covering <50% of body surface are sufficient eruption or desquamation or desquamation or other lesions covering <50% of body surface are and not confined to skin folds; pitting edema sinclude bleeding not induced by minor trauma or abrasion full thickness dermis; may include of the desquamation or desquamation eruption or desquamation confident to skin folds; pitting edema sinclude bleeding not induced by minor macular, papular or macular or papular eruption or erythema or a patchy moist desquamation event or side or patchy minor desquamation event or desquamation event or desquamation event or desquamation | Pruritus | none | relieved spontaneously | relieved spontaneously | and poorly controlled | - |
| desquamation crythema or a patchy moist desquamation club diameter and not induced by minor moderate cdema club moderate cdem | Purpura is graded in the HEM | ORRHAGE category. | | | | |
| Radiation recall reaction (reaction following chemotherapy in the absence of additional radiation port) Rash/desquamation none macular or papular cruption or crythema without associated symptoms macular or papular cruption or crythema without associated symptoms macular or papular cruption or crythema without associated symptoms or other lesions covering 50% of body surface area without sasociated with graft versus shost diseases (GVHD) for BMT studies, if specified in the protocol. Rash/desquamation None macular or papular cruption or crythema without associated symptoms or covering 225 - 50% of body surface area macular or papular cruption or crythema with puritus or other associated symptoms or covering 225 - 50% of body surface area macular or papular cruption or crythema with puritus or other associated symptoms overing 50% of body surface area sometrate to brisk desquamation overing 225 - 50% of body surface area symptomatic and not confluent moist desquamation plant thickness dermis, may include bleeding not induced by minor trauma or abrasion symptomatic generalized crythorderma or macular, papular or vesicular cruption or desquamation overing 250% of body surface area swint puritus or other associated symptoms overing 425% of body surface area without associated or propular cruption or crythema covering 225 - 50% of body surface area macular or papular cruption or desquamation overing 225 - 50% of body surface area swint puritus or other associated by minor trauma or abrasion symptomatic explainment overing 250% of body surface area swint puritus or other associated by minor trauma or abrasion symptomatic explainment overing 250% of body surface area swint puritus or other associated by minor trauma or abrasion symptomatic explainment overing 250% of body surface area swint puritus or other associated by minor trauma or abrasion symptomatic explainment overing 250% of body surface area swint puritus or other associated by minor trauma or abrasion macular or papular cruption or | Radiation dermatitis | none | | erythema or a patchy<br>moist desquamation,<br>mostly confined to skin<br>folds and creases; | desquamation ≥1.5 cm<br>diameter and not<br>confined to skin folds; | ulceration of full<br>thickness dermis; may<br>include bleeding not<br>induced by minor |
| desquamation ≥ 1.5 cm distinguishment of additional radiation of additional radiation port therapy in the absence of additional radiation previous radiation port) Rash/desquamation none macular or papular eruption or erythema without associated symptoms macular or papular eruption or erythema without associated symptoms macular or papular eruption or erythema without associated symptoms macular or papular eruption or erythema without associated symptoms macular or papular eruption or erythema evide of body surface or localized desquamation or other lesions covering <50% of body surface area Also consider Allergic reaction/hypersensitivity. Note: Stevens-Johnson syndrome is graded separately as Erythema multiforme in the DERMATOLOGY/SKIN category. Rash/dermatitis associated with high-dose chemotherapy or BMT studies. None macular or papular eruption or dry desquamation mone macular or papular eruption or erythema or a patchy moist desquamation, mostly confined to skin folds; pitting edema vibration of desquamation stellar eruption or desquamation to overing ≥50% of body surface area without associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol. More area without associated symptoms associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol. | Note: Pain associated with rad | liation dermatitis is grad | ed separately in the PAIN c | ategory as Pain due to radiat | tion. | |
| eruption or erythema with puritus or other associated symptoms covering <50% of body surface area or localized desquamation or other lesions covering <50% of body surface area Also consider Allergic reaction/hypersensitivity. Note: Stevens-Johnson syndrome is graded separately as Erythema multiforme in the DERMATOLOGY/SKIN category. Rash/dermatitis associated with high-dose chemotherapy or BMT studies. None macular or papular eruption or desquamation with high-dose chemotherapy or BMT studies. None macular or papular eruption or erythema or a patchy moist desquamation, mostly confined to skin folds and creases; moderate edema None macular or papular eruption or erythema or a patchy moist desquamation confined to skin folds and creases; moderate edema None acular or papular eruption or erythema or a patchy moist desquamation confined to skin folds and creases; moderate edema Rash/desquamation None associated with graft versus host disease (GVHD) for surface area without associated symptoms covering ≥25 - <50% of body surface or localized desquamation or or evithema with pruritus or other associated symptoms associated symptoms covering ≥25 - <50% of body surface or localized desquamation or or evithema covering ≥25 - <50% of body surface or localized desquamation or or localized desquamation or or localized desquamation or or localized desquamation or or localized desquamation covering ≥25 - <50% of body surface area Also consider Allergic reaction/hypersensitivity. | Radiation recall reaction<br>(reaction following<br>chemotherapy in the absence<br>of additional radiation<br>therapy that occurs in a<br>previous radiation port) | none | | erythema or a patchy<br>moist desquamation,<br>mostly confined to skin<br>folds and creases; | desquamation ≥1.5 cm<br>diameter and not<br>confined to skin folds; | ulceration of full<br>thickness dermis; may<br>include bleeding not<br>induced by minor |
| Note: Stevens-Johnson syndrome is graded separately as Erythema multiforme in the DERMATOLOGY/SKIN category. Rash/dermatitis associated with high-dose chemotherapy or BMT studies. Rash/desquamation Rash/desquamation Rash/desquamation None macular or papular eruption or erythema covering <25% of body surface or localized desquamation, mostly confined to skin folds; pitting edema macular or papular eruption or erythema associated symptoms covering ≥25 -<50% of body surface or localized desquamation, or desquamation, or desquamation or other lesions covering ≥25 -<50% of body surface area skin necrosis or ulcerative desquamation ≥1.5 cm diameter and not confined to skin folds; pitting edema symptomatic generalized erythorderma or symptomatic generalized erythorderma or symptomatic macular, papular or vesicular eruption, with bullous formation, or desquamation, or desquamation or other lesions covering ≥25 -<50% of body surface area skin necrosis or ulcerative desquamation skin necrosis or ulcerative desquamation or full thickness dermit; may include spontaneous bleeding not induced by minor trauma or abrasion macular or papular eruption or erythema associated symptoms covering ≥25 -<50% of body surface or localized desquamation or other lesions covering ≥25 -<50% of body surface area skin necrosis or ulcerative desquamation or full thickness dermit; may include spontaneous bleeding not induced by minor trauma or abrasion macular or papular eruption or erythema associated symptoms covering ≥25 -<50% of body surface area skin necrosis or ulcerative desquamation, mostly confined to skin folds, pitting edema symptomatic generalized erythorderma or symptomatic generalized erythorderma or symptomatic macular, papular or vesicular eruption, with bullous formation, or desquamation, or desquamation or or desquamation or or desquamation covering ≥50% of body surface area | Rash/desquamation | none | eruption or erythema<br>without associated | eruption or erythema<br>with pruritus or other<br>associated symptoms<br>covering <50% of body<br>surface or localized<br>desquamation or other<br>lesions covering <50% | generalized erythroderma or macular, papular or vesicular eruption or desquamation covering ≥50% of body surface | dermatitis or ulcerativ |
| Rash/dermatitis associated with high-dose chemotherapy or BMT studies. Rash/desquamation Rash/desquamation Rash/desquamation None macular or papular eruption or erythema covering <25% of body surface area without the protocol. Rash/desquamation Rome macular or papular eruption or erythema covering ≥25 - <50% of body surface area moderate to brisk erythema or a patchy moist desquamation, mostly confined to skin folds; pitting edema to confined to skin folds; pitting edema to in diudced by minor trauma or abrasion macular or papular eruption or erythema covering <25% of body surface area without associated symptoms moderate to brisk erythema or a patchy moist desquamation, mostly confined to skin folds; pitting edema to confined to skin folds; pitting edema symptomatic generalized eruption or erythema with pruritus or other associated symptoms covering ≥25 - <50% of body surface or localized desquamation or other lesions covering ≥25 - <50% of body surface area skin necrosis or ulcera tion of full thickness dermis; may include spontaneous bleeding not induced by minor trauma or abrasion macular or papular eruption or erythema with pruritus or other associated symptoms covering ≥25 - <50% of body surface or localized desquamation or other lesions covering ≥25 - <50% of body surface area skin necrosis or ulcera tion of full thickness dermis; may include spontaneous bleeding not induced by minor trauma or abrasion macular or papular eruption or erythema with pruritus or other associated symptoms covering ≥25 - <50% of body surface area symptomatic generalized erythoderma or symptomatic macular, papular or vesicular eruption, with bullous formation, or desquamation covering ≥50% of body surface area ≥50% of body surface area | Also consider Allergic reaction | n/hypersensitivity. | | | | |
| with high-dose chemotherapy or BMT studies. Rash/desquamation None macular or papular eruption or erythema covering <25% of body surface area without the protocol. Rash/desquamation None macular or papular eruption or erythema covering ≥25 - <50% of body surface area without associated symptoms covering ≥25 - <50% of body surface area without or other lesions covering ≥25 - <50% of body surface area without formation, or desquamation covering ≥25 - <50% of body surface area without associated symptoms covering ≥25 - <50% of body surface area without associated symptoms covering ≥25 - <50% of body surface area without formation, or desquamation or other lesions covering ≥25 - <50% of body surface area without formation, or desquamation covering ≥50% of body surface area without formation covering ≥50% of body surface area without confined to skin folds: pitting edema with induced by minor trauma or abrasion covering c | Note: Stevens-Johnson syndro | ome is graded separately | as Erythema multiforme in | n the DERMATOLOGY/SK | IN category. | |
| associated with graft versus host disease (GVHD) for covering <25% of body surface area without associated symptoms the protocol. BMT studies, if specified in surface area without associated symptoms the protocol. BMT studies, if specified in surface area without associated symptoms to covering ≥25 - <50% of body surface or localized desquamation or other lesions covering ≥25 - <50% of body surface area Equation or erythema with pruritus or other associated symptoms symptomatic macular, papular or vesicular eruption, with bullous formation, or desquamation covering ≥50% of body surface area Equation or erythema with pruritus or other associated symptoms symptomatic macular, papular or vesicular eruption, with bullous formation or other lesions covering ≥25 - <50% of body surface area | Rash/dermatitis associated<br>with high-dose<br>chemotherapy or BMT<br>studies. | none | | erythema or a patchy<br>moist desquamation,<br>mostly confined to skin<br>folds and creases; | desquamation ≥1.5 cm<br>diameter and not<br>confined to skin folds; | dermis; may include<br>spontaneous bleeding<br>not induced by minor |
| Also consider Allansia pagatian/hymoreansitivity | Rash/desquamation<br>associated with graft versus<br>host disease (GVHD) for<br>BMT studies, if specified in<br>the protocol. | None | eruption or erythema<br>covering <25% of body<br>surface area without | eruption or erythema<br>with pruritus or other<br>associated symptoms<br>covering ≥25 - <50% of<br>body surface or<br>localized desquamation<br>or other lesions<br>covering ≥25 - <50% of | generalized<br>erythroderma or<br>symptomatic macular,<br>papular or vesicular<br>eruption, with bullous<br>formation, or<br>desquamation covering<br>≥50% of body surface | dermatitis or ulcerative<br>dermatitis or bullous |
| Also consider Allergic reaction/hypersensitivity. | Also consider Allergic reaction | n/hypersensitivity. | | | | |
| Note: Stevens-Johnson syndrome is graded separately as Erythema multiforme in the DERMATOLOGY/SKIN category. | Note. Stevens-Johnson Syndro | ome is graded separately | as Li yuicina munifoline n | THE DERIVIATOROUT/SK | in category. | |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

CA139387 Clinical Protocol

| | | Gr | rade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Urticaria<br>(hives, welts, wheals) | none | requiring no medication | requiring PO or topical<br>treatment or IV<br>medication or steroids<br>for <24 hours | requiring IV medication<br>or steroids for ≥24<br>hours | - |
| Wound-infectious | none | cellulitis | superficial infection | infection requiring IV antibiotics | necrotizing fasciitis |
| Wound-non-infectious | none | incisional separation | incisional hernia | fascial disruption without evisceration | fascial disruption with evisceration |
| Dermatology/Skin - Other<br>(Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | ENDO | CRINE | | |
| Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) | absent | - | present | - | - |
| Also consider Hyperglycemia, | Hypokalemia. | | | | |
| Feminization of male | absent | - | - | present | - |
| Gynecomastia | none | mild | pronounced or painful | pronounced or painful<br>and requiring surgery | - |
| Hot flashes/flushes | none | mild or no more than 1<br>per day | moderate and greater<br>than 1 per day | - | - |
| Hypothyroidism | absent | asymptomatic,TSH<br>elevated, no therapy<br>given | symptomatic or thyroid<br>replacement treatment<br>given | patient hospitalized for<br>manifestations of<br>hypothyroidism | myxedema coma |
| Masculinization of female | absent | - | - | present | - |
| SIADH (syndrome of inappropriate antidiuretic hormone) | absent | - | - | present | - |
| Endocrine - Other<br>(Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | GASTROIN | NTESTINAL | | |
| Amylase is graded in the MET | ABOLIC/LABORAT | ORY category. | | | |
| Anorexia | none | loss of appetite | oral intake significantly decreased | requiring IV fluids | requiring feeding tube<br>or parenteral nutrition |
| Ascites (non-malignant) | none | asymptomatic | symptomatic, requiring diuretics | symptomatic, requiring therapeutic paracentesis | life-threatening<br>physiologic<br>consequences |
| Colitis | none | - | abdominal pain with<br>mucus and/or blood in<br>stool | abdominal pain, fever,<br>change in bowel habits<br>with ileus or peritoneal<br>signs, and radiographic<br>or biopsy<br>documentation | perforation or requiring surgery or toxic megacolon |
| Also consider Hemorrhage/ble<br>Rectal bleeding/hematochezia | | 4 thrombocytopenia, Hemorr | hage/bleeding without grad | e 3 or 4 thrombocytopenia, | Melena/GI bleeding, |
| Constipation | none | requiring stool softener<br>or dietary modification | requiring laxatives | obstipation requiring<br>manual evacuation or<br>enema | obstruction or toxic megacolon |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Dehydration | none | dry mucous membranes<br>and/or diminished skin<br>turgor | requiring IV fluid replacement (brief) | requiring IV fluid replacement (sustained) | physiologic<br>consequences requiring<br>intensive care;<br>hemodynamic collapse |
| Also consider Diarrhea, Vomit | ing, Stomatitis/pharyng | itis (oral/pharyngeal mucos | itis), Hypotension. | | |
| Diarrhea patients without colostomy: | none | increase of <4<br>stools/day over pre-<br>treatment | increase of 4-6<br>stools/day, or nocturnal<br>stools | increase of ≥7<br>stools/day or<br>incontinence; or need<br>for parenteral support<br>for dehydration | physiologic<br>consequences requiring<br>intensive care; or<br>hemodynamic collapse |
| patients with a colostomy: | none | mild increase in loose,<br>watery colostomy<br>output compared with<br>pretreatment | moderate increase in<br>loose, watery colostomy<br>output compared with<br>pretreatment, but not<br>interfering with normal<br>activity | severe increase in loose,<br>watery colostomy<br>output compared with<br>pretreatment, interfering<br>with normal activity | physiologic<br>consequences, requiring<br>intensive care; or<br>hemodynamic collapse |
| Diarrhea associated with<br>graft versus host disease<br>(GVHD) for BMT studies, if<br>specified in the protocol. | None | >500 - ≤1000mL of<br>diarrhea/day | >1000 - ≤1500mL of<br>diarrhea/day | >1500mL of<br>diarrhea/day | severe abdominal pain<br>with or without ileus |
| For pediatric BMT studies, if specified in the protocol. | | >5 - ≤10 mL/kg of<br>diarrhea/day | >10 - ≤15 mL/kg of<br>diarrhea/day | >15 mL/kg of<br>diarrhea/day | - |
| Also consider Hemorrhage/ble Hypotension. | eding with grade 3 or 4 | thrombocytopenia, Hemorr | hage/bleeding without grade | 3 or 4 thrombocytopenia, P | ain, Dehydration, |
| Duodenal ulcer (requires radiographic or endoscopic documentation) | none | - | requiring medical<br>management or non-<br>surgical treatment | uncontrolled by<br>outpatient medical<br>management; requiring<br>hospitalization | perforation or bleeding,<br>requiring emergency<br>surgery |
| Dyspepsia/heartburn | none | mild | moderate | severe | - |
| Dysphagia, esophagitis,<br>odynophagia (painful<br>swallowing) | none | mild dysphagia, but can<br>eat regular diet | dysphagia, requiring<br>predominantly pureed,<br>soft, or liquid diet | dysphagia, requiring IV<br>hydration | complete obstruction<br>(cannot swallow saliva)<br>requiring enteral or<br>parenteral nutritional |
| | | | | | support, or perforation |
| Note: If the adverse event is ra | diation-related, grade ei | ther under Dysphagia-esoph | nageal related to radiation or | Dysphagia-pharyngeal rela | support, or perforation |
| Note: If the adverse event is ra Dysphagia-esophageal related to radiation | diation-related, grade <u>ei</u><br>none | ther under Dysphagia-esopl<br>mild dysphagia, but can<br>eat regular diet | ageal related to radiation or<br>dysphagia, requiring<br>predominantly pureed,<br>soft, or liquid diet | Dysphagia-pharyngeal relationship Dysphagia, requiring feeding tube, IV hydration or hyperalimentation | support, or perforation |
| Dysphagia- <u>esophageal</u> | none | mild dysphagia, but can<br>eat regular diet | dysphagia, requiring predominantly pureed, | Dysphagia, requiring<br>feeding tube, IV<br>hydration or | support, or perforation<br>ted to radiation.<br>complete obstruction<br>(cannot swallow saliva);<br>ulceration with bleeding<br>not induced by minor<br>trauma or abrasion or |
| Dysphagia- <u>esophageal</u><br>related to radiation | none<br>ation, Mucositis due to r | mild dysphagia, but can<br>eat regular diet | dysphagia, requiring predominantly pureed, | Dysphagia, requiring<br>feeding tube, IV<br>hydration or | support, or perforation<br>ted to radiation.<br>complete obstruction<br>(cannot swallow saliva);<br>ulceration with bleeding<br>not induced by minor<br>trauma or abrasion or |
| Dysphagia- <u>esophageal</u> related to radiation Also consider Pain due to radia | none<br>ation, Mucositis due to r | mild dysphagia, but can<br>eat regular diet | dysphagia, requiring predominantly pureed, | Dysphagia, requiring<br>feeding tube, IV<br>hydration or | support, or perforation ted to radiation. complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or perforation complete obstruction (cannot swallow saliva); |
| Dysphagia- <u>esophageal</u> related to radiation Also consider Pain due to radia Note: Fistula is graded separate | none ation, Mucositis due to r ely as Fistula-esophagea | mild dysphagia, but can eat regular diet radiation. al. mild dysphagia, but can eat regular diet | dysphagia, requiring predominantly pureed, soft, or liquid diet dysphagia, requiring predominantly pureed, | Dysphagia, requiring feeding tube, IV hydration or hyperalimentation dysphagia, requiring feeding tube, IV hydration or | support, or perforation ted to radiation. complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or perforation complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or |
| Dysphagia- <u>esophageal</u> related to radiation Also consider Pain due to radia Note: Fistula is graded separate Dysphagia- <u>pharyngeal</u> related to radiation | none ation, Mucositis due to r ely as Fistula-esophagea none ation, Mucositis due to r | mild dysphagia, but can eat regular diet radiation. mild dysphagia, but can eat regular diet | dysphagia, requiring predominantly pureed, soft, or liquid diet dysphagia, requiring predominantly pureed, | Dysphagia, requiring feeding tube, IV hydration or hyperalimentation dysphagia, requiring feeding tube, IV hydration or | support, or perforation ted to radiation. complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or perforation complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or |
| Dysphagia- <u>esophageal</u> related to radiation Also consider Pain due to radia Note: Fistula is graded separate Dysphagia- <u>pharyngeal</u> related to radiation Also consider Pain due to radia | none ation, Mucositis due to r ely as Fistula-esophagea none ation, Mucositis due to r | mild dysphagia, but can eat regular diet radiation. mild dysphagia, but can eat regular diet | dysphagia, requiring predominantly pureed, soft, or liquid diet dysphagia, requiring predominantly pureed, | Dysphagia, requiring feeding tube, IV hydration or hyperalimentation dysphagia, requiring feeding tube, IV hydration or | support, or perforation ted to radiation. complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or perforation complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Fistula-pharyngeal | none | - | - | present | requiring surgery |
| Fistula-rectal/anal | none | - | - | present | requiring surgery |
| Flatulence | none | mild | moderate | - | - |
| Gastric ulcer<br>(requires radiographic or<br>endoscopic documentation) | none | - | requiring medical<br>management or non-<br>surgical treatment | bleeding without<br>perforation, uncon-<br>trolled by outpatient<br>medical management;<br>requiring hospitalization<br>or surgery | perforation or bleeding,<br>requiring emergency<br>surgery |
| Also consider Hemorrhage/ble | eding with grade 3 or 4 | thrombocytopenia, Hemorr | hage/bleeding without grade | e 3 or 4 thrombocytopenia. | |
| Gastritis | none | - | requiring medical<br>management or non-<br>surgical treatment | uncontrolled by out-<br>patient medical<br>management; requiring<br>hospitalization or<br>surgery | life-threatening<br>bleeding, requiring<br>emergency surgery |
| Also consider Hemorrhage/ble | eding with grade 3 or 4 | thrombocytopenia, Hemorr | hage/bleeding without grade | e 3 or 4 thrombocytopenia. | |
| Hematemesis is graded in the l | HEMORRHAGE catego | ory. | | | |
| Hematochezia is graded in the | HEMORRHAGE categ | ory as Rectal bleeding/hem | atochezia. | | |
| Ileus (or neuroconstipation) | none | - | intermittent, not<br>requiring intervention | requiring non-surgical intervention | requiring surgery |
| | | | requiring intervention | intervention | |
| Mouth dryness | normal | mild | moderate | - | - |
| Mucositis Notes: Mucositis not due to rac | diation is graded in the ( | GASTROINTESTINAL cat<br>he RENAL/GENITOURIN | moderate | titis, Esophagitis, Gastritis, S | |
| Mucositis Notes: Mucositis not due to rac (oral/pharyngeal mucos | diation is graded in the ( | GASTROINTESTINAL cat<br>he RENAL/GENITOURIN | moderate egory for specific sites: Col. | titis, Esophagitis, Gastritis, S | |
| Mucositis Notes: Mucositis <u>not due to rac</u> (oral/pharyngeal mucos Radiation-related muco | diation is graded in the ditis), and Typhlitis; or t sitis is graded as Mucos | GASTROINTESTINAL cat<br>the RENAL/GENITOURINA<br>titis due to radiation. | moderate egory for specific sites: Col. ARY category for Vaginitis. patchy pseudomembra- nous reaction (patches generally ≤1.5 cm in diameter and non- | confluent pseudomembranous reaction (contiguous patches generally >1.5 cm in | necrosis or deep<br>ulceration; may include<br>bleeding not induced by<br>minor trauma or |
| Mucositis Notes: Mucositis not due to rac (oral/pharyngeal mucos Radiation-related muco Mucositis due to radiation | diation is graded in the ditis), and Typhlitis; or t sitis is graded as Mucos none | GASTROINTESTINAL cat<br>the RENAL/GENITOURINA<br>titis due to radiation. | moderate egory for specific sites: Col. ARY category for Vaginitis. patchy pseudomembra- nous reaction (patches generally ≤1.5 cm in diameter and non- | confluent pseudomembranous reaction (contiguous patches generally >1.5 cm in | necrosis or deep<br>ulceration; may include<br>bleeding not induced by<br>minor trauma or |
| Mucositis Notes: Mucositis <u>not due to rac</u> (oral/pharyngeal mucos Radiation-related muco Mucositis due to radiation Also consider Pain due to radia Notes: Grade radiation mucosi | diation is graded in the ditis), and Typhlitis; or t sitis is graded as Mucos none | GASTROINTESTINAL cat<br>the RENAL/GENITOURINA<br>sitis due to radiation.<br>erythema of the mucosa | moderate egory for specific sites: Col. ARY category for Vaginitis. patchy pseudomembra- nous reaction (patches generally ≤1.5 cm in diameter and non- contiguous) | confluent pseudomembranous reaction (contiguous patches generally >1.5 cm in | necrosis or deep<br>ulceration; may include<br>bleeding not induced by<br>minor trauma or<br>abrasion |
| Mucositis Notes: Mucositis <u>not due to rac</u> (oral/pharyngeal mucos Radiation-related muco Mucositis due to radiation Also consider Pain due to radia Notes: Grade radiation mucosi Dysphagia related to rac | diation is graded in the ditis), and Typhlitis; or t sitis is graded as Mucos none | GASTROINTESTINAL cat<br>the RENAL/GENITOURINA<br>sitis due to radiation.<br>erythema of the mucosa | moderate egory for specific sites: Col. ARY category for Vaginitis. patchy pseudomembra- nous reaction (patches generally ≤1.5 cm in diameter and non- contiguous) | confluent pseudomembranous reaction (contiguous patches generally >1.5 cm in diameter) | necrosis or deep<br>ulceration; may include<br>bleeding not induced by<br>minor trauma or<br>abrasion |
| Mucositis Notes: Mucositis <u>not due to rac</u> (oral/pharyngeal mucos Radiation-related mucos Mucositis due to radiation Also consider Pain due to radia Notes: Grade radiation mucosi Dysphagia related to rac the site of treatment. Nausea Pancreatitis | diation is graded in the ditis), and Typhlitis; or to sitis is graded as Mucos none ation. tis of the larynx here. diation is also graded as | GASTROINTESTINAL cat<br>the RENAL/GENITOURINA<br>sitis due to radiation. erythema of the mucosa either Dysphagia-esophage | moderate egory for specific sites: Col- ARY category for Vaginitis. patchy pseudomembra- nous reaction (patches generally ≤1.5 cm in diameter and non- contiguous) al related to radiation or Dy oral intake significantly | confluent pseudomembranous reaction (contiguous patches generally >1.5 cm in diameter) sphagia-pharyngeal related to no significant intake, | necrosis or deep<br>ulceration; may include<br>bleeding not induced by<br>minor trauma or<br>abrasion |
| Mucositis Notes: Mucositis not due to rac (oral/pharyngeal mucos Radiation-related muco Mucositis due to radiation Also consider Pain due to radia Notes: Grade radiation mucosi Dysphagia related to rac the site of treatment. | diation is graded in the ditis), and Typhlitis; or to sitis is graded as Mucos none ation. tis of the larynx here. diation is also graded as none | GASTROINTESTINAL cat<br>the RENAL/GENITOURINA<br>sitis due to radiation. erythema of the mucosa either Dysphagia-esophage | moderate egory for specific sites: Col- ARY category for Vaginitis. patchy pseudomembra- nous reaction (patches generally ≤1.5 cm in diameter and non- contiguous) al related to radiation or Dy oral intake significantly | confluent pseudomembranous reaction (contiguous patches generally >1.5 cm in diameter) sphagia-pharyngeal related to no significant intake, requiring IV fluids abdominal pain with pancreatic enzyme | necrosis or deep ulceration; may include bleeding not induced by minor trauma or abrasion or radiation, depending on complicated by shock (acute circulatory |
| Mucositis Notes: Mucositis not due to rac (oral/pharyngeal mucos Radiation-related muco Mucositis due to radiation Also consider Pain due to radia Notes: Grade radiation mucosi Dysphagia related to rac the site of treatment. Nausea Pancreatitis | diation is graded in the dittis), and Typhlitis; or t sittis is graded as Mucos none ation. tis of the larynx here. diation is also graded as none none | GASTROINTESTINAL cathe RENAL/GENITOURINAtitis due to radiation. erythema of the mucosa either Dysphagia-esophage able to eat | moderate egory for specific sites: Col- ARY category for Vaginitis. patchy pseudomembra- nous reaction (patches generally ≤1.5 cm in diameter and non- contiguous) al related to radiation or Dy oral intake significantly | confluent pseudomembranous reaction (contiguous patches generally >1.5 cm in diameter) sphagia-pharyngeal related to no significant intake, requiring IV fluids abdominal pain with pancreatic enzyme | necrosis or deep ulceration; may include bleeding not induced by minor trauma or abrasion or radiation, depending on complicated by shock (acute circulatory |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Proctitis | none | increased stool<br>frequency, occasional<br>blood-streaked stools or<br>rectal discomfort<br>(including hemorrhoids)<br>not requiring<br>medication | increased stool<br>frequency, bleeding,<br>mucus discharge, or<br>rectal discomfort<br>requiring medication;<br>anal fissure | increased stool fre-<br>quency/diarrhea requir-<br>ing parenteral support;<br>rectal bleeding requir-<br>ing transfusion; or per-<br>sistent mucus discharge,<br>necessitating pads | perforation, bleeding or<br>necrosis or other life-<br>threatening<br>complication requiring<br>surgical intervention<br>(e.g., colostomy) |
| Also consider Hemorrhage/ble | eeding with grade 3 or 4 | thrombocytopenia, Hemorr | hage/bleeding without grade | e 3 or 4 thrombocytopenia, l | Pain due to radiation. |
| Notes: Fistula is graded separa | ately as Fistula-rectal/an | al. | | | |
| Proctitis occurring mor<br>Appendix IV) | e than 90 days after the | start of radiation therapy is | graded in the RTOG/EORTO | C Late Radiation Morbidity | Scoring Scheme. (See |
| Salivary gland changes | none | slightly thickened<br>saliva; may have<br>slightly altered taste<br>(e.g., metallic);<br>additional fluids may be<br>required | thick, ropy, sticky<br>saliva; markedly altered<br>taste; alteration in diet<br>required | - | acute salivary gland<br>necrosis |
| Sense of smell | normal | slightly altered | markedly altered | - | - |
| Stomatitis/pharyngitis<br>(oral/pharyngeal mucositis) | none | painless ulcers,<br>erythema, or mild<br>soreness in the absence<br>of lesions | painful erythema,<br>edema, or ulcers, but<br>can eat or swallow | painful erythema,<br>edema, or ulcers<br>requiring IV hydration | severe ulceration or<br>requires parenteral or<br>enteral nutritional<br>support or prophylactic<br>intubation |
| For BMT studies, if specified in the protocol. | none | painless ulcers,<br>erythema, or mild<br>soreness in the absence<br>of lesions | painful erythema,<br>edema or ulcers but can<br>swallow | painful crythema,<br>edema, or ulcers<br>preventing swallowing<br>or requiring hydration<br>or parenteral (or enteral)<br>nutritional support | severe ulceration<br>requiring prophylactic<br>intubation or resulting<br>in documented<br>aspiration pneumonia |
| Note: Radiation-related mucos | sitis is graded as Mucos | itis due to radiation. | | | |
| Taste disturbance<br>(dysgeusia) | normal | slightly altered | markedly altered | - | - |
| Typhlitis<br>(inflammation of the cecum) | none | - | - | abdominal pain,<br>diarrhea, fever, and<br>radiographic or biopsy<br>documentation | perforation, bleeding or<br>necrosis or other life-<br>threatening<br>complication requiring<br>surgical intervention<br>(e.g., colostomy) |
| Also consider Hemorrhage/blo<br>neutropenia. | eeding with grade 3 or 4 | thrombocytopenia, Hemorr | hage/bleeding without grade | e 3 or 4 thrombocytopenia, I | Hypotension, Febrile |
| Vomiting | none | 1 episode in 24 hours<br>over pretreatment | 2-5 episodes in 24 hours<br>over pretreatment | ≥6 episodes in 24 hours<br>over pretreatment; or<br>need for IV fluids | requiring parenteral<br>nutrition; or physiologiconsequences requiring<br>intensive care;<br>hemodynamic collapse |
| Also consider Dehydration. | | | | | |
| Weight gain is graded in the C | CONSTITUTIONAL SY | MPTOMS category. | | | |
| Weight loss is graded in the C | ONSTITUTIONAL SY | MPTOMS category. | | | |
| Gastrointestinal - Other<br>(Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

Paclitaxel CA139387 BMS-181339 Clinical Protocol

> CTC Version 2.0 Publish Date: April 30, 1999

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| HEMORRHAGE | | | | | |
| Notes: Transfusion in this section refers to pRBC infusion. | | | | | |
| For any bleeding with grade 3 or 4 platelets (<50,000), always grade Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia. Also consider Platelets, Transfusion: pRBCs, and Transfusion: platelets in addition to grading severity by grading the site or type of bleeding. | | | | | |
| | sis, Hemorrhage/bleedi | | at incorporates the site of ble<br>wer GI bleeding, Petechiae/p | | |
| | | | de the specific site. If the sit<br>nia and specify the site or typ | | e platelet count is |
| Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia | none | mild without<br>transfusion | | requiring transfusion | catastrophic bleeding,<br>requiring major non-<br>elective intervention |
| Also consider Platelets, Hemog (Specify site,). | globin, Transfusion: pla | telets, Transfusion: pRBCs, | site or type of bleeding. If t | the site is not listed, grade as | s Hemorrhage-Other |
| Note: This adverse event must | t be graded for any blee | ding with grade 3 or 4 throi | nbocytopenia. | | |
| Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia | none | mild without<br>transfusion | | requiring transfusion | catastrophic bleeding<br>requiring major non-<br>elective intervention |
| Also consider Platelets, Hemog | globin, Transfusion: pla | telets, Transfusion: pRBCs, | Hemorrhage - Other (Speci | fy site,). | |
| Note: Bleeding in the absence<br>HEMORRHAGE category | | ocytopenia is graded here o<br>r in the HEMORRHAGE ca | | e of bleeding is not listed els | ewhere in the |
| CNS hemorrhage/bleeding | none | - | - | bleeding noted on CT or<br>other scan with no<br>clinical consequences | hemorrhagic stroke or<br>hemorrhagic vascular<br>event (CVA) with<br>neurologic signs and<br>symptoms |
| Epistaxis | none | mild without<br>transfusion | - | requiring transfusion | catastrophic bleeding,<br>requiring major non-<br>elective intervention |
| Hematemesis | none | mild without<br>transfusion | - | requiring transfusion | catastrophic bleeding,<br>requiring major non-<br>elective intervention |
| Hematuria<br>(in the absence of vaginal<br>bleeding) | none | microscopic only | intermittent gross<br>bleeding, no clots | persistent gross<br>bleeding or clots; may<br>require catheterization<br>or instrumentation, or<br>transfusion | open surgery or necrosis<br>or deep bladder<br>ulceration |
| Hemoptysis | none | mild without<br>transfusion | | requiring transfusion | catastrophic bleeding,<br>requiring major non-<br>elective intervention |
| Hemorrhage/bleeding associated with surgery | none | mild without<br>transfusion | - | requiring transfusion | catastrophic bleeding,<br>requiring major non-<br>elective intervention |
| Note: Expected blood loss at th | e time of surgery is not | graded as an adverse event | - | | |
| Melena/GI bleeding | none | mild without<br>transfusion | - | requiring transfusion | catastrophic bleeding,<br>requiring major non-<br>elective intervention |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| | | G | rade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Petechiae/purpura<br>(hemorrhage/bleeding into<br>skin or mucosa) | none | rare petechiae of skin | petechiae or purpura in<br>dependent areas of skin | generalized petechiae or<br>purpura of skin or<br>petechiae of any<br>mucosal site | - |
| Rectal bleeding/<br>hematochezia | none | mild without<br>transfusion or<br>medication | persistent, requiring<br>medication (e.g., steroid<br>suppositories) and/or<br>break from radiation<br>treatment | requiring transfusion | catastrophic bleeding,<br>requiring major non-<br>elective intervention |
| Vaginal bleeding | none | spotting, requiring <2<br>pads per day | requiring ≥2 pads per<br>day, but not requiring<br>transfusion | requiring transfusion | catastrophic bleeding,<br>requiring major non-<br>elective intervention |
| Hemorrhage - Other (Specify site,) | none | mild without<br>transfusion | - | requiring transfusion | catastrophic bleeding,<br>requiring major non-<br>elective intervention |
| | | НЕР | PATIC | | |
| Alkaline phosphatase | WNL | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Bilirubin | WNL | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN |
| Bilirubin associated with<br>graft versus host disease<br>(GVHD) for BMT studies, if<br>specified in the protocol. | normal | ≥2 - <3 mg/100 mL | ≥3 - <6 mg/100 mL | ≥6 - <15 mg/100 mL | ≥15 mg/100 mL |
| GGT<br>(γ - Glutamyl transpeptidase) | WNL | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Hepatic enlargement | absent | - | - | present | - |
| Note: Grade Hepatic enlargem | ent only for treatr | nent related adverse event includ | ing Veno-Occlusive Disease | | |
| Hypoalbuminemia | WNL | <lln -="" 3="" dl<="" g="" td=""><td>≥2 - &lt;3 g/dL</td><td>&lt;2 g/dL</td><td>-</td></lln> | ≥2 - <3 g/dL | <2 g/dL | - |
| Liver dysfunction/ failure (clinical) | normal | - | - | asterixis | encephalopathy or coma |
| Portal vein flow | normal | - | decreased portal vein flow | reversal/retrograde<br>portal vein flow | - |
| SGOT (AST)<br>(serum glutamic oxaloacetic<br>transaminase) | WNL | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| SGPT (ALT)<br>(serum glutamic pyruvic<br>transaminase) | WNL | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Hepatic - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | INFECTION/FEBR | ILE NEUTROPE | NIA | |
| Catheter-related infection | none | mild, no active<br>treatment | moderate, localized<br>infection, requiring<br>local or oral treatment | severe, systemic<br>infection, requiring IV<br>antibiotic or antifungal<br>treatment or<br>hospitalization | life-threatening sepsis<br>(e.g., septic shock) |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

CA139387

| | | G | rade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Febrile neutropenia<br>(fever of unknown origin<br>without clinically or<br>microbiologically<br>documented infection) | none | - | - | Present | Life-threatening sepsis<br>(e.g., septic shock) |
| (ANC <1.0 x 10 <sup>9</sup> /L, fever ≥38.5°C) | | | | | |
| Also consider Neutrophils. | | | | | |
| Note: Hypothermia instead of | f fever may be associa | ted with neutropenia and is g | raded here. | | |
| Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia | none | - | - | present | life-threatening sepsis<br>(e.g., septic shock) |
| (ANC <1.0 x 10 <sup>9</sup> /L) | | | | | |
| Also consider Neutrophils. | | | | | |
| Notes: Hypothermia instead o | of fever may be associ | ated with neutropenia and is g | graded here. | | |
| In the absence of docu | mented infection grad | le 3 or 4 neutropenia with fev | er is graded as Febrile neutro | ppenia. | |
| Infection with unknown ANC | none | - | - | present | life-threatening sepsis<br>(e.g., septic shock) |
| Note: This adverse event crite | erion is used in the rar | e case when ANC is unknown | 1. | | |
| Infection without neutropenia | none | mild, no active<br>treatment | moderate, localized<br>infection, requiring<br>local or oral treatment | severe, systemic<br>infection, requiring IV<br>antibiotic or antifungal<br>treatment, or<br>hospitalization | life-threatening sepsis<br>(e.g., septic shock) |
| Also consider Neutrophils. | | | | | |
| Wound-infectious is graded in | the DERMATOLOG | GY/SKIN category. | | | |
| Infection/Febrile Neutropenia - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | LYMP | HATICS | | |
| Lymphatics | normal | mild lymphedema | moderate lymphedema<br>requiring compression;<br>lymphocyst | severe lymphedema<br>limiting function;<br>lymphocyst requiring<br>surgery | severe lymphedema<br>limiting function with<br>ulceration |
| Lymphatics - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | METABOLIC/ | LABORATORY | | |
| Acidosis<br>(metabolic or respiratory) | normal | pH <normal, but="" td="" ≥7.3<=""><td>-</td><td>pH &lt;7.3</td><td>pH &lt;7.3 with life-<br/>threatening physiologic<br/>consequences</td></normal,> | - | pH <7.3 | pH <7.3 with life-<br>threatening physiologic<br>consequences |
| Alkalosis<br>(metabolic or respiratory) | normal | pH >normal, but ≤7.5 | - | pH >7.5 | pH >7.5 with life-<br>threatening physiologic<br>consequences |
| Amylase | WNL | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN |
| Bicarbonate | WNL | <lln -="" 16="" dl<="" meq="" td=""><td>11 - 15 mEq/dL</td><td>8 - 10 mEq/dL</td><td>&lt;8 mEq/dL</td></lln> | 11 - 15 mEq/dL | 8 - 10 mEq/dL | <8 mEq/dL |


Revised March 23, 1998

| | Grade | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| CPK<br>(creatine phosphokinase) | WNL | >ULN - 2.5 x ULN | >2.5 - 5 x ULN | >5 - 10 x ULN | >10 x ULN |
| Hypercalcemia | WNL | >ULN - 11.5 mg/dL<br>>ULN - 2.9 mmol/L | >11.5 - 12.5 mg/dL<br>>2.9 - 3.1 mmol/L | >12.5 - 13.5 mg/dL<br>>3.1 - 3.4 mmol/L | >13.5 mg/dL<br>>3.4 mmol/L |
| Hypercholesterolemia | WNL | >ULN - 300 mg/dL<br>>ULN - 7.75 mmol/L | >300 - 400 mg/dL<br>>7.75 - 10.34 mmol/L | >400 - 500 mg/dL<br>>10.34 - 12.92 mmol/L | >500 mg/dL<br>>12.92 mmol/L |
| Hyperglycemia | WNL | >ULN - 160 mg/dL<br>>ULN - 8.9 mmol/L | >160 - 250 mg/dL<br>>8.9 - 13.9 mmol/L | >250 - 500 mg/dL<br>>13.9 - 27.8 mmol/L | >500 mg/dL<br>>27.8 mmol/L or<br>acidosis |
| Hyperkalemia | WNL | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L | >7.0 mmol/L |
| Hypermagnesemia | WNL | >ULN - 3.0 mg/dL<br>>ULN - 1.23 mmol/L | - | >3.0 - 8.0 mg/dL<br>>1.23 - 3.30 mmol/L | >8.0 mg/dL<br>>3.30 mmol/L |
| Hypernatremia | WNL | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L | >160 mmol/L |
| Hypertriglyceridemia | WNL | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 10 x ULN | >10 x ULN |
| Hyperuricemia | WNL | >ULN - ≤10 mg/dL<br>≤0.59 mmol/L without<br>physiologic<br>consequences | - | >ULN - ≤10 mg/dL<br>≤0.59 mmol/L with<br>physiologic<br>consequences | >10 mg/dL<br>>0.59 mmol/L |
| Also consider Tumor lysis s | yndrome, Renal fai | lure, Creatinine, Hyperkalemia. | | | |
| Hypocalcemia | WNL | <lln -="" 8.0="" dl<br="" mg=""><lln -="" 2.0="" l<="" mmol="" td=""><td>7.0 - &lt;8.0 mg/dL<br/>1.75 - &lt;2.0 mmol/L</td><td>6.0 - &lt;7.0 mg/dL<br/>1.5 - &lt;1.75 mmol/L</td><td>&lt;6.0 mg/dL<br/>&lt;1.5 mmol/L</td></lln></lln> | 7.0 - <8.0 mg/dL<br>1.75 - <2.0 mmol/L | 6.0 - <7.0 mg/dL<br>1.5 - <1.75 mmol/L | <6.0 mg/dL<br><1.5 mmol/L |
| Hypoglycemia | WNL | <lln -="" 55="" dl<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>40 - &lt;55 mg/dL<br/>2.2 - &lt;3.0 mmol/L</td><td>30 - &lt;40 mg/dL<br/>1.7 - &lt;2.2 mmol/L</td><td>&lt;30 mg/dL<br/>&lt;1.7 mmol/L</td></lln></lln> | 40 - <55 mg/dL<br>2.2 - <3.0 mmol/L | 30 - <40 mg/dL<br>1.7 - <2.2 mmol/L | <30 mg/dL<br><1.7 mmol/L |
| Hypokalemia | WNL | <lln -="" 3.0="" l<="" mmol="" td=""><td>-</td><td>2.5 - &lt;3.0 mmol/L</td><td>&lt;2.5 mmol/L</td></lln> | - | 2.5 - <3.0 mmol/L | <2.5 mmol/L |
| Hypomagnesemia | WNL | <lln -="" 1.2="" dl<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>0.9 - &lt;1.2 mg/dL<br/>0.4 - &lt;0.5 mmol/L</td><td>0.7 - &lt;0.9 mg/dL<br/>0.3 - &lt;0.4 mmol/L</td><td>&lt;0.7 mg/dL<br/>&lt;0.3 mmol/L</td></lln></lln> | 0.9 - <1.2 mg/dL<br>0.4 - <0.5 mmol/L | 0.7 - <0.9 mg/dL<br>0.3 - <0.4 mmol/L | <0.7 mg/dL<br><0.3 mmol/L |
| Hyponatremia | WNL | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>120 - &lt;130 mmol/L</td><td>&lt;120 mmol/L</td></lln> | - | 120 - <130 mmol/L | <120 mmol/L |
| Hypophosphatemia | WNL | <lln -2.5="" dl<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>≥2.0 - &lt;2.5 mg/dL<br/>≥0.6 - &lt;0.8 mmol/L</td><td>≥1.0 - &lt;2.0 mg/dL<br/>≥0.3 - &lt;0.6 mmol/L</td><td>&lt;1.0 mg/dL<br/>&lt;0.3 mmol/L</td></lln></lln> | ≥2.0 - <2.5 mg/dL<br>≥0.6 - <0.8 mmol/L | ≥1.0 - <2.0 mg/dL<br>≥0.3 - <0.6 mmol/L | <1.0 mg/dL<br><0.3 mmol/L |
| Hypothyroidism is graded in | the ENDOCRINE | category. | | | |
| Lipase | WNL | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN |
| Metabolic/Laboratory -<br>Other (Specify, | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | MUSCULO | SKELETAL | | |
| Arthralgia is graded in the P | AIN category. | | | | |
| Arthritis | none | mild pain with<br>inflammation, crythema<br>or joint swelling but not<br>interfering with<br>function | moderate pain with<br>inflammation,<br>erythema, or joint<br>swelling interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain with<br>inflammation,<br>erythema, or joint<br>swelling and interfering<br>with activities of daily<br>living | disabling |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Muscle weakness<br>(not due to neuropathy) | normal | asymptomatic with<br>weakness on physical<br>exam | symptomatic and<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | symptomatic and<br>interfering with<br>activities of daily living | bedridden or disabling |
| Myalgia [tenderness or pain in | muscles] is grade | ed in the PAIN category. | | | |
| Myositis<br>(inflammation/damage of<br>muscle) | none | mild pain, not<br>interfering with<br>function | pain interfering with<br>function, but not<br>interfering with<br>activities of daily living | pain interfering with<br>function and interfering<br>with activities of daily<br>living | bedridden or disabling |
| Also consider CPK. | | | | | |
| Note: Myositis implies muscle | damage (i.e., ele | vated CPK). | | | |
| Osteonecrosis<br>(avascular necrosis) | none | asymptomatic and<br>detected by imaging<br>only | symptomatic and<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | symptomatic and<br>interfering with<br>activities of daily living | symptomatic; or<br>disabling |
| Musculoskeletal - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | NEURO | DLOGY | | |
| Aphasia, receptive and/or exp | ressive, is graded | under Speech impairment in the N | | | |
| Arachnoiditis/meningismus/<br>radiculitis | absent | mild pain not interfering with function | moderate pain<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | severe pain interfering<br>with activities of daily<br>living | unable to function or<br>perform activities of<br>daily living; bedridden<br>paraplegia |
| Also consider Headache, Vom | iting, Fever. | | | | |
| Ataxia (incoordination) | normal | asymptomatic but<br>abnormal on physical<br>exam, and not<br>interfering with<br>function | mild symptoms<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | moderate symptoms<br>interfering with<br>activities of daily living | bedridden or disabling |
| CNS cerebrovascular ischemia | none | - | - | transient ischemic event<br>or attack (TIA) | permanent event (e.g.,<br>cerebral vascular<br>accident) |
| CNS hemorrhage/bleeding is § | graded in the HEN | MORRHAGE category. | | | |
| Cognitive disturbance/<br>learning problems | none | cognitive disability; not<br>interfering with<br>work/school<br>performance;<br>preservation of<br>intelligence | cognitive disability;<br>interfering with<br>work/school<br>performance; decline of<br>1 SD (Standard<br>Deviation) or loss of<br>developmental<br>milestones | cognitive disability;<br>resulting in significant<br>impairment of<br>work/school<br>performance; cognitive<br>decline >2 SD | inability to work/frank<br>mental retardation |


Revised March 23, 1998

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Confusion | normal | confusion or<br>disorientation or<br>attention deficit of brief<br>duration; resolves<br>spontaneously with no<br>sequelae | confusion or<br>disorientation or<br>attention deficit<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | confusion or delirium<br>interfering with<br>activities of daily living | harmful to others or<br>self; requiring<br>hospitalization |
| Cranial neuropathy is graded | in the NEUROLOGY | category as Neuropathy-crani | al. | | |
| Delusions | normal | - | - | present | toxic psychosis |
| Depressed level of consciousness | normal | somnolence or sedation<br>not interfering with<br>function | somnolence or sedation<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | obtundation or stupor;<br>difficult to arouse;<br>interfering with<br>activities of daily living | coma |
| Note: Syncope (fainting) is gr | raded in the NEUROI | LOGY category. | | | |
| Dizziness/lightheadedness | none | not interfering with function | interfering with<br>function, but not<br>interfering with<br>activities of daily living | interfering with activities of daily living | bedridden or disabling |
| Dysphasia, receptive and/or e | expressive, is graded u | nder Speech impairment in the | NEUROLOGY category. | | |
| Extrapyramidal/<br>involuntary movement/<br>restlessness | none | mild involuntary<br>movements not<br>interfering with<br>function | moderate involuntary<br>movements interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe involuntary<br>movements or torticollis<br>interfering with<br>activities of daily living | bedridden or disabling |
| Hallucinations | normal | - | - | present | toxic psychosis |
| Headache is graded in the PA | IN category. | | | | |
| Insomnia | normal | occasional difficulty<br>sleeping not interfering<br>with function | difficulty sleeping<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | frequent difficulty<br>sleeping, interfering<br>with activities of daily<br>living | - |
| Note: This adverse event is g | raded when insomnia | is related to treatment. If pain | or other symptoms interfere | with sleep do NOT grade as | insomnia. |
| Irritability<br>(children <3 years of age) | normal | mild; easily consolable | moderate; requiring increased attention | severe; inconsolable | - |
| Leukoencephalopathy<br>associated radiological<br>findings | none | mild increase in SAS (subarachnoid space) and/or mild ventriculomegaly; and/or small (+/- multiple) focal T2 hyperintensities, involving periventricular white matter or <1/3 of susceptible areas of cerebrum | moderate increase in SAS; and/or moderate ventriculomegaly; and/or focal T2 hyperintensities extending into centrum ovale; or involving 1/3 to 2/3 of susceptible areas of cerebrum | severe increase in SAS;<br>severe<br>ventriculomegaly; near<br>total white matter T2<br>hyperintensities or<br>diffuse low attenuation<br>(CT); focal white matter<br>necrosis (cystic) | severe increase in SAS;<br>severe<br>ventriculomegaly;<br>diffuse low attenuation<br>with calcification (CT);<br>diffuse white matter<br>necrosis (MRI) |
| Memory loss | normal | memory loss not<br>interfering with<br>function | memory loss interfering<br>with function, but not<br>interfering with<br>activities of daily living | memory loss interfering<br>with activities of daily<br>living | amnesia |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Mood alteration-anxiety, agitation | normal | mild mood alteration<br>not interfering with<br>function | moderate mood<br>alteration interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe mood alteration<br>interfering with<br>activities of daily living | suicidal ideation or<br>danger to self |
| Mood alteration-depression | normal | mild mood alteration<br>not interfering with<br>function | moderate mood<br>alteration interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe mood alteration<br>interfering with<br>activities of daily living | suicidal ideation or<br>danger to self |
| Mood alteration-euphoria | normal | mild mood alteration<br>not interfering with<br>function | moderate mood<br>alteration interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe mood alteration<br>interfering with<br>activities of daily living | danger to self |
| Neuropathic pain is graded in | the PAIN category. | | | | |
| Neuropathy-cranial | absent | - | present, not interfering<br>with activities of daily<br>living | present, interfering with activities of daily living | life-threatening,<br>disabling |
| Neuropathy-motor | normal | subjective weakness but<br>no objective findings | mild objective<br>weakness interfering<br>with function, but not<br>interfering with<br>activities of daily living | objective weakness<br>interfering with<br>activities of daily living | paralysis |
| Neuropathy-sensory | normal | loss of deep tendon<br>reflexes or paresthesia<br>(including tingling) but<br>not interfering with<br>function | objective sensory loss<br>or paresthesia<br>(including tingling),<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | sensory loss or<br>paresthesia interfering<br>with activities of daily<br>living | permanent sensory loss<br>that interferes with<br>function |
| Nystagmus | absent | present | - | - | - |
| Also consider Vision-double v | vision. | | | | |
| Personality/behavioral | normal | change, but not<br>disruptive to patient or<br>family | disruptive to patient or family | disruptive to patient and<br>family; requiring mental<br>health intervention | harmful to others or<br>self; requiring<br>hospitalization |
| Pyramidal tract dysfunction<br>(e.g., ↑ tone, hyperreflexia,<br>positive Babinski, ↓ fine<br>motor coordination) | normal | asymptomatic with<br>abnormality on physical<br>examination | symptomatic or<br>interfering with<br>function but not<br>interfering with<br>activities of daily living | interfering with<br>activities of daily living | bedridden or disabling;<br>paralysis |
| Seizure(s) | none | - | seizure(s) self-limited<br>and consciousness is<br>preserved | seizure(s) in which<br>consciousness is altered | seizures of any type<br>which are prolonged,<br>repetitive, or difficult to<br>control (e.g., status<br>epilepticus, intractable<br>epilepsy) |
| Speech impairment<br>(e.g., dysphasia or aphasia) | normal | - | awareness of receptive<br>or expressive dysphasia,<br>not impairing ability to<br>communicate | receptive or expressive<br>dysphasia, impairing<br>ability to communicate | inability to communicate |
| Syncope (fainting) | absent | - | - | present | - |
| Also consider CAPDIOVASC | THE AR CARRHYTHM | IIA) Vasovagal enisode CN | S cerebrovascular ischemia. | | |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Tremor | none | mild and brief or<br>intermittent but not<br>interfering with<br>function | moderate tremor<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | severe tremor<br>interfering with<br>activities of daily living | - |
| Vertigo | none | not interfering with function | interfering with<br>function, but not<br>interfering with<br>activities of daily living | interfering with activities of daily living | bedridden or disabling |
| Neurology - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | OCULAR | R/VISUAL | | |
| Cataract | none | asymptomatic | symptomatic, partial<br>visual loss | symptomatic, visual<br>loss requiring treatment<br>or interfering with<br>function | - |
| Conjunctivitis | none | abnormal ophthalmologic changes, but asymptomatic or symptomatic without visual impairment (i.e., pain and irritation) | symptomatic and<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | symptomatic and<br>interfering with<br>activities of daily living | - |
| Dry eye | normal | mild, not requiring treatment | moderate or requiring artificial tears | - | - |
| Glaucoma | none | increase in intraocular<br>pressure but no visual<br>loss | increase in intraocular<br>pressure with retinal<br>changes | visual impairment | unilateral or bilateral<br>loss of vision<br>(blindness) |
| Keratitis<br>(corneal inflammation/<br>corneal ulceration) | none | abnormal<br>ophthalmologic changes<br>but asymptomatic or<br>symptomatic without<br>visual impairment (i.e.,<br>pain and irritation) | symptomatic and<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | symptomatic and<br>interfering with<br>activities of daily living | unilateral or bilateral<br>loss of vision<br>(blindness) |
| Tearing (watery eyes) | none | mild: not interfering<br>with function | moderate: interfering<br>with function, but not<br>interfering with<br>activities of daily living | interfering with activities of daily living | - |
| Vision-blurred vision | normal | - | symptomatic and<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | symptomatic and<br>interfering with<br>activities of daily living | - |
| Vision-double vision<br>(diplopia) | normal | - | symptomatic and<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | symptomatic and<br>interfering with<br>activities of daily living | - |
| Vision-flashing<br>lights/floaters | normal | mild, not interfering<br>with function | symptomatic and<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | symptomatic and<br>interfering with<br>activities of daily living | - |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Vision-night blindness<br>(nyctalopia) | normal | abnormal electro-<br>retinography but<br>asymptomatic | symptomatic and<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | symptomatic and<br>interfering with<br>activities of daily living | - |
| Vision-photophobia | normal | - | symptomatic and<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | symptomatic and<br>interfering with<br>activities of daily living | - |
| Ocular/Visual - Other (Specify,) | normal | mild | moderate | severe | unilateral or bilateral<br>loss of vision<br>(blindness) |
| | | PA | IN | | |
| Abdominal pain or cramping | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Arthralgia<br>(joint pain) | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Arthritis (joint pain with clinic | al signs of inflammatio | n) is graded in the MUSCUI | LOSKELETAL category. | | |
| Bone pain | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Chest pain<br>(non-cardiac and non-<br>pleuritic) | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Dysmenorrhea | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Dyspareunia | none | mild pain not interfering with function | moderate pain interfering with sexual activity | severe pain preventing sexual activity | - |
| Dysuria is graded in the RENA | AL/GENITOURINARY | category. | | | |
| Earache (otalgia) | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Headache | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |


Revised March 23, 1998

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Hepatic pain | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Myalgia<br>(muscle pain) | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Neuropathic pain<br>(e.g., jaw pain, neurologic<br>pain, phantom limb pain,<br>post-infectious neuralgia, or<br>painful neuropathies) | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Pain due to radiation | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Pelvic pain | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Pleuritic pain | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Rectal or perirectal pain<br>(proctalgia) | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Tumor pain<br>(onset or exacerbation of<br>tumor pain due to treatment) | none | mild pain not interfering with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Tumor flare is graded in the SY | YNDROME category. | | | | |
| Pain - Other<br>(Specify,) | none | mild | moderate | severe | disabling |
| | PULMONARY | | | | |
| Adult Respiratory Distress<br>Syndrome (ARDS) | absent | - | - | - | present |
| Apnea | none | - | - | present | requiring intubation |


Revised March 23, 1998

23

| | | Gr | rade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Carbon monoxide diffusion capacity (DL <sub>CO</sub> ) | ≥90% of pretreatment or normal value | ≥75 - <90% of<br>pretreatment or normal<br>value | ≥50 - <75% of<br>pretreatment or normal<br>value | ≥25 - <50% of<br>pretreatment or normal<br>value | <25% of pretreatment<br>or normal value |
| Cough | absent | mild, relieved by non-<br>prescription medication | requiring narcotic antitussive | severe cough or<br>coughing spasms,<br>poorly controlled or<br>unresponsive to<br>treatment | - |
| Dyspnea (shortness of breath) | normal | - | dyspnea on exertion | dyspnea at normal level of activity | dyspnea at rest or<br>requiring ventilator<br>support |
| FEV <sub>1</sub> | ≥90% of pretreatment or normal value | ≥75 - <90% of<br>pretreatment or normal<br>value | ≥50 - <75% of pretreatment or normal value | ≥25 - <50% of<br>pretreatment or normal<br>value | <25% of pretreatment<br>or normal value |
| Hiccoughs (hiccups, singultus) | none | mild, not requiring treatment | moderate, requiring treatment | severe, prolonged, and refractory to treatment | - |
| Нурохіа | normal | - | decreased O <sub>2</sub> saturation with exercise | decreased O <sub>2</sub> saturation<br>at rest, requiring<br>supplemental oxygen | decreased O <sub>2</sub> saturation<br>requiring pressure<br>support (CPAP) or<br>assisted ventilation |
| Pleural effusion<br>(non-malignant) | none | asymptomatic and not requiring treatment | symptomatic, requiring diuretics | symptomatic, requiring O <sub>2</sub> or therapeutic thoracentesis | life-threatening (e.g.,<br>requiring intubation) |
| Pleuritic pain is graded in the | PAIN category. | | | | |
| Pneumonitis/pulmonary infiltrates | none | radiographic changes<br>but asymptomatic or<br>symptoms not requiring<br>steroids | radiographic changes<br>and requiring steroids or<br>diuretics | radiographic changes<br>and requiring oxygen | radiographic changes<br>and requiring assisted<br>ventilation |
| Pneumothorax | none | no intervention required | chest tube required | sclerosis or surgery<br>required | life-threatening |
| Pulmonary embolism is grade | d as Thrombosis/embol | ism in the CARDIOVASCU | LAR (GENERAL) category | 7. | |
| Pulmonary fibrosis | none | radiographic changes,<br>but asymptomatic or<br>symptoms not requiring<br>steroids | requiring steroids or<br>diuretics | requiring oxygen | requiring assisted<br>ventilation |
| Note: Radiation-related pulmo | onary fibrosis is graded | in the RTOG/EORTC Late l | Radiation Morbidity Scoring | Scheme-Lung. (See Apper | ndix IV) |
| Voice changes/stridor/larynx<br>(e.g., hoarseness, loss of<br>voice, laryngitis) | normal | mild or intermittent<br>hoarseness | persistent hoarseness,<br>but able to vocalize;<br>may have mild to<br>moderate edema | whispered speech, not<br>able to vocalize; may<br>have marked edema | marked dyspnea/stridor<br>requiring tracheostomy<br>or intubation |
| Notes: Cough from radiation is | s graded as cough in the | e PULMONARY category. | | | |
| | | rynx is graded as Grade 4 M<br>graded as Grade 4 Hemopt | | | category. Radiation- |
| Pulmonary - Other<br>(Specify, ) | none | mild | moderate | severe | life-threatening or<br>disabling |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| | | Gı | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| RENAL/GENITOURINARY | | | | | |
| Bladder spasms | absent | mild symptoms, not<br>requiring intervention | symptoms requiring antispasmodic | severe symptoms<br>requiring narcotic | - |
| Creatinine | WNL | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 6.0 x ULN | >6.0 x ULN |
| Note: Adjust to age-approprie | ate levels for pediatric p | patients. | | | |
| Dysuria<br>(painful urination) | none | mild symptoms<br>requiring no<br>intervention | symptoms relieved with<br>therapy | symptoms not relieved<br>despite therapy | - |
| Fistula or GU fistula<br>(e.g., vaginal, vesicovaginal) | none | - | - | requiring intervention | requiring surgery |
| Hemoglobinuria | - | present | - | - | - |
| Hematuria (in the absence of | vaginal bleeding) is gra | ded in the HEMORRHAGE | category. | | |
| Incontinence | none | with coughing,<br>sneezing, etc. | spontaneous, some control | no control (in the absence of fistula) | - |
| Operative injury to bladder<br>and/or ureter | none | - | injury of bladder with<br>primary repair | sepsis, fistula, or<br>obstruction requiring<br>secondary surgery; loss<br>of one kidney; injury<br>requiring anastomosis<br>or re-implantation | septic obstruction of<br>both kidneys or<br>vesicovaginal fistula<br>requiring diversion |
| Proteinuria | normal or <0.15<br>g/24 hours | 1+ or 0.15 - 1.0 g/24<br>hours | 2+ to 3+ or 1.0 - 3.5<br>g/24 hours | 4+ or >3.5 g/24 hours | nephrotic syndrome |
| Note: If there is an inconsister | ncy between absolute v | alue and dip stick reading, us | se the absolute value for grad | ling. | |
| Renal failure | none | - | - | requiring dialysis, but reversible | requiring dialysis and irreversible |
| Ureteral obstruction | none | unilateral, not requiring surgery | - | bilateral, not requiring surgery | stent, nephrostomy<br>tube, or surgery |
| Urinary electrolyte wasting (e.g., Fanconi's syndrome, renal tubular acidosis) | none | asymptomatic, not requiring treatment | mild, reversible and<br>manageable with oral<br>replacement | reversible but requiring IV replacement | irreversible, requiring continued replacement |
| Also consider Acidosis, Bicar | bonate, Hypocalcemia, | Hypophosphatemia. | | | |
| Urinary frequency/urgency | normal | increase in frequency or<br>nocturia up to 2 x<br>normal | increase >2 x normal<br>but <hourly< td=""><td>hourly or more with<br/>urgency, or requiring<br/>catheter</td><td>-</td></hourly<> | hourly or more with<br>urgency, or requiring<br>catheter | - |
| Urinary retention | normal | hesitancy or dribbling,<br>but no significant<br>residual urine; retention<br>occurring during the<br>immediate<br>postoperative period | hesitancy requiring medication or occasional in/out catheterization (<4 x per week), or operative bladder atony requiring indwelling catheter beyond immediate postoperative period but for <6 weeks | requiring frequent in/out catheterization (≥4 x per week) or urological intervention (e.g., TURP, suprapubic tube, urethrotomy) | bladder rupture |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Urine color change<br>(not related to other dietary<br>or physiologic cause e.g.,<br>bilirubin, concentrated urine,<br>hematuria) | normal | asymptomatic, change<br>in urine color | - | - | - |
| Vaginal bleeding is graded in | the HEMORRHAC | E category. | | | |
| Vaginitis<br>(not due to infection) | none | mild, not requiring<br>treatment | moderate, relieved with treatment | severe, not relieved<br>with treatment, or<br>ulceration not requiring<br>surgery | ulceration requiring<br>surgery |
| Renal/Genitourinary - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | SECONDARY | MALIGNANCY | | |
| Secondary Malignancy - Other (Specify type,) excludes metastasis from initial primary | none | - | - | - | present |
| | \$ | SEXUAL/REPRODU | JCTIVE FUNCTI | ON | |
| Dyspareunia is graded in the F | PAIN category. | | | | |
| Dysmenorrhea is graded in the | PAIN category. | | | | |
| Erectile impotence | normal | mild (erections<br>impaired but<br>satisfactory) | moderate (erections<br>impaired, unsatisfactory<br>for intercourse) | no erections | - |
| | | _ | _ | sterile | - |
| Female sterility | normal | | | | |
| Female sterility Feminization of male is grade | | NE category. | | | |
| • | | NE category. occasionally irregular or lengthened interval, but continuing menstrual cycles | very irregular, but<br>continuing menstrual<br>cycles | persistent amenorrhea | - |
| Feminization of male is grade | d in the ENDOCRI | occasionally irregular or<br>lengthened interval, but<br>continuing menstrual | continuing menstrual | persistent amenorrhea | - |
| Feminization of male is graded<br>Irregular menses<br>(change from baseline) | d in the ENDOCRI | occasionally irregular or<br>lengthened interval, but<br>continuing menstrual<br>cycles | continuing menstrual cycles | | - |
| Feminization of male is grade<br>Irregular menses<br>(change from baseline) | d in the ENDOCRI normal normal | occasionally irregular or<br>lengthened interval, but<br>continuing menstrual<br>cycles<br>decrease in interest | continuing menstrual cycles severe loss of interest oligospermia | -<br>azoospermia | - |
| Feminization of male is grade<br>Irregular menses<br>(change from baseline)<br>Libido | d in the ENDOCRI normal normal | occasionally irregular or<br>lengthened interval, but<br>continuing menstrual<br>cycles<br>decrease in interest | continuing menstrual cycles severe loss of interest oligospermia | -<br>azoospermia | - |
| Feminization of male is graded Irregular menses (change from baseline) Libido Male infertility Masculinization of female is g | normal normal - craded in the ENDO | occasionally irregular or lengthened interval, but continuing menstrual cycles decrease in interest - OCRINE category. | continuing menstrual cycles severe loss of interest oligospermia (low sperm count) requiring treatment and/or interfering with sexual function, | -<br>azoospermia | disabling |
| Feminization of male is grade Irregular menses (change from baseline) Libido Male infertility Masculinization of female is g Vaginal dryness Sexual/Reproductive Function - Other | normal normal raded in the ENDO normal normal | occasionally irregular or lengthened interval, but continuing menstrual cycles decrease in interest - OCRINE category. mild | continuing menstrual cycles severe loss of interest oligospermia (low sperm count) requiring treatment and/or interfering with sexual function, dyspareunia moderate | - azoospermia (no sperm) - severe | - |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Autoimmune reactions are g | raded in the ALLERGY/ | IMMUNOLOGY category. | | | |
| DIC (disseminated intravasc | ular coagulation) is grad | ed in the COAGULATION of | category. | | |
| Fanconi's syndrome is grade | d as Urinary electrolyte | wasting in the RENAL/GEN | ITOURINARY category. | | |
| Renal tubular acidosis is gra | ded as Urinary electrolyt | e wasting in the RENAL/GE | NITOURINARY category. | | |
| Stevens-Johnson syndrome ( | erythema multiforme) is | graded in the DERMATOLO | OGY/SKIN category. | | |
| SIADH (syndrome of inappr | opriate antidiuretic horn | one) is graded in the ENDO | CRINE category. | | |
| Thrombotic microangiopath | y (e.g., thrombotic throm | bocytopenic purpura/TTP or | hemolytic uremic syndrome | e/HUS) is graded in the CO | AGULATION category. |
| Tumor flare | none | mild pain not interfering<br>with function | moderate pain; pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain; pain or<br>analgesics interfering<br>with function and<br>interfering with<br>activities of daily living | Disabling |
| Also consider Hypercalcemi | a. | | | | |
| Note: Tumor flare is characterized by a constellation of symptoms and signs in direct relation to initiation of therapy (e.g., anti-estrogens/androgens or additional hormones). The symptoms/signs include tumor pain, inflammation of visible tumor, hypercalcemia, diffuse bone pain, and other electrolyte disturbances. | | | | | |
| Tumor lysis syndrome | absent | - | - | present | - |
| Also consider Hyperkalemia | , Creatinine. | | | | |
| Urinary electrolyte wasting ( | e.g., Fanconi's syndrom | e, renal tubular acidosis) is g | raded in the RENAL/GENIT | OURINARY category. | |
| Syndromes - Other (Specify,) | none | mild | moderate | severe | life-threatening or disabling |


Date: 25-May-2005

Revised March 23, 1998

27

Paclitaxel CA139387 BMS-181339 Clinical Protocol

> CTC Version 2.0 Publish Date: April 30, 1999

# Appendix I Adverse Event Module

To be implemented at the request of the study sponsor or principal investigator in the protocol or by protocol amendment when more detailed information is considered pertinent.

| Adverse Event: | Date of Treatment: | | Course Number: |
|---|---|---|---|
| Date of onset: | | | Grade at onset: |
| Date of first change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Did adverse event resolve? If so, date of resolution of adverse event: | Yes | No | |
| Date of last observation (if prior to recovery): | | | |
| Reason(s) observations stopped (if prior to recovery): | | | |
| Was patient retreated? If yes, was treatment delayed for recovery? Date of next treatment? | Yes | No | |
| Dose reduced for next treatment? | Yes | No | |
| Additional Comments: | | | |
| If module is being activated for new adver | rse event not currently in G | CTC, please provi | de definitions for adverse event grading: |
| Grade 0 = | | | |
| Grade 1 = | | | |
| Grade 2 = | | | |
| Grade 3 = | | | |
| Grade 4 = | | | |


Revised March 23, 1998

Paclitaxel CA139387 Clinical Protocol BMS-181339

CTC Version 2.0 Publish Date: April 30, 1999

## Appendix II

#### Infection Module

| To<br>am | be implemented at the request of the study sponsor or principal investigator in the protocol or by protocol endment when more detailed information is considered pertinent. |
|---|---|
| 1. | Use the Common Toxicity Criteria definitions to grade the severity of the infection. |
| 2. | Specify type of infection from the following (CHOOSE ONE): |
| | BACTERIAL FUNGAL PROTOZOAL VIRAL UNKNOWN |
| 3. | Specify site of infection from the following (CHOOSE ALL THAT APPLY): |
| | BLOOD CULTURE POSITIVE BONE INFECTION CATHETER (intravenous) CATHETER (intravenous), tunnel infection CENTRAL NERVOUS SYSTEM INFECTION EAR INFECTION EYE INFECTION GASTROINTESTINAL INFECTION ORAL INFECTION PNEUMONIA SKIN INFECTION UPPER RESPIRATORY INFECTION URINARY TRACT INFECTION VAGINAL INFECTION INFECTION, not otherwise specified (Specify site,) |
| | Specify organism, if known: |
| 5. | Prophylactic antibiotic, antifungal, or antiviral therapy administration |
| | Yes No |
| | If prophylaxis was given prior to infection, please specify below: |
| | Antibiotic prophylaxis |
| | Antifungal prophylaxis |
| | Antiviral prophylaxis |
| | Other prophylaxis |


Revised March 23, 1998

## Appendix III Performance Status Scales/Scores

#### PERFORMANCE STATUS CRITERIA Karnofsky and Lansky performance scores are intended to be multiples of 10. ECOG (Zubrod) Karnofsky Lansky\* Score Description Score Description Score Description 100 100 Normal, no complaints, no Fully active, normal, evidence of disease. Fully active, able to carry on 0 all pre-disease performance Minor restrictions in physically without restriction. 90 Able to carry on normal activity; minor signs or strenuous activity. symptoms of disease. Normal activity with effort; 80 Active, but tires more quickly some signs or symptoms of Restricted in physically disease. strenuous activity but ambulatory and able to carry Cares for self, unable to carry 70 Both greater restriction of and less time out work of a light or on normal activity or do active spent in play activity. sedentary nature, e.g., light housework, office work. work. Requires occasional Up and around, but minimal active play; assistance, but is able to care keeps busy with quieter activities. Ambulatory and capable of all selfcare but unable to carry for most of his/her needs. out any work activities. Up Requires considerable Gets dressed, but lies around much of and about more than 50% of the day; no active play; able to participate in all quiet play and assistance and frequent waking hours. medical care. activities. 40 Disabled, requires special care 40 Mostly in bed; participates in quiet and assistance activities Capable of only limited 3 selfcare, confined to bed or chair more than 50% of Severely disabled, hospitalization indicated. 30 In bed; needs assistance even for quiet waking hours. Death not imminent. Often sleeping; play entirely limited to very passive activities. 20 Very sick, hospitalization 20 indicated. Death not imminent. Completely disabled. Cannot carry on any selfcare. Totally 4 confined to bed or chair. Moribund, fatal processes 10 No play; does not get out of bed. progressing rapidly.

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

 $<sup>^{\</sup>star}$ The conversion of the Lansky to ECOG scales is intended for NCI reporting purposes only.

#### Appendix IV

#### RTOG/EORTC Late Radiation Morbidity Scoring Scheme

Use for adverse event occurring greater than 90 days after radiation therapy.

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Bladder-<br>Late RT Morbidity Scoring | No change from baseline | Slight epithelial<br>atrophy/minor<br>telangiectasia<br>(microscopic hematuria) | Moderate frequency/<br>generalized<br>telangiectasia/<br>intermittent<br>macroscopic hematuria | Severe frequency and<br>dysuria/severe<br>generalized<br>telangiectasia (often<br>with petechiae);<br>frequent hematuria;<br>reduction in bladder<br>capacity (<150 mL) | Necrosis/contracted<br>bladder (capacity <100<br>mL)/severe<br>hemorrhagic cystitis |
| Bone-<br>Late RT Morbidity Scoring | No change from baseline | Asymptomatic; no growth retardation; reduced bone density | Moderate pain or<br>tenderness; growth<br>retardation; irregular<br>bone sclerosis | Severe pain or<br>tenderness; complete<br>arrest of bone growth;<br>dense bone sclerosis | Necrosis/<br>spontaneous fracture |
| Brain-<br>Late RT Morbidity Scoring | No change from baseline | Mild headache; slight lethargy | Moderate headache;<br>great lethargy | Severe headaches;<br>severe CNS dysfunction<br>(partial loss of power or<br>dyskinesia) | Seizures or paralysis;<br>coma |
| Esophagus-<br>Late RT Morbidity Scoring | No change from baseline | Mild fibrosis; slight<br>difficulty in swallowing<br>solids; no pain on<br>swallowing | Unable to take solid<br>food normally;<br>swallowing semi-solid<br>food; dilation may be<br>indicated | Severe fibrosis; able to<br>swallow only liquids;<br>may have pain on<br>swallowing; dilation<br>required | Necrosis/<br>perforation; fistula |
| Eye-<br>Late RT Morbidity Scoring | No change from baseline | Asymptomatic cataract;<br>minor corneal<br>ulceration or keratitis | Symptomatic cataract;<br>moderate corneal<br>ulceration; minor<br>retinopathy or glaucoma | Severe keratitis; severe<br>retinopathy or<br>detachment; severe<br>glaucoma | Panophthalmitis;<br>blindness |
| Heart-<br>Late RT Morbidity Scoring | No change from baseline | Asymptomatic or mild<br>symptoms; transient T<br>wave inversion and ST<br>changes; sinus<br>tachycardia >110 (at<br>rest) | Moderate angina on<br>effort; mild pericarditis;<br>normal heart size;<br>persistent abnormal T<br>wave and ST changes;<br>low QRS | Severe angina;<br>pericardial effusion;<br>constrictive pericarditis;<br>moderate heart failure;<br>cardiac enlargement;<br>EKG abnormalities | Tamponade/severe heart<br>failure/severe<br>constrictive pericarditis |
| Joint-<br>Late RT Morbidity Scoring | No change from baseline | Mild joint stiffness;<br>slight limitation of<br>movement | Moderate stiffness;<br>intermittent or moderate<br>joint pain; moderate<br>limitation of movement | Severe joint stiffness;<br>pain with severe<br>limitation of movement | Necrosis/complete fixation |
| Kidney-<br>Late RT Morbidity Scoring | No change from baseline | Transient albuminuria;<br>no hypertension; mild<br>impairment of renal<br>function; urea 25 - 35<br>mg%; creatinine 1.5 -<br>2.0 mg%; creatinine<br>clearance >75% | Persistent moderate<br>albuminuria (2+); mild<br>hypertension; no related<br>anemia; moderate<br>impairment of renal<br>function; urea >36 - 60<br>mg%; creatinine<br>clearance >50 - 74% | Severe albuminuria;<br>severe hypertension;<br>persistent anemia (<10<br>g%); severe renal<br>failure; urea >60 mg%;<br>creatinine >4 mg%;<br>creatinine clearance<br><50% | Malignant hypertension;<br>uremic coma/urea<br>>100% |
| Larynx-<br>Late RT Morbidity Scoring | No change from baseline | Hoarseness; slight arytenoid edema | Moderate arytenoid edema; chondritis | Severe edema; severe chondritis | Necrosis |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

#### Appendix IV (continued)

#### RTOG/EORTC Late Radiation Morbidity Scoring Scheme

Use for adverse event occurring greater than 90 days after radiation therapy.

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Liver-<br>Late RT Morbidity Scoring | No change from baseline | Mild lassitude; nausea;<br>dyspepsia; slightly<br>abnormal liver function | Moderate symptoms;<br>some abnormal liver<br>function tests; serum<br>albumin normal | Disabling hepatic<br>insufficiency; liver<br>function tests grossly<br>abnormal; low albumin;<br>edema or ascites | Necrosis/hepatic coma<br>or encephalopathy |
| Lung-<br>Late RT Morbidity Scoring | No change from baseline | Asymptomatic or mild<br>symptoms (dry cough);<br>slight radiographic<br>appearances | Moderate symptomatic<br>fibrosis or pneumonitis<br>(severe cough); low<br>grade fever; patchy<br>radiographic<br>appearances | Severe symptomatic<br>fibrosis or pneumonitis;<br>dense radiographic<br>changes | Severe respiratory<br>insufficiency/<br>continuous O <sub>2</sub> /assisted<br>ventilation |
| Mucous membrane-<br>Late RT Morbidity Scoring | No change from baseline | Slight atrophy and dryness | Moderate atrophy and telangiectasia; little mucus | Marked atrophy with complete dryness; severe telangiectasia | Ulceration |
| Salivary glands-<br>Late RT Morbidity Scoring | No change from baseline | Slight dryness of<br>mouth; good response<br>on stimulation | Moderate dryness of mouth; poor response on stimulation | Complete dryness of mouth; no response on stimulation | Fibrosis |
| Skin-<br>Late RT Morbidity Scoring | No change from baseline | Slight atrophy;<br>pigmentation change;<br>some hair loss | Patchy atrophy;<br>moderate telangiectasia;<br>total hair loss | Marked atrophy; gross telangiectasia | Ulceration |
| Small/Large intestine-<br>Late RT Morbidity Scoring | No change from baseline | Mild diarrhea; mild<br>cramping; bowel<br>movement 5 x daily;<br>slight rectal discharge<br>or bleeding | Moderate diarrhea and colic; bowel movement >5 x daily; excessive rectal mucus or intermittent bleeding | Obstruction or bleeding, requiring surgery | Necrosis/perforation<br>fistula |
| Spinal cord-<br>Late RT Morbidity Scoring | No change from baseline | Mild Lhermitte's syndrome | Severe Lhermitte's syndrome | Objective neurological findings at or below cord level treatment | Mono-, para-,<br>quadriplegia |
| Subcutaneous tissue-<br>Late RT Morbidity Scoring | No change from baseline | Slight induration<br>(fibrosis) and loss of<br>subcutaneous fat | Moderate fibrosis but<br>asymptomatic; slight<br>field contracture; <10%<br>linear reduction | Severe induration and<br>loss of subcutaneous<br>tissue; field contracture<br>>10% linear<br>measurement | Necrosis |
| Radiation - Other (Specify,) | None | Mild | Moderate | Severe | Life-threatening or disabling |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

#### Appendix V

#### BMT-Specific Adverse Events

Summary of BMT-Specific Adverse Events that may be used **if specified by the protocol**. These differ from the standard CTC and may be more relevant to the transplant setting. They are listed here for the convenience of investigators writing transplant protocols. They are also included in the CTC document.

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Bilirubin associated with graft versus host disease for BMT studies . | normal | ≥2 - <3 mg/100 mL | ≥3 - <6 mg/100 mL | ≥6 - <15 mg/100 mL | ≥15 mg/100 mL |
| Diarrhea associated with graft versus host disease (GVHD) for BMT studies. | none | >500 - ≤1000mL of<br>diarrhea/day | >1000 - ≤1500mL of<br>diarrhea/day | >1500mL of<br>diarrhea/day | severe abdominal pain with or without ileus |
| Diarrhea for pediatric BMT studies. | | >5 - ≤10 mL/kg of<br>diarrhea/day | >10 - ≤15 mL/kg of<br>diarrhea/day | >15 mL/kg of<br>diarrhea/day | - |
| Hepatic enlargement | absent | - | - | present | - |
| Leukocytes (total WBC) for BMT studies. | WNL | ≥2.0 - <3.0 X 10 <sup>9</sup> /L<br>≥2000 - <3000/mm <sup>3</sup> | $\geq 1.0 - <2.0 \times 10^9 / L$<br>$\geq 1000 - <2000 / mm^3$ | $\geq 0.5 - < 1.0 \times 10^9 / L$<br>$\geq 500 - < 1000 / mm^3$ | <0.5 x 10 <sup>9</sup> /L<br><500/mm <sup>3</sup> |
| Leukocytes (total WBC) for pediatric BMT studies (using age, race and sex normal values). | | ≥75 - <100% LLN | ≥50 - <75% LLN | ≥25 - 50% LLN | <25% LLN |
| Lymphopenia for pediatric<br>BMT studies (using age,<br>race and sex normal values). | mm <sup>3</sup> | ≥75-<100%LLN | ≥50-<75%LLN | ≥25-<50%LLN | <25%LLN |
| Neutrophils/granulocytes<br>(ANC/AGC) for BMT<br>studies. | WNL | ≥1.0 - <1.5 x 10 <sup>9</sup> /L<br>≥1000 - <1500/mm <sup>3</sup> | ≥0.5 - <1.0 x 10 <sup>9</sup> /L<br>≥500 - <1000/mm <sup>3</sup> | ≥0.1 - <0.5 x 10 <sup>9</sup> /L<br>≥100 - <500/mm <sup>3</sup> | <0.1 x 10 <sup>9</sup> /L<br><100/mm <sup>3</sup> |
| Platelets for BMT studies. | WNL | ≥50.0 - <75.0 x 10 <sup>9</sup> /L<br>≥50,000 - <75,000/mm <sup>3</sup> | ≥20.0 - <50.0 x 10 <sup>9</sup> /L<br>≥20,000 - <50,000/mm <sup>3</sup> | ≥10.0 - <20.0 x 10 <sup>9</sup> /L<br>≥10,000 - <20,000/mm <sup>3</sup> | <10.0 x 10 <sup>9</sup> /L<br><10,000/mm <sup>3</sup> |
| Rash/dermatitis associated with high-dose chemotherapy or BMT studies. | none | faint erythema or dry<br>desquamation | moderate to brisk<br>crythema or a patchy<br>moist desquamation,<br>mostly confined to skin<br>folds and creases;<br>moderate edema | confluent moist<br>desquamation, ≥1.5 cm<br>diameter, not confined<br>to skin folds; pitting<br>edema | skin necrosis or<br>ulceration of full<br>thickness dermis; may<br>include spontaneous<br>bleeding not included by<br>minor trauma or<br>abrasion |
| Rash/desquamation<br>associated with graft versus<br>host disease (GVHD) for<br>BMT studies. | none | macular or papular<br>eruption or erythema<br>covering <25% of body<br>surface area without<br>associated symptoms | macular or papular eruption or erythema with pruritus or other associated symptoms covering ≥25 - <50% of body surface or localized desquamation or other lesions covering ≥25 - <50% of body surface area | symptomatic<br>generalized<br>erythroderma or<br>symptomatic macular,<br>papular or vesicular<br>eruption, with bullous<br>formation, or<br>desquamation covering<br>≥50% of body surface<br>area | generalized exfoliative<br>dermatitis or ulcerative<br>dermatitis or bullous<br>formation |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998

#### Appendix V (Continued)

#### **BMT-Specific Adverse Events**

Summary of BMT-Specific Adverse Events that may be used **if specified by the protocol**. These differ from the standard CTC and may be more relevant to the transplant setting. They are listed here for the convenience of investigators writing transplant protocols. They are also included in the CTC document.

| | Grade | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Stomatitis/pharyngitis<br>(oral/pharyngeal mucositis)<br>for BMT studies. | none | painless ulcers,<br>erythema, or mild<br>soreness in the absence<br>of lesions | painful erythema,<br>edema or ulcers but can<br>swallow | painful erythema,<br>edema, or ulcers<br>preventing swallowing<br>or requiring hydration<br>or parenteral (or enteral)<br>nutritional support | severe ulceration<br>requiring prophylactic<br>intubation or resulting<br>in documented<br>aspiration pneumonia |
| Transfusion: Platelets for BMT studies. | none | 1 platelet transfusion in<br>24 hours | 2 platelet transfusions in<br>24 hours | ≥3 platelet transfusions<br>in 24 hours | platelet transfusions and<br>other measures required<br>to improve platelet<br>increment; platelet<br>transfusion<br>refractoriness associated<br>with life-threatening<br>bleeding. (e.g., HLA or<br>cross matched platelet<br>transfusions) |
| Transfusion: pRBCs for BMT studies. | none | ≤2 u pRBC in 24 hours<br>elective or planned | 3 u pRBC in 24 hours<br>elective or planned | ≥4 u pRBC in 24 hours | hemorrhage or<br>hemolysis associated<br>with life-threatening<br>anemia; medical<br>intervention required to<br>improve hemoglobin |
| Transfusion: pRBCs for pediatric BMT studies. | none | ≤15mL/kg in 24 hours<br>elective or planned | >15 - ≤30mL/kg in 24<br>hours elective or<br>planned | >30mL/kg in 24 hours | hemorrhage or<br>hemolysis associated<br>with life-threatening<br>anemia; medical<br>intervention required to<br>improve hemoglobin |
| Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura/TTP or hemolytic uremic syndrome/HUS) for BMT studies. | - | evidence of RBC<br>destruction<br>(schistocytosis) without<br>clinical consequences | evidence of RBC<br>destruction with<br>elevated creatinine (≤3<br>x ULN) | evidence of RBC<br>destruction with<br>creatinine (>3 x ULN)<br>not requiring dialysis | evidence of RBC<br>destruction with renal<br>failure requiring<br>dialysis and/or<br>encephalopathy |
| Weight gain associated with<br>Veno-Occlusive Disease<br>(VOD) for BMT studies. | <2% | ≥2 - <5% | ≥5 - <10% | ≥10% or as ascites | ≥10% or fluid retention<br>resulting in pulmonary<br>failure |


34

Revised March 23, 1998

Paclitaxel CA139387 BMS-181339 Clinical Protocol

> CTC Version 2.0 Publish Date: April 30, 1999

#### Appendix VI

#### BMT Complex/Multicomponent Events

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Note: The grading of Complex/Multicomponent Events in bone marrow transplant will be defined in the protocol. The grading scale must use the CTC criteria for grading the specific component events (adverse events). | | | | | |
| Failure to engraft | absent | mild | moderate | severe | life-threatening |
| | Also consider Hemoglobin, Neutrophils/granulocytes (ANC/AGC), Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol, Platelets, Platelets for BMT studies, if specified in the protocol | | | | |
| Graft versus host disease | absent | mild | moderate | severe | life-threatening |
| Also consider Fatigue, Rash/desquamation, Rash/desquamation associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol, Diarrhea for patients without colostomy, Diarrhea for patients with colostomy, Diarrhea associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol, Diarrhea for pediatric BMT studies, if specified in the protocol, Bilirubin, Bilirubin associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol | | | | | |
| Stem cell infusion complications | absent | mild | moderate | severe | life-threatening |
| Also consider Allergic reaction/hypersensitivity, Conduction abnormality/Atrioventricular heart block, Nodal/junctional arrhythmia/dysrhythmia, Prolonged QTc interval (QTc >0.48 seconds), Sinus bradycardia, Sinus tachycardia, Supraventricular arrhythmias (SVT/atrial fibrillation/flutter), Vasovagal episode, Ventricular arrhythmia (PVCs/bigeminy/trigeminy/ventricular tachycardia), Cardiovascular/Arrhythmia - Other (Specify, | | | | | |
| Veno-Occlusive Disease<br>(VOD) | absent | mild | moderate | severe | life-threatening |
| | | | | | ubin, Bilirubin associated with graft<br>al failure, Hepatic enlargement |

Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 DCTD, NCI, NIH, DHHS March 1998 Revised March 23, 1998